# Statistical Analysis Plan

A Phase III, Multi-Center, Randomized, Open-Label, Active-Controlled Trial to Compare the Efficacy and Safety of Recombinant Human Granulocyte Colony Stimulating Factor-Fc Fusion Protein (F-627) and Recombinant Human Granulocyte Colony Stimulating Factor (GRAN®) in the Prophylactic Treatment for Chemotherapy-Induced Neutropenia

Protocol Number SP11631

**Sponsor** Generon (Shanghai) Corporation Ltd.

**CRO** Fountain Medical Development Ltd.

Version Number 1.0

**Date** Dec. 06, 2019


Protocol Number: SP11631 Version: 1.0 Statistical Analysis Plan Version Date: Dec. 6, 2019

## TABLE OF CONTENTS

| 1 INTRODUCTION 7 1.1 Study Objectives 7 1.1.1 Primary objective 7 1.1.2 Secondary objective 8 1.1.3 Safety objective 8 1.1.4 Exploratory objective 8 1.2 Study Endpoints 8 1.2.1 Primary efficacy endpoint 8 1.2.2 Secondary efficacy endpoints 8 1.2.3 Exploratory efficacy endpoint 8 1.2.4 Safety endpoint 8 1.3 Study Design 9 1.3.1 Overall design 9 1.3.2 Randomization and blinding 13 1.3.3 Subject replacement 13 1.3.4 Sample size 13 2 BASIC PRINCIPLES FOR STATISTICAL ANALYSIS 13 2.1 General Principles 13 2.2 Definition of Analysis Set 14 2.3.1 Definition of baseline 14 2.3.2 Definition of study period 15 2.3.3 Definition of study period 15 2.3.4 Missing data processing principles 15 2.3.4 I Missing ANC data 15 2.3.5 Other data processing principles 16 2.3.5 Other data processing princ |
|---|
| 1.1.1 Primary objective 7 1.1.2 Secondary objectives 7 1.1.3 Safety objective 8 1.1.4 Exploratory objective 8 1.2 Study Endpoints 8 1.2.1 Primary efficacy endpoint 8 1.2.2 Secondary efficacy endpoints 8 1.2.3 Exploratory efficacy endpoint 8 1.2.4 Safety endpoint 8 1.3 Study Design 9 1.3.1 Overall design 9 1.3.2 Randomization and blinding 13 1.3.3 Subject replacement 13 1.3.4 Sample size 13 2 BASIC PRINCIPLES FOR STATISTICAL ANALYSIS 13 2.1 General Principles 13 2.2 Definition of Analysis Set 14 2.3 Data Processing Principles 14 2.3.1 Definition of baseline 14 2.3.2 Definition of study period 15 2.3.3 Definition of analysis window period 15 2.3.4 Missing ANC data 15 2.3.5 Other data processing principles 17 2.3.6 Data processing principles for unscheduled visits 17 2.4 Multiple Comparison 17 <tr< th=""></tr<> |
| 1.1.1 Primary objective 7 1.1.2 Secondary objectives 7 1.1.3 Safety objective 8 1.1.4 Exploratory objective 8 1.2 Study Endpoints 8 1.2.1 Primary efficacy endpoint 8 1.2.2 Secondary efficacy endpoints 8 1.2.3 Exploratory efficacy endpoint 8 1.2.4 Safety endpoint 8 1.3 Study Design 9 1.3.1 Overall design 9 1.3.2 Randomization and blinding 13 1.3.3 Subject replacement 13 1.3.4 Sample size 13 2 BASIC PRINCIPLES FOR STATISTICAL ANALYSIS 13 2.1 General Principles 13 2.2 Definition of Analysis Set 14 2.3 Data Processing Principles 14 2.3.1 Definition of baseline 14 2.3.2 Definition of study period 15 2.3.3 Definition of analysis window period 15 2.3.4 Missing ANC data 15 2.3.5 Other data processing principles 15 2.3.5 Other data processing principles for unscheduled visits 17 2.4 Multiple Comparison 17 |
| 1.1.2 Secondary objectives 7 1.1.3 Safety objective 8 1.1.4 Exploratory objective 8 1.2 Study Endpoints 8 1.2.1 Primary efficacy endpoint 8 1.2.2 Secondary efficacy endpoints 8 1.2.3 Exploratory efficacy endpoint 8 1.2.4 Safety endpoint 8 1.3 Study Design 9 1.3.1 Overall design 9 1.3.2 Randomization and blinding 13 1.3.3 Subject replacement 13 1.3.4 Sample size 13 2 BASIC PRINCIPLES FOR STATISTICAL ANALYSIS 13 2.1 General Principles 13 2.2 Definition of Analysis Set 14 2.3 Data Processing Principles 14 2.3.1 Definition of baseline 14 2.3.2 Definition of study period 15 2.3.4 Missing ANC data 15 2.3.4 Dissing ANC data 15 2.3.5 Other data processing |
| 1.1.3 Safety objective 8 1.1.4 Exploratory objective 8 1.2 Study Endpoints 8 1.2.1 Primary efficacy endpoint 8 1.2.2 Secondary efficacy endpoint 8 1.2.3 Exploratory efficacy endpoint 8 1.2.4 Safety endpoint 8 1.2.4 Safety endpoint 8 1.3.1 Overall design 9 1.3.1 Overall design 9 1.3.2 Randomization and blinding 13 1.3.3 Subject replacement 13 1.3.4 Sample size 13 2 BASIC PRINCIPLES FOR STATISTICAL ANALYSIS 13 2.1 General Principles 13 2.2 Definition of Analysis Set 14 2.3 Data Processing Principles 14 2.3.1 Definition of study period 15 2.3.2 Definition of study period 15 2.3.3 Definition of study period 15 2.3.4 Missing ANC data 15 2.3.5 Other data |
| 1.1.4 Exploratory objective 8 1.2 Study Endpoints 8 1.2.1 Primary efficacy endpoint 8 1.2.2 Secondary efficacy endpoints 8 1.2.3 Exploratory efficacy endpoint 8 1.2.4 Safety endpoint 8 1.3 Study Design 9 1.3.1 Overall design 9 1.3.2 Randomization and blinding 13 1.3.3 Subject replacement 13 1.3.4 Sample size 13 2 BASIC PRINCIPLES FOR STATISTICAL ANALYSIS 13 2.1 General Principles 13 2.2 Definition of Analysis Set 14 2.3.1 Definition of baseline 14 2.3.2 Definition of baseline 14 2.3.3 Definition of study period 15 2.3.4 Missing data processing principles 15 2.3.4 Imputation of missing dates 16 2.3.5 Other data processing principles 17 2.3.6 Data processing principles for unscheduled visits 17 2.4 Multiple Comparison 17 2.5 Subgroup Analysis 17 2.6 Combination of Study Sites 18 |
| 1.2 Study Endpoints 8 1.2.1 Primary efficacy endpoint 8 1.2.2 Secondary efficacy endpoints 8 1.2.3 Exploratory efficacy endpoint 8 1.2.4 Safety endpoint 8 1.3 Study Design 9 1.3.1 Overall design 9 1.3.2 Randomization and blinding 13 1.3.3 Subject replacement 13 1.3.4 Sample size 13 2 BASIC PRINCIPLES FOR STATISTICAL ANALYSIS 13 2.1 General Principles 13 2.2 Definition of Analysis Set 14 2.3 Data Processing Principles 14 2.3.1 Definition of baseline 14 2.3.2 Definition of study period 15 2.3.3 Definition of analysis window period 15 2.3.4 Missing data processing principles 15 2.3.4.2 Imputation of missing dates 15 2.3.5 Other data processing principles 17 2.3.6 Data processing principles for unscheduled visits 17 2.4 Multiple Comparison 17 2.5 Subgroup Analysis 17 2.6 Combination of Study Sites 18 |
| 1.2.1 Primary efficacy endpoint. 8 1.2.2 Secondary efficacy endpoints 8 1.2.3 Exploratory efficacy endpoint. 8 1.2.4 Safety endpoint. 8 1.3 Study Design 9 1.3.1 Overall design. 9 1.3.2 Randomization and blinding. 13 1.3.3 Subject replacement 13 1.3.4 Sample size 13 2 BASIC PRINCIPLES FOR STATISTICAL ANALYSIS 13 2.1 General Principles 13 2.2 Definition of Analysis Set 14 2.3 Data Processing Principles 14 2.3.1 Definition of baseline 14 2.3.2 Definition of study period 15 2.3.3 Definition of analysis window period 15 2.3.4 Missing data processing principles 15 2.3.4.1 Missing ANC data 15 2.3.5 Other data processing principles 17 2.3.6 Data processing principles for unscheduled visits 17 2.4 Multiple Comparison 17 2.5 Subgroup Analysis 17 2.6 Combination of Study Sites 18 |
| 1.2.2 Secondary efficacy endpoints 8 1.2.3 Exploratory efficacy endpoint 8 1.2.4 Safety endpoint 8 1.3 Study Design 9 1.3.1 Overall design 9 1.3.2 Randomization and blinding 13 1.3.3 Subject replacement 13 1.3.4 Sample size 13 2 BASIC PRINCIPLES FOR STATISTICAL ANALYSIS 13 2.1 General Principles 13 2.2 Definition of Analysis Set 14 2.3 Data Processing Principles 14 2.3.1 Definition of baseline 14 2.3.2 Definition of study period 15 2.3.3 Definition of analysis window period 15 2.3.4 Missing data processing principles 15 2.3.4.1 Missing ANC data 15 2.3.4.2 Imputation of missing dates 15 2.3.5 Other data processing principles for unscheduled visits 17 2.4 Multiple Comparison 17 2.5 Subgroup Analysis 17 2.6 Combination of Study Sites 18 |
| 1.2.3 Exploratory efficacy endpoint 8 1.2.4 Safety endpoint 8 1.3 Study Design 9 1.3.1 Overall design 9 1.3.2 Randomization and blinding 13 1.3.3 Subject replacement 13 1.3.4 Sample size 13 2 BASIC PRINCIPLES FOR STATISTICAL ANALYSIS 13 2.1 General Principles 13 2.2 Definition of Analysis Set 14 2.3 Data Processing Principles 14 2.3.1 Definition of baseline 14 2.3.2 Definition of study period 15 2.3.3 Definition of analysis window period 15 2.3.4 Missing data processing principles 15 2.3.4.1 Missing ANC data 15 2.3.5 Other data processing principles 15 2.3.5 Other data processing principles 17 2.4 Multiple Comparison 17 2.5 Subgroup Analysis 17 2.6 Combination of Study Sites 18 |
| 1.2.4 Safety endpoint 8 1.3 Study Design 9 1.3.1 Overall design 9 1.3.2 Randomization and blinding 13 1.3.3 Subject replacement 13 1.3.4 Sample size 13 2 BASIC PRINCIPLES FOR STATISTICAL ANALYSIS 13 2.1 General Principles 13 2.2 Definition of Analysis Set 14 2.3 Data Processing Principles 14 2.3.1 Definition of baseline 14 2.3.2 Definition of study period 15 2.3.3 Definition of analysis window period 15 2.3.4 Missing data processing principles 15 2.3.4.1 Missing ANC data 15 2.3.4.2 Imputation of missing dates 16 2.3.5 Other data processing principles 17 2.3.6 Data processing principles for unscheduled visits 17 2.4 Multiple Comparison 17 2.5 Subgroup Analysis 17 2.6 Combination of Study Sites 18 |
| 1.3 Study Design 9 1.3.1 Overall design 9 1.3.2 Randomization and blinding 13 1.3.3 Subject replacement 13 1.3.4 Sample size 13 2 BASIC PRINCIPLES FOR STATISTICAL ANALYSIS 13 2.1 General Principles 13 2.2 Definition of Analysis Set 14 2.3 Data Processing Principles 14 2.3.1 Definition of baseline 14 2.3.2 Definition of study period 15 2.3.3 Definition of analysis window period 15 2.3.4 Missing data processing principles 15 2.3.4.1 Missing ANC data 15 2.3.5 Other data processing principles 16 2.3.5 Other data processing principles 17 2.3.6 Data processing principles for unscheduled visits 17 2.4 Multiple Comparison 17 2.5 Subgroup Analysis 17 2.6 Combination of Study Sites 18 |
| 1.3.1 Overall design 9 1.3.2 Randomization and blinding 13 1.3.3 Subject replacement 13 1.3.4 Sample size 13 2 BASIC PRINCIPLES FOR STATISTICAL ANALYSIS 13 2.1 General Principles 13 2.2 Definition of Analysis Set 14 2.3 Data Processing Principles 14 2.3.1 Definition of baseline 14 2.3.2 Definition of study period 15 2.3.3 Definition of analysis window period 15 2.3.4 Missing data processing principles 15 2.3.4.1 Missing ANC data 15 2.3.5 Other data processing principles 16 2.3.5 Other data processing principles for unscheduled visits 17 2.4 Multiple Comparison 17 2.5 Subgroup Analysis 17 2.6 Combination of Study Sites 18 |
| 1.3.3 Subject replacement 13 1.3.4 Sample size 13 2 BASIC PRINCIPLES FOR STATISTICAL ANALYSIS 13 2.1 General Principles 13 2.2 Definition of Analysis Set 14 2.3 Data Processing Principles 14 2.3.1 Definition of baseline 14 2.3.2 Definition of study period 15 2.3.3 Definition of analysis window period 15 2.3.4 Missing data processing principles 15 2.3.4.1 Missing ANC data 15 2.3.4.2 Imputation of missing dates 16 2.3.5 Other data processing principles 17 2.3.6 Data processing principles for unscheduled visits 17 2.4 Multiple Comparison 17 2.5 Subgroup Analysis 17 2.6 Combination of Study Sites 18 |
| 1.3.4 Sample size 13 2 BASIC PRINCIPLES FOR STATISTICAL ANALYSIS 13 2.1 General Principles 13 2.2 Definition of Analysis Set 14 2.3 Data Processing Principles 14 2.3.1 Definition of baseline 14 2.3.2 Definition of study period 15 2.3.3 Definition of analysis window period 15 2.3.4 Missing data processing principles 15 2.3.4.1 Missing ANC data 15 2.3.4.2 Imputation of missing dates 16 2.3.5 Other data processing principles 17 2.3.6 Data processing principles for unscheduled visits 17 2.4 Multiple Comparison 17 2.5 Subgroup Analysis 17 2.6 Combination of Study Sites 18 |
| 2 BASIC PRINCIPLES FOR STATISTICAL ANALYSIS 13 2.1 General Principles 13 2.2 Definition of Analysis Set 14 2.3 Data Processing Principles 14 2.3.1 Definition of baseline 14 2.3.2 Definition of study period 15 2.3.3 Definition of analysis window period 15 2.3.4 Missing data processing principles 15 2.3.4.1 Missing ANC data 15 2.3.4.2 Imputation of missing dates 16 2.3.5 Other data processing principles 17 2.3.6 Data processing principles for unscheduled visits 17 2.4 Multiple Comparison 17 2.5 Subgroup Analysis 17 2.6 Combination of Study Sites 18 |
| 2.1 General Principles 13 2.2 Definition of Analysis Set 14 2.3 Data Processing Principles 14 2.3.1 Definition of baseline 14 2.3.2 Definition of study period 15 2.3.3 Definition of analysis window period 15 2.3.4 Missing data processing principles 15 2.3.4.1 Missing ANC data 15 2.3.4.2 Imputation of missing dates 16 2.3.5 Other data processing principles 17 2.3.6 Data processing principles for unscheduled visits 17 2.4 Multiple Comparison 17 2.5 Subgroup Analysis 17 2.6 Combination of Study Sites 18 |
| 2.1 General Principles 13 2.2 Definition of Analysis Set 14 2.3 Data Processing Principles 14 2.3.1 Definition of baseline 14 2.3.2 Definition of study period 15 2.3.3 Definition of analysis window period 15 2.3.4 Missing data processing principles 15 2.3.4.1 Missing ANC data 15 2.3.4.2 Imputation of missing dates 16 2.3.5 Other data processing principles 17 2.3.6 Data processing principles for unscheduled visits 17 2.4 Multiple Comparison 17 2.5 Subgroup Analysis 17 2.6 Combination of Study Sites 18 |
| 2.2 Definition of Analysis Set142.3 Data Processing Principles142.3.1 Definition of baseline142.3.2 Definition of study period152.3.3 Definition of analysis window period152.3.4 Missing data processing principles152.3.4.1 Missing ANC data152.3.4.2 Imputation of missing dates162.3.5 Other data processing principles172.3.6 Data processing principles for unscheduled visits172.4 Multiple Comparison172.5 Subgroup Analysis172.6 Combination of Study Sites18 |
| 2.3 Data Processing Principles142.3.1 Definition of baseline142.3.2 Definition of study period152.3.3 Definition of analysis window period152.3.4 Missing data processing principles152.3.4.1 Missing ANC data152.3.4.2 Imputation of missing dates162.3.5 Other data processing principles172.3.6 Data processing principles for unscheduled visits172.4 Multiple Comparison172.5 Subgroup Analysis172.6 Combination of Study Sites18 |
| 2.3.1 Definition of baseline142.3.2 Definition of study period152.3.3 Definition of analysis window period152.3.4 Missing data processing principles152.3.4.1 Missing ANC data152.3.4.2 Imputation of missing dates162.3.5 Other data processing principles172.3.6 Data processing principles for unscheduled visits172.4 Multiple Comparison172.5 Subgroup Analysis172.6 Combination of Study Sites18 |
| 2.3.2 Definition of study period 15 2.3.3 Definition of analysis window period 15 2.3.4 Missing data processing principles 15 2.3.4.1 Missing ANC data 15 2.3.4.2 Imputation of missing dates 16 2.3.5 Other data processing principles 17 2.3.6 Data processing principles for unscheduled visits 17 2.4 Multiple Comparison 17 2.5 Subgroup Analysis 17 2.6 Combination of Study Sites 18 |
| 2.3.3 Definition of analysis window period 15 2.3.4 Missing data processing principles 15 2.3.4.1 Missing ANC data 15 2.3.4.2 Imputation of missing dates 16 2.3.5 Other data processing principles 17 2.3.6 Data processing principles for unscheduled visits 17 2.4 Multiple Comparison 17 2.5 Subgroup Analysis 17 2.6 Combination of Study Sites 18 |
| 2.3.4 Missing data processing principles 15 2.3.4.1 Missing ANC data 15 2.3.4.2 Imputation of missing dates 16 2.3.5 Other data processing principles 17 2.3.6 Data processing principles for unscheduled visits 17 2.4 Multiple Comparison 17 2.5 Subgroup Analysis 17 2.6 Combination of Study Sites 18 |
| 2.3.4.1 Missing ANC data 15 2.3.4.2 Imputation of missing dates 16 2.3.5 Other data processing principles 17 2.3.6 Data processing principles for unscheduled visits 17 2.4 Multiple Comparison 17 2.5 Subgroup Analysis 17 2.6 Combination of Study Sites 18 |
| 2.3.4.2 Imputation of missing dates |
| 2.3.5 Other data processing principles172.3.6 Data processing principles for unscheduled visits172.4 Multiple Comparison172.5 Subgroup Analysis172.6 Combination of Study Sites18 |
| 2.3.6 Data processing principles for unscheduled visits172.4 Multiple Comparison172.5 Subgroup Analysis172.6 Combination of Study Sites18 |
| 2.4 Multiple Comparison172.5 Subgroup Analysis172.6 Combination of Study Sites18 |
| 2.6 Combination of Study Sites 18 |
| • |
| 3 STATISTICAL ANALYSIS |
| 3.1 Basic Subject Information 18 |
| 3.1.1 Enrollment and study completion |
| 3.1.2 Protocol deviation |
| 3.1.3 Demographics and baseline characteristics 18 |
| 3.1.4 Medical history, history of breast cancer surgery, and concomitant non-drug treatment19 |
| 3.1.5 Prior medications and concomitant medications |
| 3.1.6 Exposure to drugs |
| 3.2 Efficacy Analysis/Pharmacokinetic Analysis |
| 3.2.1 Primary efficacy analysis 21 |
| 3.2.1.1 Primary analysis 21 |

| Protocol Number: SP11631 | Statistica | al Ana | lysis | Pla | n |
|--------------------------|------------|--------|-------|-----|------|
| Version: 1.0 | Version | Date: | Dec. | 6, | 2019 |

| | 3.2.1.2 Sensitivity analysis | 21 |
|---|---|---|
| | 3.2.2 Secondary efficacy analysis | |
| | 3.2.2.1 Incidence rate of grade 3 or grade 4 neutropenia in each cycle | |
| | 3.2.2.2 Durations (days) of grade 3 or 4 neutropenia in cycles 2–4 | |
| | 3.2.2.3 Incidence rate and duration (days) of grade 4 neutropenia in each cycle | 22 |
| | 3.2.2.4 Overall duration (days) of grade 3 or 4 neutropenia in overall 4 cycles | 22 |
| | 3.2.2.5 Incidence rate and duration (days) of grade 2 or greater neutropenia in each cycle | 22 |
| | 3.2.2.6 Incidence rate of febrile neutropenia (FN) | 23 |
| | 3.2.2.7 ANC - time profile | 23 |
| | 3.2.2.8 ANC nadir | |
| | 3.2.2.9 Time (days) of ANC nadir recovers to 2.0 × 10 <sup>9</sup> /L in each cycle | 23 |
| | 3.3 Safety Analysis | |
| | 3.3.1 Adverse event | |
| | 3.3.2 Laboratory measurements | |
| | 3.3.3 Vital signs, physical examination, ECG, and abdominal ultrasound | |
| | 3.3.3.1 Vital signs | |
| | 3.3.3.2 Physical examination | |
| | 3.3.3.3 Electrocardiogram (ECG) | |
| | 3.3.3.4 Abdominal ultrasound | |
| | 3.3.4 Other safety analysis | |
| | 3.4 Exploratory Analysis of F-627 Immunogenicity | |
| | 3.5 Interim Analysis | 28 |
| 4 | MODIFICATIONS TO THE ORIGINAL ANALYSIS PLAN | 28 |
| 5 | REFERENCES | 28 |
| A | ppendix 1 SAS Procedures for Imputation of Monotone Missing ANC Data | 29 |

# **ABBREVIATIONS**

| Abbreviations | Definition |
|---|---|
| AE | Adverse event |
| ANC | Absolute neutrophil count |
| ATC | Anatomical Therapeutic Chemical (ATC) Classification System |
| BMI | Body mass index |
| BSA | Body surface area |
| CI | Confidence interval |
| CRF | Case Report Form |
| CTCAE | Common Terminology Criteria for Adverse Events |
| EC | Epirubicin + Cyclophosphamide (Name of Chemotherapy Regimen) |
| FAS | Full analysis set |
| Hb | Hemoglobin |
| ICH | International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use |
| ITT | Intent-to-treat |
| MedDRA | Medical Dictionary for Regulatory Activities |
| NCI CTC | National Cancer Institute Common Terminology Criteria |
| PLT | Platelet |
| PP | Per-protocol |
| PT | Preferred term |
| SAE | Serious adverse event |
| SAP | Statistical Analysis Plan |
| SE | Standard error |
| SD | Standard deviation |
| SOC | System organ class |
| SS | Safety analysis set |
| TEAE | Treatment-emergent adverse event |
| WHODD | World Health Organization Drug Dictionary |


#### 1 INTRODUCTION

This is a Statistical Analysis Plan (SAP) that provides data processing principles and statistical analysis methods to analyze and report the efficacy and safety of the phase III clinical trial (protocol number: SP11631) sponsored by Generon (Shanghai) Corporation Ltd.

This SAP is prepared based on the protocol numbered SP11631 (version/date: 4.1/Aug. 7, 2018).

#### 1.1 Study Objectives

## 1.1.1 Primary objective

The primary objective of this study is to compare the efficacy of recombinant human granulocyte colony stimulating factor-Fc fusion protein (F-627) versus recombinant human granulocyte colony stimulating factor (GRAN®) in the first cycle of prophylactic treatment in subjects with breast cancer receiving EC chemotherapy. The primary endpoint is the duration (days) of grade 3 (moderate) or 4 (severe) neutropenia in cycle 1, that is, the number of days with absolute neutrophil count (ANC)  $< 1.0 \times 10^9$ /L in cycle 1.

## 1.1.2 Secondary objectives

Secondary objectives include:

- The incidence rate of grade 3 or 4 neutropenia (ANC  $< 1.0 \times 10^9/L$  and  $< 0.5 \times 10^9/L$ , respectively) in each cycle
- The durations (days) of grade 3 or 4 neutropenia (ANC  $< 1.0 \times 10^9/L$  and  $< 0.5 \times 10^9/L$ , respectively) in cycles 2–4
- The incidence rate and duration (days) of grade 4 neutropenia (ANC  $< 0.5 \times 10^9/L$ ) in each cycle
- The overall duration (days) of grade 3 and 4 neutropenia (ANC  $< 1.0 \times 10^9$ /L and ANC  $< 0.5 \times 10^9$ /L, respectively) in overall 4 cycles
- The incidence rate and duration (days) of grade 2 or greater neutropenia (ANC  $< 1.5 \times 10^9/L$ ) in each cycle
- The incidence rate of febrile neutropenia (FN) (defined as ANC < 1.0×10<sup>9</sup>/L; a single measurement of body temperature > 38.3 °C or a temperature ≥ 38.0 °C sustained over 1 hr)
- ANC-time profile
- The ANC nadir from day 3 to day 13 of cycle 1
- The time (days) of ANC nadir recovers to  $2.0 \times 10^9/L$  or greater (ANC  $\ge 2.0 \times 10^9/L$ ) in each cycle


## 1.1.3 Safety objective

To evaluate the safety of F-627 and GRAN<sup>®</sup>. Safety endpoints include adverse events (AEs)/serious adverse events (SAEs), laboratory measurements, 12-lead ECG, abdominal ultrasound, physical examinations, vital signs, and symptoms. GRAN<sup>®</sup> was used as the active comparator.

## 1.1.4 Exploratory objective

To evaluate the immunogenic potential of F-627 by testing serum anti-F-627 antibodies.

#### 1.2 Study Endpoints

#### 1.2.1 Primary efficacy endpoint

The primary endpoint is the duration (days) of grade 3 (moderate) or 4 (severe) neutropenia, that is, the number of days in which ANC is  $< 1.0 \times 10^9/L$  in cycle 1. The equation for calculating the duration (days) is as follows:

Duration (days) = (the last day with ANC  $< 1.0 \times 10^9/L$  during the first 13 days of the cycle) – (the first day with ANC  $< 1.0 \times 10^9/L$  during the first 13 days of the cycle) + 1

Note: In the absence of ANC  $< 1.0 \times 10^9 / L$  record during the first 13 days of the cycle, the duration (days) = 0. The data from central laboratory is preferred for the ANC analysis. If the ANC data in both central laboratory and local laboratory are missing, the missing data will be imputed. See Section 2.3.4.1 for the imputation method.

## 1.2.2 Secondary efficacy endpoints

The secondary efficacy endpoints are the same as that of the secondary objectives.

The duration calculation method of neutrophil-related endpoints in each cycle is the same as that of the primary efficacy endpoint.

The rates in secondary efficacy endpoints are calculated based on the evaluable number of subjects, that is, the denominator of each cycle rate is the number of subjects with evaluable data of this cycle in the corresponding population set; and the denominator of the entire treatment period rate is the number of subjects with evaluable post-baseline data in the corresponding population set.

For the calculation of the time (days) of ANC nadir recovers to  $2.0 \times 10^9/L$  in each cycle, the minimum value is the ANC nadir during the day 3 to 13 of each cycle. In the absence of ANC  $< 2.0 \times 10^9/L$  record during the day 3 to 13 of the cycle, the recovery time = 0 day. If more than one nadir is recorded during the day 3 to 13 of the cycle, the first one will be used.

## 1.2.3 Exploratory efficacy endpoint

Same as the exploratory objective.

## 1.2.4 Safety endpoint

Same as the safety objective.


#### 1.3 Study Design

## 1.3.1 Overall design

This is a multi-center, randomized, open-label, active-controlled phase III clinical trial. A total of 240 postoperative subjects with breast cancer will be enrolled to receive at least 4 cycles of EC chemotherapy, namely: epirubicin (Ellence®) 100 mg/m² + cyclophosphamide 600 mg/m², i.v. on day 1 of each cycle, repeat cycle every 21 days for 4 cycles. After completing the evaluation for the overall 4 cycles, subjects will receive subsequent treatments according to routine clinical practice. The investigator must ensure that the first cycle of treatment follows the recommended dosages for chemotherapy. In cycles 2–4, dose delays and reductions due to toxicities other than myelotoxicity (such as cardiotoxicity) are permitted. Dosages are permitted to be individualized based on subject's condition.

As shown in the flow diagram in Figure 1, patients will be randomized in a 1:1 ratio to F-627 arm or GRAN® arm before the start of chemotherapy on day 1 of cycle 1. Treatment allocation will remain unchanged during the entire treatment period (4 cycles). On day 3 of each cycle, that is,  $48 \pm 4$  hrs after the start of chemotherapy, subjects will receive F-627 (20 mg/dose, s.c.) or GRAN® (5  $\mu$ g/kg/day, s.c., once daily [ $\pm 4$  hrs] for  $\leq 2$  weeks or until ANC recovers to  $5.0 \times 10^9$ /L from nadir [the investigator may refer to the ANC results from the Department of Laboratory Medicine of each study site to decide when to discontinue GRAN®]). All laboratory measurements will be performed at individual study sites except for the routine blood test (ANC) in cycle 1, which is performed at the central laboratory. AEs/SAEs will be recorded, along with the results of laboratory measurements, 12-lead ECGs, and abdominal ultrasounds.

The last visit will be completed 3 weeks after the last chemotherapy dose. A follow-up visit by telephone will be completed 30 days after the last dose. The schedule of study procedures is detailed in Table 1.




Figure 1. Study flow diagram


 Table 1
 Schedule of study procedures

| Treatment | Screening | | Cycles 1–4 | | End of study |
|---|---|---|---|---|---|
| period<br>Items | period<br>Day –21 to<br>Day –1 | Day 1 | Day 3 | Days 3–21 | Day 21 of cycle 4 <sup>j</sup> |
| Informed consent form | × | | | | |
| Inclusion/<br>exclusion criteria | × | | | | |
| Tumor history | × | | | | |
| Concomitant diseases | × | × | × | × | × |
| Combined medications | × | × | × | × | × |
| Physical examination <sup>a</sup> | × | × | | | × |
| Weight and height <sup>b</sup> | × | × | | | × |
| Blood pressure and heart rate | × | × | | | × |
| Body temperature <sup>c</sup> | × | × | × | × | × |
| Abdominal ultrasound <sup>d</sup> | × | × | | | × |
| 12-lead ECG <sup>d</sup> | × | × | | | × |
| Echocardiography | × | | | | |
| Chest X-ray or CT | × | | | | |
| Laboratory measurements | | | | | |
| Routine blood teste | × | × | × | × | × |
| Clinical chemistry | × | × | | | × |
| Urinalysis | × | × | | | × |
| Pregnancy test | × | | | | × |
| Serum Anti-F-627<br>Antibodies <sup>f</sup> | | × | | | × |
| Chemotherapy <sup>g</sup> | | × | | | |
| Study drugsh | | | × | × | |
| Adverse eventi | × | × | × | × | × |

## Notes:

- a. A complete physical examination is required during screening. Corresponding physical examinations on day 1 of cycles 1–4 (vital organs) are completed based on subject condition;
- b. Height is only measured during screening. Weight is measured on day 1 of each cycle (measurements within 3 days of the cycle are acceptable) and at the end of the study;
- c. Body temperature is measured during screening, on day 1 of each cycle, and at the end of the study. On days 3–21 of each cycle, temperature is measured as clinically indicated when ANC  $< 1.0 \times 10^9/L$ ;
- d. Abdominal ultrasound is performed during screening or before the start of cycle 1 and at the end of the study. The time window for abdominal ultrasound is +/- 3 days. The 12-lead ECG is performed during screening (ECGs performed within 7 days prior to randomization can be used as the result for cycle 1), before the start of each cycle, and at the end of the study. The time window for 12-lead ECG is +/-3 days;


e. Routine blood test is performed on days 3, 5, 7, 8, 9, 10, 11, 13, 15, and 21 of cycle 1 and on days 3, 5, 7, 9, 11, 13, 15, and 21 of cycles 2–4. Laboratory measurements (routine blood test, clinical chemistry, urinalysis, and pregnancy test) within 7 days before the chemotherapy in cycle 1 (day 1) are acceptable. The time window for laboratory measurements (routine blood test, clinical chemistry, routine urinalysis, and pregnancy test) before cycles 2–4 is –3 days:

- f. Blood samples are collected on day 1 (± 1 day) of each cycle, on day 21 (± 1 day) of cycle 4, and 90 days (± 7 days) after the last visit (day 21 of cycle 4) to test the serum anti-F-627 antibodies. Results of the test on day 1 of cycle 1 are used as the baseline data
- g. The investigator will decide on the dose and time of the next chemotherapy based on the subject's actual conditions. Results of routine blood test must meet the following criteria prior to the start of chemotherapy of the next cycle:  $ANC \ge 2.0 \times 10^9/L$ ,  $PLT \ge 80 \times 10^9/L$ , and liver and renal functions in accordance with "Inclusion Criteria". A 14-day recovery period is permitted if these criteria are not met prior to the scheduled chemotherapy in cycles 2, 3, and 4. If the criteria described above are still not met after 14 days, the subject will not be enrolled in the study of cycle 2, cycle 3, or cycle 4.
- h. On day 3 of each cycle ( $48 \pm 4$  hours after the start of chemotherapy), subjects will receive F-627 20 mg subcutaneously or GRAN® ( $5 \mu g/kg/day$ , s.c., once daily [ $\pm 4$  hrs] for  $\leq 2$  weeks or until ANC recovers to  $5.0 \times 10^9/L$  from nadir [the investigator may refer to ANC results from the Department of Laboratory Medicine of each study site to decide when to discontinue GRAN®1):
- i. AEs are evaluated according to NCI CTCAE 4.03. AEs that occur within 30 days after the last dose are included in the safety evaluation. SAEs should be reported;
- j. The last visit should be completed on day 21 (± 1 day) of cycle 4. A follow-up visit by telephone should be completed in 30 days (± 3 days) after the last dose;

Notes: Routine blood tests in cycle 1 and all serum anti-F-627 antibody assays are performed at the central laboratory. Routine blood test, clinical chemistry, pregnancy test, and urinalysis during screening, cycles 2–4, and at the end of the study are performed at the study sites. In cycle 1, when necessary, investigators can conduct routine blood test at their respective study sites based on subject's condition, in order to provide necessary treatment to prevent the risks from neutropenia. Appropriate measures are taken for chemotherapy-related toxicities based on the investigator's clinical judgment and routine clinical practice.


#### 1.3.2 Randomization and blinding

This is a randomized and open-label trial. No blinding is applied in this study. Each subject will be assigned with a random number by an independent statistician who does not participate in the study. A randomized allocation table will be generated by block randomization through PLAN using SAS 9.4. Central randomization will be performed in this study using the Interactive Web-Response System (IWRS). After eligible patients provide a signed informed consent form (ICF), authorized investigators will log in to the IWRS system and key in relevant information, and subjects will be randomized to 2 different arms, i.e. F-627 or GRAN® through the system.

#### 1.3.3 Subject replacement

In this trial, there is no plan on replacing any subject who terminates the trial early.

#### 1.3.4 Sample size

The primary endpoint is the duration (days) of grade 3 or 4 neutropenia in cycle 1. The non-inferiority margin for F-627 and GRAN<sup>®</sup> is defined to be 1 day<sup>3-5</sup>. Although the maximum standard deviations for the two F-627 phase II clinical trials (SP-CDR-1-1302 and GC-627-02) were 1.33 and 1.58 days, respectively, it is conservatively assumed that the standard deviation for this study is 1.75 days. In the case of a one-sided  $\alpha = 0.025$  and a power of 95%, 94 subjects are required for each arm; and in consideration of a 15–20% drop-out rate, 120 subjects are required for each arm (a total of 240 subjects).

#### 2 BASIC PRINCIPLES FOR STATISTICAL ANALYSIS

#### 2.1 General Principles

Statistical analyses will be performed using SAS 9.4 or above. Unless otherwise stated, two-sided 95% CI will be used. All data in the database will be tabulated. Unless otherwise stated, all summary tables will be summarized according to the scheduled visits. The unscheduled visits will be tabulated only. Data are tabulated by treatment arm, subject number, and test time point. Continuous variables are summarized by descriptive statistics, including number of cases, mean, median, standard deviation, minimum, and maximum. Classification parameters are described by the number of cases, number of missing cases, number of classified cases, and percentages. Unless otherwise stated, percentages are calculated with non-missing data as the denominator.

For the principle of decimal places, unless otherwise stated, the minimum and maximum values are rounded to the same decimal places as the data collected; one more decimal place than the data collected is required for means and medians, and two more for standard deviations and standard errors; no value with more than 3 decimal places is allowed. The differences estimated by Hodges-Lehmann are rounded to 1 decimal place and the confidence intervals (CIs) are rounded to 2 decimal places. Rates (%) and rate differences (%) are rounded to 1 decimal place, and CIs of rates (%) and rate differences (%) are rounded to 2 decimal places.


Unless otherwise stated, a one-sided test with a significance level of  $\alpha = 0.025$  is used in the non-inferiority test, and a two-sided test with a significance level of  $\alpha = 0.05$  is used in other tests. All P values are rounded to three decimal places. If a P value is less than 0.001, it is expressed as "< 0.001". If a P value is greater than 0.999, it is expressed as "> 0.999".

## 2.2 Definition of Analysis Set

Efficacy analysis is performed based on full analysis set and per-protocol set. Safety analysis is performed based on safety analysis set. Definitions of each analysis set are as follows:

Full analysis set (FAS): All randomized subjects who have received the study drug and underwent at least one post-baseline efficacy evaluation. The FAS is primarily used for efficacy evaluation.

Per-protocol (PP) set A: Subjects in FAS and without serious protocol deviations, serious medication noncompliance, loss to follow-up, or withdrawal during cycle 1. The PP set A is used for PP set analyses of endpoints only related to cycle 1.

Per-protocol set B: subjects in FAS and without serious protocol deviations, serious medication noncompliance, loss to follow-up, or withdrawal in any cycle. The PP set B is used for PP set analyses of endpoints only related to overall cycles. The PP set is primarily used for efficacy evaluation.

Safety set (SS): All randomized subjects who have received at least one dose of the study drugs. The SS is primarily used for safety evaluation.

Immunogenicity analysis set: subjects with at least one result of serum anti-F-627 antibody assay after F-627 treatment.

Serious protocol deviations are confirmed before the database locking. The definitions of serious protocol deviations are as follows:

- Serious violations of inclusion/exclusion criteria;
- Administration of a wrong study drug (not the originally randomized treatment);
- Administration of a wrong dose:
- Other serious protocol deviations considered by the sponsor.

## 2.3 Data Processing Principles

#### 2.3.1 Definition of baseline

Unless otherwise stated, baseline for the entire trial is defined as the last effective value prior to the first chemotherapy (including the day of the first chemotherapy). The baseline of laboratory measurements (routine blood test, clinical chemistry, urinalysis) in cycles 2–4 is defined as the last effective value measured within –3 days (including the day of starting the chemotherapy in that cycle) before the start of chemotherapy in that cycle; for data collected at the same day, the one from the central laboratory is preferred.


The descriptive statistics of baseline characteristics are based on a population without missing results. The change from baseline is defined as the difference between visit observations and baseline results.

For the serum anti-F-627 antibody, the test result on day 1 of cycle 1 is the baseline.

In the absence of such defined value above, the baseline is missing.

## 2.3.2 Definition of study period

The calculation of study period is about calculating the time interval between the event occurrence date and the start date of chemotherapy with reference to the start date of chemotherapy.

If the event occurrence date is at or after the start date of chemotherapy, the study period = event occurrence date - start date of chemotherapy (day 1) + 1.

If the event occurrence date is before the start date of chemotherapy, the study period = event occurrence date - start date of chemotherapy (day 1).

## 2.3.3 Definition of analysis window period

The analysis window period is defined in accordance with the baseline (as defined above) and only for the routine blood test, clinical chemistry, and urinalysis during the visit on day 1 of each cycle. For other laboratory measurements during the visits not on day 1 of each cycle, unless otherwise stated, the analysis is performed according to the scheduled visits and no window period is defined.

#### 2.3.4 Missing data processing principles

#### 2.3.4.1 Missing ANC data

As stated above, the ANC on day 1 of each cycle is the baseline of that cycle according to the window period (as defined above) principle. For data collected at the same visit, the one from the central laboratory is preferred for analysis. In the absence of ANC data in both central laboratory and local laboratory, the missing data will be imputed. The imputation method is as follows:

If the baseline ANC of cycle 1 is missing, the mean baseline value of FAS is imputed.

Imputation method for other missing ANC data is as follows (for scheduled visits only):

- 1) If ANC data between cycles are missing, the missing data of the first 13 days of each cycle are imputed by linear interpolation.
- 2) For the subsequent monotone missing ANC due to the withdrawal within the first 13 days in cycle 1, if the last ANC  $>= 2.0 \times 10^9$ /L after ANC nadir, the last ANC is carried forward for the missing ANC of the first 13 days of cycle 1; if the last ANC is the nadir, it is not carried forward.


The monotone missing ANCs after step 2) are imputed by sequential regression, starting from the first scheduled visit (day 3 of cycle 1) after day 1 (baseline) of cycle 1. The covariates for the imputation model include age, arm, chemotherapy, and ANC on day 1 of cycle 1. The missing data of the next scheduled visit is imputed after this is completed, with the ANC of the previous visit (including the value imputed) as an additional prediction factor of the covariates of the model. In this way, the missing data are imputed until day 13 of cycle 1. See Appendix 1 for the imputation procedures by SAS.

#### 2.3.4.2 Imputation of missing dates

In general, no missing date is imputed unless part of the date is missing or otherwise stated.

#### Imputation principles for first diagnosis date:

- A missing year (or all parts are missing) is not imputed;
- If only the day is missing, it is imputed by the 15th day of that month;
- If both month and day are missing, it is imputed by Jul. 1.

#### Imputation principles for combined medication start/end date

Imputation of combined medication start date:

- If only the day is missing, it is imputed by the 1st day of that month;
- If both the month and day are missing, it is imputed by Jan. 1;
- If all the year, month, and day are missing, it is imputed by the date before the first administration date of the study drug.

Imputation of combined medication end date:

- If only the day is missing, the last day of that month is used;
- If both the month and day are missing, it is imputed by Dec. 31;
- If all the year, month, and day are missing, it is imputed by the last administration date of the study drug + 30 days.

In the case of a death, if the combined medication end date imputed is after the date of death, the date of death is used instead.

#### Imputation principles for AE start/end date

Imputation of AE start date:

- If the AE start date is entirely missing, it is imputed by the first administration date of the study drug;
- If the AE start date is partially missing, the imputation principles are as follows:


 If the year and month are known and are the same as that of the first administration date, it is imputed by the first medication date;

- o If the year and month are known but are different from that of the first administration date, it is imputed by the 1st day of that month;
- o If only the year is known and is the same as that of the first administration date, it is imputed by the first administration date of the study drug;
- o If only the year is known but is different from that of the first administration date, it is imputed by Jan. 1 of that year.

Imputation principles for AE end date:

- If the year and month are known, it is imputed by the last day of that month;
- If only the year is known, it is imputed by Dec. 31 of that year.
- If all the year, month, and day are missing, the AE end date is imputed by the last administration date of the study drug + 30 days.

In the case of a death, if the AE end date imputed is after the date of death, the date of death is used instead.

## 2.3.5 Other data processing principles

When describing data for routine blood test, if the results are below the lower limit of instrument measurement, then 0 is used for the statistical analysis. For data collected at the same visit, the one from the central laboratory is preferred for analysis. If two or more measurements are performed at the same visit in the central laboratory or study site, the first effective result is used. All measurement results will be tabulated.

## 2.3.6 Data processing principles for unscheduled visits

The measurements of unscheduled visits are included in the baseline (including the baseline of each cycle) summary. In any other phase, unless otherwise stated, only the data from scheduled visits are summarized, and the measurement results from unscheduled visits will be tabulated only and not included in the statistical analysis.

#### 2.4 Multiple Comparison

In this study, no multiple comparison is performed.

#### 2.5 Subgroup Analysis

In this study, no subgroup analysis is performed.


#### 2.6 Combination of Study Sites

This is a multi-center study. Data collected from different study sites are pooled for analysis. Due to the large number of study sites and the small number of subjects per site, the study site is not included as a covariate in any statistical model.

## 3 STATISTICAL ANALYSIS

#### 3.1 Basic Subject Information

#### 3.1.1 Enrollment and study completion

All subjects enrolled are included in the analysis. The statistical analysis of the enrollment and study completion are performed based on the randomized treatment arm.

Information on subject screening, randomization, study completion and withdrawal of each cycle are summarized for the study/each treatment arm, causes of withdrawals are summarized by category, and the number of cases and percentages are calculated respectively. The causes of withdrawals are presented in a table based on the orders in the CRF. All subject dispositions are tabulated for analysis.

Information on subject screening, randomization, and subjects receiving at least one dose of study drug in each study site is summarized.

Statistical analyses on the number of cases and percentages of FAS, PP set A, PP set B, and SS are performed.

#### 3.1.2 Protocol deviation

To determine whether the protocol has been well performed, all subject data on the Case Report Form (CRF) should be reviewed for serious protocol deviations prior to database lock. All possible serious protocol deviations should be reviewed and evaluated by the investigator and sponsor.

This analysis is based on the randomized set. All serious protocol deviations will be summarized by category and will be tabulated for analysis. In the case of a summary description or tabulated analysis of serious protocol deviations, the time of the protocol deviation will be considered (whether occurred in cycle 1).

See the chapter "Definition of Analysis Set" for the definition of serious protocol deviation.

#### 3.1.3 Demographics and baseline characteristics

Descriptive statistics of demographics and baseline characteristics are summarized for FAS, PP set A, and PP set B at baseline.

For baseline demographics, descriptive statistics of quantitative parameters, including age, height, weight, BMI, BSA, and the time (days) from diagnosing breast cancer to signing ICF are summarized by the number of subjects, mean, standard deviation, median, minimum, and maximum in each treatment arm, separately. Descriptive statistics of qualitative parameters, including gender, ethnicity, ECOG performance status, tumor TNM staging, and tumor clinical staging are summarized by the number of subjects and percentage in each treatment arm, separately.


Where:

Age (years) = (Date of signing ICF – Date of birth + 1)/365.25.

BSA =  $0.007184 \times \text{weight (kg)}^{0.425} \times \text{height (cm)}^{0.725}$ 

BMI  $(kg/m^2) = W(kg)/H^2(m)$ , where, the unit of BMI is  $kg/m^2$ ; W means weight (kg); H means height (m).

In addition, the demographics and disease characteristics at baseline will be tabulated.

#### 3.1.4 Medical history, history of breast cancer surgery, and concomitant non-drug treatment

This analysis is based on FAS. Medical history is summarized by prior disease and concomitant disease separately. A prior disease is a disease resolved before the start of the first chemotherapy. A concomitant disease is a disease which occurs after the start of the first chemotherapy or which occurs before the start of the first chemotherapy but continues after the start of the first chemotherapy. A disease should be judged as a prior disease if there are justifiable reasons. Otherwise, it is judged as a concomitant disease. Medical history, history of breast cancer surgery, and concomitant non-drug treatment are coded using Medical Dictionary for Regulatory Activities (MedDRA) 20.1 or the latest version before database locking, and the number of subjects and percentages are summarized by System Organ Class (SOC) and Preferred Term (PT), separately.

Medical history, history of breast cancer surgery, and concomitant non-drug treatment will be tabulated separately.

#### 3.1.5 Prior medications and concomitant medications

This analysis is based on FAS. The World Health Organization Drug Dictionary (WHODD) (Version: Jun. 01, 2017) or the latest version before database locking is used for coding. Combined medications subjects in FAS received are summarized in prior medications and concomitant medications by Anatomical Therapeutic Chemical (ATC) Classification System level 2 (in descending order of overall frequency) and PT (in descending order of overall frequency) separately. In addition, data of the prior medications and concomitant medications will be tabulated separately.

Prior medication is defined as a medication that has already been discontinued before the first chemotherapy. Concomitant medication is defined as a medication other than the study drug and given from the first chemotherapy to day 21 of cycle 4. A medication is considered a prior medication if its end date coincides with the date of the first chemotherapy. If the start date of the combined medication is missing, it will be imputed according to the imputation principles for combined medications specified in 2.3.4 "Missing data processing principles" of this SAP.

The prior medications and concomitant medications will all be tabulated.


#### 3.1.6 Exposure to drugs

This analysis is based on SS. The use of study drugs (F-627 and GRAN®) and adjuvant chemotherapy agents (epirubicin and cyclophosphamide) are described by treatment cycle and the entire treatment period as follows:

## F-627and GRAN®

- Total number of treatment
- Actual total dose
- Actual dose intensity
- Relative dose intensity (%) = (Actual dose intensity/Planned dose intensity) × 100%

## Epirubicin + Cyclophosphamide

- Total days of treatment
- Actual dose intensity
- Actual total dose (mg)
- Relative dose intensity (%) = (Actual dose intensity/Planned dose intensity) × 100%

A description on the relative dose intensity of these drugs will be summarized based on the following criteria: > 110%, > 100-110%, > 90-100%, > 80-90%, > 70-80%, > 60-70%, > 50-60%, and  $\le 50\%$ .

Among which, the actual dose intensity of F-627 (mg/dose) = actual dose/actual number of doses; the actual dose intensity of GRAN® ( $\mu$ g/kg/day) = actual total dose/body weight/days of dosing, and when calculating the actual dose intensity of GRAN®, the subject's body weight is the last effective value measured before the administration of study drugs in each cycle (including the day of administration); the actual dose intensity of chemotherapeutic agents (mg/m²) = actual dose/body surface area (BSA)/actual number of doses. According to the Takahira formula, BSA = 0.007184 × body weight (kg)<sup>0.425</sup> × height (cm)<sup>0.725</sup>. When calculating the actual dose intensity of epirubicin and cyclophosphamide, the subject's body weight and height are the last effective values measured before the start of chemotherapy in each cycle (including the day of chemotherapy).

After the completion of the study, the total dose of each study drug and adjuvant chemotherapy agent will be summarized for the entire study.

All information on study drugs will be tabulated by treatment arm, subject number, treatment stage, date of drug administration, total dose of actual medication, and route of administration, respectively.

Similarly, data of adjuvant chemotherapy agents (epirubicin, cyclophosphamide) will be tabulated and described.


#### 3.2 Efficacy Analysis/Pharmacokinetic Analysis

## 3.2.1 Primary efficacy analysis

## 3.2.1.1 Primary analysis

The primary efficacy endpoint will test the non-inferiority of F-627 to GRAN<sup>®</sup> in terms of the duration (days) of grade 3 neutropenia (including grade 4 or severe neutropenia) in cycle 1.

Primary efficacy analysis will be performed using both PP set A and FAS. Priority is given to the FAS analysis results while PP set A is used for a sensitivity analysis. The hypotheses for non-inferiority between F-627 and GRAN® are as follows:

```
H<sub>0</sub>: \muF-627 (20 mg/dose) -\muGRAN<sup>®</sup> > 1 day; H<sub>1</sub>: \muF-627 (20 mg/dose) -\muGRAN<sup>®</sup> \leq 1 day
```

The non-inferiority margin is specified as 1 day and the test is one-sided with a significance level of  $\alpha$  = 0.025. The difference (F-627–GRAN®) of the primary efficacy endpoint between the two arms and its upper limit of one-sided 97.5% CI will be estimated using the Hodges–Lehmann method. If the upper limit of one-sided 97.5% CI of the inter-arm difference (F-627–GRAN®) in the duration of grade 3 or 4 neutropenia is  $\leq$  1 day, the ineffective hypothesis  $H_0$  will be rejected, and the non-inferiority hypothesis  $H_1$  is established and it can be deemed that F-627 is not inferior to GRAN®.

SAS code analyzed using Hodges–Lehmann is as follows:

proc npar1way hl(refclass=2) alpha=0.05 data=adef1; /\* "refclass=2" means the comparator arm (trtn=2) is used as a reference\*/

```
class trtn;
var aval;
ods select WilcoxonScores HodgesLehmann;
run;
```

#### 3.2.1.2 Sensitivity analysis

In addition to the use of PP set A in the sensitivity analysis of the primary endpoint, analysis on missing ANC data without imputation in the FAS will also be performed to evaluate the robustness of the primary endpoint results.

## 3.2.2 Secondary efficacy analysis

The specific endpoints and methods of secondary efficacy analysis are as follows: The statistical analysis on the secondary efficacy endpoints in cycle 1 is performed using both FAS and PP set A; the statistical analysis on the secondary efficacy endpoints in cycles 2–4 is performed using both FAS and PP set B.


#### 3.2.2.1 Incidence rate of grade 3 or grade 4 neutropenia in each cycle

The incidence rates of grade 3 or 4 neutropenia of F-627 and GRAN® (ANC  $< 1.0 \times 10^9$ /L and ANC  $< 0.5 \times 10^9$ /L, respectively) in cycle 1 are compared using Fisher's exact test. In each cycle, if a subject develops one case of neutropenia, it will be documented once. Incidence rate = Number of subjects with neutropenia/Total number of analyzed subjects.

For cycles 2–4, the analysis is performed using a method similar with that used in cycle 1.

The incidence rates of grade 3 or 4 neutropenia of F-627 and GRAN® in cycles 1–4 are summarized, along with the P values corresponding to the comparison between F-627 and GRAN®.

## 3.2.2.2 Durations (days) of grade 3 or 4 neutropenia in cycles 2-4

The durations (days) of grade 3 or 4 neutropenia of F-627 and GRAN® (ANC  $< 1.0 \times 10^9$ /L and ANC  $< 0.5 \times 10^9$ /L, respectively) in cycles 2–4 are summarized.

Similar as the method used in the primary efficacy analysis, the 95% CI of the mean difference of the durations of grade 3 neutropenia between F-627 and GRAN® in cycles 2–4 is given using the Hodges-Lehmann method.

## 3.2.2.3 Incidence rate and duration (days) of grade 4 neutropenia in each cycle

The incidence rates of grade 4 neutropenia (ANC  $< 0.5 \times 10^9/L$ ) of F-627 and GRAN® are compared using the method similar to that used for the incidence rate of grade 3 or grade 4 neutropenia in 3.2.2.1 and the comparison is summarized.

The durations (days) of grade 4 neutropenia (ANC <  $0.5 \times 10^9$ /L) of F-627 and GRAN® are compared using the method similar to that used for the duration (days) of grade 3 or 4 neutropenia in 3.2.2.2 and the comparison is summarized.

#### 3.2.2.4 Overall duration (days) of grade 3 or 4 neutropenia in overall 4 cycles

The difference of durations between F-627 and GRAN<sup>®</sup> is compared using the method similar to that used for the duration (days) of grade 3 or 4 neutropenia (ANC  $< 1.0 \times 10^9$ /L and  $< 0.5 \times 10^9$ /L, respectively) in 3.2.2.2 and the comparison is summarized.

The overall duration is the sum of the durations (days) of grade 3 or 4 neutropenia in overall 4 cycles.

The overall duration of the 4 cycles = duration (days) of grade 3 or 4 neutropenia in cycle 1 + duration (days) of grade 3 or 4 neutropenia in cycle 2 + duration (days) of grade 3 or 4 neutropenia in cycle 3 + duration (days) of grade 3 or 4 neutropenia in cycle 4.

## 3.2.2.5 Incidence rate and duration (days) of grade 2 or greater neutropenia in each cycle

The incidence rates of grade 2 or greater neutropenia (ANC  $< 1.5 \times 10^9$ /L) of F-627 and GRAN® are compared using the method similar to that used for the incidence rate of grade 3 or grade 4 neutropenia in 3.2.2.1 and the comparison is summarized.


The durations (days) of grade 2 or greater neutropenia (ANC  $< 1.5 \times 10^9/L$ ) of F-627 and GRAN® are compared using the method similar to that used for the duration (days) of grade 3 or 4 neutropenia in 3.2.2.2 and the comparison is summarized.

## 3.2.2.6 Incidence rate of febrile neutropenia (FN)

FN is defined as ANC  $< 1.0 \times 10^9$ /L, and body temperature in a single measurement > 38.3 °C or a fever  $\ge 38.0$  °C lasting for greater than 1 hr.

To calculate the incidence rate, FN which occurs in a subject throughout the study is recorded only once even if it occurs more than one time. Incidence rate = Number of subjects experiencing FN/Total number of analyzed subjects.

The frequency and incidence rate of FN are summarized by different treatment arms and cycles using the method similar to that used for the incidence rate of grade 3 or 4 neutropenia in 3.2.2.1. The differences between F-627 and GRAN® are compared using Fisher's exact test and the comparison is summarized

#### 3.2.2.7 ANC - time profile

The efficacies of F-627 and GRAN® are compared by plotting the ANC-time logarithmic curves of treatment arms in cycle 1 and cycles 2–4.

#### 3.2.2.8 ANC nadir

The ANC nadir on days 3–13 of cycles 1–4 is compared between different treatment arms. The analysis is performed using the same analysis method for the primary efficacy endpoint to calculate 95% CI.

## 3.2.2.9 Time (days) of ANC nadir recovers to $2.0 \times 10^9/L$ in each cycle

The time (days) of ANC recovers to  $2.0 \times 10^9$ /L from nadir in cycles 1–4 is compared between different treatment arms. The analysis is performed using the same analysis method for the primary efficacy endpoint to present 95% CI and is summarized.

If ANC nadir is  $< 2.0 \times 10^9/L$  during the first 13 days of a cycle, the recovery time = the date on which ANC is  $\ge 2.0 \times 10^9/L$  - the date of ANC nadir + 1.

If ANC nadir is  $\ge 2.0 \times 10^9$ /L during the first 13 days of a cycle, the recovery time = 0 day.

## 3.3 Safety Analysis

All safety analyses are based on SS. Parameters for safety analysis include AEs, laboratory measurements, vital signs, electrocardiogram (ECG), and abdominal ultrasound. In safety analysis, the result of the last visit is the measurements obtained at the last scheduled visit (including end of study visit/withdrawal visit) during the study.

#### 3.3.1 Adverse event

AEs are summarized according to MedDRA 20.1 and coded based on the latest version thereof before


#### database locking.

In this study, all SAEs that occur from signing ICF and randomization until 30 days after the last dose of the study drug will be recorded, including AEs that occurred prior to the randomization and worsened during the treatment period, regardless of whether they are collected from the investigator's observation or self-reported by the subject.

A treatment-emergent adverse event (TEAE) is (1) an AE which occurred on or worsened after the first dose of study drug (including chemotherapy) or (2) an AE which occurred before the first dose of study drug (including chemotherapy) but worsened after the first dose of study drug.

Number of TEAE cases refers to the number of subjects experienced TEAE. In statistical summary of TEAE cases, if a subject experienced the same TEAE more than once, he/she is considered to have experienced the TEAE. If a subject experienced more than one TEAE, then the subject will only be included in the most severe TEAE category in statistical analysis.

The number of TEAEs refers to the frequency of the occurrence of TEAE. The number of TEAEs is counted by PT. If two TEAEs occurred in the same subject have the same PT but differ in the time of onset, they are considered as different TEAEs and are counted as 2 events when summarizing the number of TEAE. If two TEAEs occurred in the same subject one after another (the end date of the previous AE is the onset date of the next AE), they are considered as one TEAE with the greatest severity grade and are counted as 1 event when summarizing the number of TEAE.

Firstly, the incidence rates (including number of cases and number of events) of AEs, TEAEs, study drug-related TEAEs, grade 3 or greater (as per NCI CTCAE V4.03) TEAEs, study drug-related grade 3 or greater TEAEs, TEAEs leading to permanent discontinuation, SAEs, and study drug-related SAEs or death throughout the treatment will be summarized by treatment arms, respectively.

Secondly, the incidence rate (number of cases) of the following AEs occurring in each treatment arm throughout the treatment will be described by SOC and PT:

- TEAEs
- Study drug-related TEAEs
- Grade 3 or greater TEAEs
- Study drug-related grade 3 or greater TEAEs
- TEAEs graded as per NCI CTCAE V4.03
- Study drug-related TEAEs graded as per NCI CTCAE V4.03
- TEAEs leading to permanent discontinuation
- SAEs
- Study drug-related SAEs


Deaths

• TEAEs with an incidence rate of > 5%

All AEs as well as study drug-related TEAEs and SAEs are tabulated.

#### 3.3.2 Laboratory measurements

For data collected at the same visit, the one from the central laboratory is preferred for analysis. The missing ANC data will not be imputed for the safety analysis. Laboratory measurements include:

- Routine blood test: complete blood count, including red blood cells (RBCs), hemoglobin, white blood cells (WBCs), platelet count, neutrophils, lymphocytes, monocytes, basophils, eosinophils, hematocrit, mean corpuscular volume, mean corpuscular hemoglobin concentration, mean corpuscular hemoglobin, etc.;
- Clinical chemistry: total protein, albumin, blood glucose, blood urea nitrogen, creatinine, alkaline phosphatase (ALP), lactate dehydrogenase, total bilirubin, aspartate transaminase (AST), γ-glutamyl transpeptidase, alanine transaminase (ALT), Ca, P, K, Na, etc.;
- Urine analysis (urinalysis): pH, urine specific gravity, urine protein, cast, hemocytes, urine WBCs (qualitative), urine glucose, urine ketones, urine RBCs (microscopy), urine WBCs (microscopy), etc.;
- Serum pregnancy test: for any female subject of child-bearing potential, including those who have had tubal ligation.

The laboratory measurements results in routine blood test and the quantitative parameters of clinical chemistry and urinalysis (urine specific gravity and pH) at baseline and at post-baseline time points will be descriptively analyzed by treatment arms, and the changes from baseline in laboratory measurements at post-baseline time points will be given (for routine blood test, the changes from baseline to post-baseline time points in each cycle will be calculated).

Note: Urea in clinical chemistry is counted as blood urea nitrogen, and the data measured and unit are converted according to "blood urea nitrogen = urea". Descriptive statistics of the urine RBCs (microscopy) and urine WBCs (microscopy) in urinalysis will not be summarized and will be tabulated only.

All laboratory measurements made on day 1 of cycle 1 will be included in baseline summary according to the baseline definition and will not be summarized separately.

Routine blood tests made on day 1 of each cycle will be included in the baseline of that cycle according to the baseline definition in each cycle and will not be summarized separately. Other laboratory measurements (including clinical chemistry and urinalysis) made on day 1 of cycles 2–4 will be summarized by the scheduled visits according to the definition of analysis window period.


Based on the normal ranges provided by the central laboratory, results of laboratory measurement (quantitative parameters of routine blood test, clinical chemistry, and urinalysis [urine specific gravity and pH]) are classified as low (below the lower limit of normal range), normal (within the normal range), and high (above the upper limit of normal range). The test results of urinalysis qualitative parameters at baseline and at post-baseline time points will be classified and summarized. The clinical evaluation results of urinalysis parameters at baseline and at post-baseline time points will be classified and summarized.

Data showing "negative" or "positive" in urinalysis are directly classified while other non-quantitative data are classified according to the following principles:

- (1) Qualitative parameters are classified as "positive" if they are: "normal (Chinese version source: 正常)", "NORMAL", "normal (Chinese version source: normal)", "NORMAL", "-", or "Neg".
- Qualitative parameters are classified as "positive" if they are: "+", "++", "+++", "++++", "++++", "++++", "1+", "2+", "3+", "4+", "trace", "±", "weakly positive", "positive 1+", "positive 2+", "positive (1+)", "positive (1+)", "positive (2+)", or "positive (3+)".
- Quantitative analysis will be performed on pH and urine specific gravity. If there are uncertain descriptions such as ">", "<", "greater than", or "less than", the upper or lower limit of the result will be used for the analysis. For example, if the result is "≤ 5.0" or "≥ 5.0", then 5.0 will be used for the analysis.

All laboratory measurement results will be tabulated.

#### 3.3.3 Vital signs, physical examination, ECG, and abdominal ultrasound

The results of vital signs, physical examination, ECG, and abdominal ultrasound performed on day 1 of cycle 1 will be included in the baseline and will not be summarized separately, while those from other visits will be summarized as scheduled visits.

## 3.3.3.1 Vital signs

Vital signs include blood pressure, body temperature, heart rate, and weight. Parameters of vital signs measured at baseline and at post-baseline time points (day 1 of cycles 1–4) will be descriptively analyzed by treatment arms, respectively, and changes from baseline of each parameter at post-baseline time points will be given. The number of cases, mean, standard deviation, median, maximum, and minimum will be calculated. Results of vital signs will be tabulated.


#### 3.3.3.2 Physical examination

Physical examinations include lymph nodes, neck, ears, nose, eyes, throat, cardiovascular system, skin and mucous membranes, limbs, nervous system, musculoskeletal system, etc. Results of physical examinations (normal, abnormal without clinical significance, abnormal with clinical significance, and not tested) at baseline and at post-baseline time points (day 1 of cycles 1–4) will be summarized and described by treatment arms, and the shift change table from baseline to each visit will be given. The abnormalities will be tabulated.

#### 3.3.3.3 Electrocardiogram (ECG)

ECG examination parameters include PR interval, QRS interval, RR interval, QT interval, QTc, and heart rate. PQ interval will not be summarized separately. If both PR interval and PQ interval data are available in the same visit, the data of PR interval will be used for analysis. If only the data of PQ interval are available, it will be used as the data of PR interval. The ECG results during visits will be summarized by treatment arms. The number of cases, mean, standard deviation, median, maximum, and minimum will be quantitatively calculated. According to the clinical evaluation results (normal, abnormal without clinical significance, and abnormal with clinical significance), the number and percentage of subjects will be summarized by the category of ECG results, and the shift change table from baseline to each visit will be given. The number and percentage of subjects with QTc > 450 msec, > 480 msec, and > 500 msec will be summarized, and the number and percentage of subjects with QTc > 30 msec, > 60 msec, and > 90 msec in the changes from baseline will be summarized. Results of all ECG parameters will be tabulated.

#### 3.3.3.4 Abdominal ultrasound

Results of abdominal ultrasound (normal, abnormal without clinical significance, and abnormal with clinical significance) at baseline and at post-baseline time points (day 1 of cycles 1–4) will be summarized and described by treatment arms, and the shift change table from baseline to each visit will be given. All abdominal ultrasound results will be tabulated.

#### 3.3.4 Other safety analysis

Pregnancy test results will be tabulated only.

#### 3.4 Exploratory Analysis of F-627 Immunogenicity

The serum samples for immunogenicity assay will only be collected from the F-627 arm. Information on the distribution of F-627 serum antibody results in immunogenicity analysis set at baseline and at post-baseline time points will be summarized and described. Blood samples are collected on day 1 ( $\pm$  1 day) of each cycle, on day 21 ( $\pm$  1 day) of cycle 4, and 90 days ( $\pm$  7 days) after the last visit (day 21 of cycle 4) to test the serum anti-F-627 antibodies. Results of the test on day 1 of cycle 1 are used as the baseline data.

The results of serum antibody assay will be tabulated.


#### 3.5 Interim Analysis

Not applicable.

## 4 MODIFICATIONS TO THE ORIGINAL ANALYSIS PLAN

The ITT set is changed to FAS based on the statistical analysis guideline.

FAS refers to all randomized subjects who have received the study drug and underwent at least one post-baseline efficacy evaluation. The FAS is primarily used for efficacy evaluation.

The definition of the ITT set is modified to all randomized set.

#### 5 REFERENCES

- The European Agency for the Evaluation of Medicinal Products (EMEA), Committee for Proprietary Medicinal Products (CPMP), ICH E9, Statistical Principles for Clinical Trials, CPMP/ICH/363/96
- Food and Drug Administration (FDA), Center for Drug Evaluation and Research (CDER), Center for Biologics Evaluation and Research (CBER), Guidance for Industry Clinical Trail Endpoints for the Approval of Cancer Drugs and Biologics, May 2007
- 3. F. A. Holmes, S. E. Jones, J. O'Shaughnessy et al. Comparable efficacy and safety profiles of once-per-cycle pegfilgrastim and daily injection filgrastim in chemotherapy-induced neutropenia: a multicenter dose-finding study in women with breast cancer. Ann Oncol. 2002; 13: 903-9.
- 4. F.A. Homes, J.A. O'Shaughnessy, S. Vukelija, et al. Blinded, Randomized, Multicenter Study to Evaluate Single Administration Pefilgrastim Once per Cycle Versus Daily Filgrastim as an Adjunct to Chemotherapy in Patients with High-Risk Stage II or Stage III/IV Breast Cancer. J Clin Oncol 2002; 20: 727-731.
- M. D. Green, H. Koelbl, J. Baselga et al. A randomized double-blind multicenter phase III study of fixed-dose single-administration pegfilgrastim versus daily filgrastim in patients receiving myelosuppressive chemotherapy. Annals of Oncology 2003; 14: 29-35.


## **Appendix 1 SAS Procedures for Imputation of Monotone Missing ANC Data**

```
*Step 1: To impute the missing data at time point 1 (day 3 of cycle 1), model estimation based on
available data at time point 1 is performed. Covariates used include age, arm, chemotherapy, and
existing ANC data;
proc mi data= anc mono out= anc mono1 nimpute=1 seed=2334764;
class prchemo trt;
by Imputation;
var age prchemo trt baseline anc1;
monotone reg(anc1= age prchemo trt ANC);
run;
*Step 2: To impute the missing data at time point 2 (day 5 of cycle 1), model estimation based on
available data at time point 2 and the data imputed at time point 1 is performed. The covariates used are
the same as those used in step 1 (including the ANC data imputed in step 1);
proc sort data= anc mono1;
by _Imputation_;
run;
proc mi data= anc mono1out= anc mono2 nimpute=1 seed=53674345;
by Imputation;
class prchemo trt;
var age prchemo trt baseline anc1 anc2;
monotone reg(anc2= age prchemo trt ANC anc1);
run;
/*The above steps are repeated for each scheduled visit until day 13 of cycle 1*/
```


| Sponsor: | Protocol Number : | Version, date : |
|-------------------------------------|-------------------|-----------------|
| Generon (Shanghai) Corporation Ltd. | SP11631 | 1.0, 2020-03-11 |

# **Table Listing Figures Shells for Statistical Analyses**

A Phase III Randomized, Multi-Centre, Open-Label, Active-Controlled Clinical Trial to Compare the Efficacy and Safety of Recombinant Human Granulocyte Colony Stimulating Factor—Fc Fusion Protein (F-627) and Recombinant Human Granulocyte Colony Stimulating Factor (GRAN®) in the Prophylactic Treatment for Chemotherapy-Induced Neutropenia

**Protocol Number:** SP11631

**Sponsor:** Generon (Shanghai) Corporation Ltd.

Fountain (Beijing) Medical Technology

CRO:

Development CO., Ltd

Version: 1.0

**Date:** 2020-03-11

|-------------------------------------|-------------------|-----------------|
| Generon (Shanghai) Corporation Ltd. | SP11631 | 1.0, 2020-03-11 |

# **Contents**

| Table 14.1.1.1 Subject Disposition – All subjects | 7 |
|---|---|
| Table 14.1.1.2 Subject Disposition by Site – All subjects | 9 |
| Table 14.1.2 Analysis Sets – Randomized Subjects | 10 |
| Table 14.1.3.1 Major Protocol Deviations during the All Treatment Periods – Randomized Subjects | 11 |
| Table 14.1.3.2 Major Protocol Deviations for Cycle 1 – Randomized Subjects | 12 |
| Γable 14.2.1 Demographics and Baseline Characteristics – FAS | |
| Table 14.2.2.1 Demographics and Baseline Characteristics – PP Analysis Set A | 15 |
| Table 14.2.2.2 Demographics and Baseline Characteristics – PP Analysis Set B. | 15 |
| Γable 14.2.3 Baseline Characteristics of the Disease – FAS | 16 |
| Table 14.2.4.1 Baseline Characteristics of the Disease – PP Analysis Set A. | 19 |
| Table 14.2.4.2 Baseline Characteristics of the Disease – PP Analysis Set B | 19 |
| Table 14.2.5 Medical History, Symptoms and Surgical History – FAS | 20 |
| Table 14.2.6 Concomitant Diseases and Symptoms - FAS | |
| Table 14.2.7 Surgical History of Breast Cancer – FAS | 21 |
| Table 14.2.8 Prior Medications – FAS | 22 |
| Table 14.2.9.1 Concomitant Medications – FAS. | 23 |
| Γable 14.2.9.2 Concomitant Non-Drug Treatments – FAS | 23 |
| Table 14.2.10 Extent of Exposure to Study Medication(F-627, GRAN®)–Safety Analysis Set | 24 |
| Table 14.2.11 Extent of Exposure to Chemotherapy drugs(Epirubicin, Cyclophosphamide) -Safety Analysis Set | 26 |
| Table 14.3.1.1 Duration of Grade 3 or 4 Neutropenia during Cycle 1 – FAS | |
| Table 14.3.1.2 Duration of Grade 3 or 4 Neutropenia during Cycle 1 – PP Analysis Set A | 28 |
| Table 14.3.1.3 Duration of Grade 3 or 4 Neutropenia during Cycle 1 – FAS. | 28 |
| Table 14.3.1.4 Sensitivity Analysis for Duration of Grade 3 or 4 Neutropenia during Cycle 1 | 29 |
| Table 14.3.2.1 The Incidence of Grade 3 or 4 Neutropenia for Cycle 1 – FAS | 30 |
| Table 14.3.2.2 The Incidence of Grade 3 or 4 Neutropenia for Cycle 1 – PP Analysis Set A | 31 |
| Table 14.3.2.3 The Incidence of Grade 3 or 4 Neutropenia for Cycle 2-4 and All Treatment Periods – FAS | 32 |
| Table 14.3.2.4 The Incidence of Grade 3 or 4 Neutropenia for Cycle 2-4 and All Treatment Periods – PP Analysis Set B | 33 |
| Table 14.3.3.1 Duration of Grade 3 or 4 Neutropenia for Cycle 2-4 and All Treatment Periods – FAS | 34 |
| Table 14.3.3.2 Duration of Grade 3 or 4 Neutropenia during Cycle 2-4 and All Treatment Periods – PP Analysis Set B | |
| Table 14.3.4.1 Duration of Grade 4 Neutropenia during Cycle 1 – FAS | |
| Table 14.3.4.2 Duration of Grade 4 Neutropenia during Cycle 1 – PP Analysis Set A | 37 |

Sponsor:
Generon (Shanghai) Corporation Ltd.

Protocol Number:
SP11631

Version, date:
1.0, 2020-03-11

| Table 14.3.4.3 | Duration of Grade 4 Neutropenia during Cycle 2-4 and All Treatment Periods – FAS. | 37 |
|---|---|---|
| Table 14.3.4.4 | Duration of Grade 4 Neutropenia during Cycle 2-4 and All Treatment Periods – PP Analysis Set B | 37 |
| Table 14.3.4.5 | The Incidence of Grade 4 Neutropenia for Cycle 1 – FAS | 38 |
| Table 14.3.4.6 | The Incidence of Grade 4 Neutropenia for Cycle 1 – PP Analysis Set A | 38 |
| Table 14.3.4.7 | The Incidence of Grade 4 Neutropenia for Cycle 2-4 and All Treatment Periods – FAS | 38 |
| Table 14.3.4.8 | The Incidence of Grade 4 Neutropenia for Cycle 2-4 and All Treatment Periods – PP Analysis Set B | 38 |
| Table 14.3.5.1 | The total Duration of Grade 3 or 4 Neutropenia during 4 Cycles – FAS | 40 |
| Table 14.3.5.2 | The total Duration of Grade 3 or 4 Neutropenia during 4 Cycles – PP Analysis Set B | 40 |
| | Duration of Grade 2 or Higher Neutropenia during Cycle 1 – FAS. | |
| Table 14.3.6.2 | Duration of Grade 2 or Higher Neutropenia during Cycle 1 – PP Analysis Set A | 41 |
| Table 14.3.6.3 | Duration of Grade 2 or Higher Neutropenia during Cycle 2-4 and All Treatment Periods – FAS | 41 |
| Table 14.3.6.4 | Duration of Grade 2 or Higher Neutropenia during Cycle 2-4 and All Treatment Periods – PP Analysis Set B | 41 |
| Table 14.3.6.5 | The Incidence of Grade 2 or Higher Neutropenia for Cycle 1 – FAS | 42 |
| Table 14.3.6.6 | The Incidence of Grade 2 or Higher Neutropenia for Cycle 1 – PP Analysis Set A | 42 |
| Table 14.3.6.7 | The Incidence of Grade 2 or Higher Neutropenia for Cycle 2-4 and All Treatment Periods – FAS | 42 |
| Table 14.3.6.8 | The Incidence of Grade 2 or Higher Neutropenia for Cycle 2-4 and All Treatment Periods – PP Analysis Set B | 42 |
| Table 14.3.7.1 | The Incidence of Febrile Neutropenia (FN) for Cycle 1 – FAS | <b>4</b> 4 |
| | The Incidence of Febrile Neutropenia (FN) for Cycle 1 – PP Analysis Set A | |
| Table 14.3.7.3 | The Incidence of Febrile Neutropenia (FN) for Cycle 2-4 and All Treatment Periods – FAS | 44 |
| | The Incidence of Febrile Neutropenia (FN) for Cycle 2-4 and All Treatment Periods – PP Analysis Set B | |
| | ANC nadir from day 3 to day 13 for Cycle 1 – FAS | |
| | ANC nadir from day 3 to day 13 for Cycle 1 – PP Analysis Set A | |
| | ANC nadir from day 3 to day 13 within a cycle for Cycle 2-4 – FAS | |
| | ANC nadir from day 3 to day 13 within a cycle for Cycle 2-4 – PP Analysis Set B | |
| | Time in days to ANC Recovery Post Nadir for Cycle 1– FAS | |
| | Time in days to ANC Recovery Post Nadir for Cycle 1 – PP Analysis Set A | |
| | Time in days to ANC Recovery Post Nadir for Cycle 2-4 and All Treatment Periods– FAS | |
| | Time in days to ANC Recovery Post Nadir for Cycle 2-4 and All Treatment Periods – PP Analysis Set B | |
| | mmunogenicity Results of F-627- Immunogenicity Analysis Set | |
| | Adverse Events – Safety Analysis Set | |
| | Adverse Events by Causality with study drug – Safety Analysis Set | |
| Table 14.5.1.3 | TEAEs by System Organ Class and Preferred Term – Safety Analysis Set | 53 |
| Table 14.5.1.4 | Study Drug Related TEAEs by System Organ Class and Preferred Term - Safety Analysis Set | 54 |

Sponsor:
Generon (Shanghai) Corporation Ltd.

Protocol Number:
SP11631

Version, date:
1.0, 2020-03-11

| Table 14.5.1.5 TEAEs with CTCAE Grade 3 or Higher by System Organ Class and Preferred Term - Safety Analysis Set | 54 |
|---|---|
| Table 14.5.1.6 Study Drug Related TEAEs with CTCAE Grade 3 or Higher by System Organ Class and Preferred Term - Safety | |
| Analysis Set | 54 |
| Table 14.5.1.7 TEAEs by System Organ Class and Preferred Term and NCI CTCAE V4.03 Grade - Safety Analysis Set | 55 |
| Table 14.5.1.8 Study Drug Related TEAEs by System Organ Class and Preferred Term and NCI CTCAE V4.03 Grade - Safety Ana | |
| Set | - |
| Table 14.5.1.9 TEAEs leading to Study Drug Withdrawn by System Organ Class and Preferred Term - Safety Analysis Set | 57 |
| Table 14.5.1.10 SAE by System Organ Class and Preferred Term - Safety Analysis Set | |
| Table 14.5.1.11 Death by System Organ Class and Preferred Term - Safety Analysis Set | 58 |
| Table 14.5.1.12 TEAEs with Incidence > 5% by System Organ Class and Preferred Term - Safety Analysis Set | 58 |
| Table 14.5.2.1.1 Summary of Hematology Results- Safety Analysis Set. | |
| Table 14.5.2.1.2 Category of Hematology Results by Baseline and Post-Baseline Visit by Cycle – Safety Analysis Set | 60 |
| Table 14.5.2.2.1 Summary of Clinical Chemistry Results – Safety Analysis Set | 61 |
| Table 14.5.2.2.2 Category of Clinical Chemistry Results by Baseline and Post-Baseline Visit – Safety Analysis Set | 61 |
| Table 14.5.2.3.1 Summary of Urinalysis Quantitative Parameters – Safety Analysis Set | |
| Table 14.5.2.3.2 Category of Urinalysis Quantitative Parameters Results by Baseline and Post-Baseline Visit – Safety Analysis Set | 61 |
| Table 14.5.2.3.3 Category of Urinalysis Qualitative Parameters Results by Baseline and Post-Baseline Visit – Safety Analysis Set | |
| Table 14.5.2.3.4 Summary of Urinalysis Clinical Evaluation by Baseline and Post-Baseline Visit – Safety Analysis Set | |
| Table 14.5.3.1 Vital Signs and Weight – Safety Analysis Set. | |
| Table 14.5.3.2 Body Temperature Results – Safety Analysis Set | 66 |
| Table 14.5.3.3.1 Physical Examination – Safety Analysis Set | 67 |
| Table 14.5.3.3.2 Shift Change of Physical Examination from Baseline to Post-Baseline – Safety Analysis Set | |
| Table 14.5.4.1 12-Lead ECG – Safety Analysis Set | |
| Table 14.5.4.2 12-Lead ECG Results in Clinical Evaluation—Safety Analysis Set | 70 |
| Table 14.5.4.3 Shift Change of 12-Lead ECG Results in Clinical Evaluation from Baseline to Post-Baseline – Safety Analysis Set | 71 |
| Table 14.5.4.4 QTc ECG Results – Safety Analysis Set | |
| Table 14.5.5.1 Results of Abdominal Ultrasound - Safety Analysis Set | 73 |
| Table 14.5.5.2 Shift Change of Abdominal Ultrasound from Baseline to Post-Baseline - Safety Analysis Set | |
| Listing 16.1.7.1 Enrollment Information and Randomization – All Subjects | |
| Listing 16.2.1.1 Disposition of Subjects –Randomized Subjects | |
| Listing 16.2.1.2 Withdrawal from Study–Randomized Subjects | 77 |
| Listing 16.2.1.3.1 Analysis Sets– Randomized Subjects | 78 |
| Listing 16.2.1.3.2 Reasons for Subjects Excluded from FAS/SS/PP Set – Randomized Subjects | 78 |

Sponsor:
Generon (Shanghai) Corporation Ltd.

Protocol Number:
SP11631

Version, date:
1.0, 2020-03-11

| Listing 1 | 16.2.1.4 Major Protocol Deviations- Randomized Subjects | . 79 |
|---|---|---|
| Listing : | 16.2.1.5 Protocol Deviations– Randomized Subjects. | . 80 |
| Listing 1 | 16.2.2.1 Demographics – FAS | . 81 |
| | 16.2.2.2 Disease Diagnosis, Chemotherapy History, Physical Status – FAS | |
| | 16.2.2.3 History of Surgery–FAS | |
| Listing : | 16.2.2.4 Prior / Concomitant Disease – FAS | . 84 |
| Listing 1 | 16.2.2.5 Cardiac Doppler Ultrasound– FAS. | . 85 |
| Listing 1 | 16.2.2.6 Chest (Lateral) Examination— FAS | . 86 |
| Listing 1 | 16.2.2.7 Concomitant medications – FAS | . 87 |
| Listing 1 | 16.2.2.8 Concomitant Non-Drug Treatments – FAS | . 88 |
| Listing 1 | 16.2.2.9 Data of Efficacy Endpoints – FAS | . 89 |
| Listing 1 | 16.2.3.1 Immunogenicity test of F-627 - Immunogenicity Analysis Set | . 90 |
| Listing 1 | 16.2.4.1.1 Exposure of Study Drug (F-627, GRAN®) for Cycle 1 – Safety Analysis Set | . 91 |
| Listing 1 | 16.2.4.1.2 Exposure of Study Drug (F-627, GRAN®) for All Treatment Periods – Safety Analysis Set | . 92 |
| Listing 1 | 16.2.4.1.3 Overdose of Study Drug (F-627, GRAN®) for All Treatment Periods – Safety Analysis Set | . 93 |
| Listing 1 | 16.2.4.1.4 Exposure of Chemotherapy drugs (Epirubicin, Cyclophosphamide) for Cycle 1– Safety Analysis Set | . 94 |
| | 16.2.4.1.5 Exposure of Chemotherapy drugs (Epirubicin, Cyclophosphamide) for All Treatment Periods – Safety Analysis Set | |
| Listing [ | 16.2.4.2.1 Adverse Event – Safety Analysis Set | . 95 |
| Listing 1 | 16.2.4.2.2 TEAE Related to Study Drug – Safety Analysis Set | . 96 |
| Listing [ | 16.2.4.2.3 Serious Adverse Event – Safety Analysis Set | . 96 |
| Listing [ | 16.2.4.2.4 Adverse Event leading to Study Drug Withdrawn – Safety Analysis Set | . 96 |
| | 16.2.4.3.1 Hematology - Safety Analysis Set | |
| Listing [ | 16.2.4.3.2 Clinical Chemistry - Safety Analysis Set | . 98 |
| Listing [ | 16.2.4.3.3 Urinalysis - Safety Analysis Set | . 99 |
| Listing [ | 16.2.4.3.4 Pregnancy Test - Safety Analysis Set | 01 |
| Listing [ | 16.2.4.4.1 Vital Signs - Safety Analysis Set. | 102 |
| Listing [ | 16.2.4.4.2 Body Temperature- Safety Analysis Set | 103 |
| Listing | 16.2.4.4.3 Physical Examination – Safety Analysis Set. | 104 |
| Listing | 16.2.4.5.1 12-Lead ECG - Safety Analysis Set | 105 |
| | 16.2.4.5.2 Abdominal Ultrasound - Safety Analysis Set | |
| | 4.1.1.1 Changes of ANC Mean (log-transformed) by Time during Cycle 1 – FAS | |
| Figure 1 | 4.1.1.2 Changes of ANC Mean (log-transformed) by Time during Cycle 1 – PP Analysis Set A | 108 |
| Figure 1 | 4 1 1 3 Changes of ANC Median (log-transformed) by Time during Cycle 1 – FAS | 108 |

| Sponsor :<br>Generon (Shanghai) Corporation Ltd. | Protocol Number :<br>SP11631 | Version, date : 1.0, 2020-03-11 | |
|---|---|---|---|
| Figure 14.1.1.4 Changes of ANC Median (lo | g-transformed) by Time during Cycle 1 – PP A | nalysis Set A | 108 |
| Figure 14.1.2.1 Changes of ANC Mean (log- | transformed) by Time during Cycle 2 – FAS | · | 108 |
| Figure 14.1.2.2 Changes of ANC Mean (log- | transformed) by Time during Cycle 2 -PP Ana | ysis Set B | 108 |
| Figure 14.1.2.3 Changes of ANC Median (lo | g-transformed) by Time during Cycle 2 – FAS | | 108 |
| Figure 14.1.2.4 Changes of ANC Median (lo | g-transformed) by Time during Cycle 2 – PP A | nalysis Set B | 108 |
| Figure 14.1.3.1 Changes of ANC Mean (log- | transformed) by Time during Cycle 3 – FAS | | 108 |
| Figure 14.1.3.2 Changes of ANC Mean (log- | transformed) by Time during Cycle 3 – PP Ana | lysis Set B | 108 |
| Figure 14.1.3.3 Changes of ANC Median (lo | g-transformed) by Time during Cycle 3 – FAS | | 108 |

|-------------------------------------|-------------------|-----------------|
| Generon (Shanghai) Corporation Ltd. | SP11631 | 1.0, 2020-03-11 |

**Table 14.1.1.1 Subject Disposition – All subjects** 

| | F-627<br>n (%) | GRAN®<br>n (%) | Total n (%) |
|---|---|---|---|
| All Screened Subjects | | | XX |
| Screening failure | | | XX |
| Randomized | XX | XX | XX |
| Received study drug at least once | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not receive study drug after random and withdrawal | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Complete the cycle 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Withdrawal in cycle 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Complete the cycle 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Withdrawal in cycle 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Complete the cycle 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Withdrawal in cycle 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Complete the cycle 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Withdrawal in cycle 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Complete the study | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Withdraw from the study | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| The reasons for withdrawal | , , | | , , |
| Screening failure | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subject withdraws voluntarily | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Occurrence of uncontrolled grade 3 or 4 adverse events related to the study drug as judged by the investigator | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subject fails to comply with the study protocol | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Termination by the investigator under safety considerations or in the best interest of the subject when the subject's condition changes | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Pregnancy | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Lost to follow-up | xx (xx.x) | xx (xx.x) | xx (xx.x) |

|---|---|---|---|
| Death | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Data Source: Data Listing 16.x.x.x

Note: Percentages are based on the number of randomized subjects in each treatment group.

| Sponsor :<br>Generon (Shanghai) Corporation Ltd. | Protocol Number :<br>SP11631 | Version, date: 1.0, 2020-03-11 |
|---|---|---|

Table 14.1.1.2 Subject Disposition by Site – All subjects

| | ibject Disposition by Site | in subjects | | |
|---|---|---|---|---|
| | Screening | Screening failure | | Receivd study drug at least once |
| Study site | | | Randomized | n (%) |
| 01 | XX | XX | XX | xx (xx.x) |
| 02 | XX | XX | XX | xx (xx.x) |
| 03 | XX | XX | XX | xx (xx.x) |
| | XX | XX | XX | xx (xx.x) |
| | XX | XX | XX | xx (xx.x) |
| | XX | XX | XX | xx (xx.x) |

Data Source: Data Listing 16.x.x.x

Note: Percentages are based on the number of randomized subjects at each site.
|---|---|---|
|---|---|---|

Table 14.1.2 Analysis Sets – Randomized Subjects

| F-627 | CDANE | |
|---|---|---|
| 1 -02/ | $GRAN^{@}$ | Total |
| (N=xx) | (N=xx) | (N=xx) |
| n(%) | n(%) | n(%) |
| xx (xx.x) | xx (xx.x) | xx (xx.x) |
| xx (xx.x) | xx (xx.x) | xx (xx.x) |
| xx (xx.x) | xx (xx.x) | xx (xx.x) |
| xx (xx.x) | xx (xx.x) | xx (xx.x) |
| xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | (N=xx)<br>n(%)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | (N=xx) (N=xx) n(%) n(%) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) |

Data Source: Data Listing 16.x.x.x

Note: N= Number of randomized subjects in each treatment group

Percentages are based on the number of randomized subjects in each treatment group.

- [1] Safety Analysis Set (SS): All subjects randomized who received at least one study drug will be included in the safety analysis set.
- [2] Full Analysis Set (FAS): All subjects randomized who received at least one study drug and had at least one post-baseline effective assessment will be included in the full analysis set
- [3] Per-Protocol (PP) Analysis Set A: All subjects from the Full Analysis Set without major protocol deviations, severe medication non-compliance, lost to follow-up or withdrawal in the cycle 1 will be included in the PP Analysis Set A.
- [4] Per-Protocol (PP) Analysis Set B: All subjects from the Full Analysis Set without major protocol deviations, severe medication non-compliance, lost to follow-up or withdrawal in all cycles will be included in the PP Analysis Set B.
- [5] Immunogenicity analysis set (IMAS) is defined as all subjects who receive at least one dose of F627 and have at least one result of serum anti-F-627 antibody collected after treatment of F-627.

|---|---|---|
| Generon (Ghanghar) Corporation Eta. | 5111051 | 1.0, 2020-03-11 |

Table 14.1.3.1 Major Protocol Deviations during the All Treatment Periods – Randomized Subjects

| <u>-</u> | F-627 | GRAN® | Total |
|---------------------------------------|-----------|-----------|-----------|
| | (N=xx) | (N=xx) | (N=xx) |
| | n(%) | n(%) | n(%) |
| At least one major protocol deviation | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| < major protocol deviations #1> | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| < major protocol deviations #2> | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| < major protocol deviations #3> | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Data Source: Data Listing 16.x.x.x

Note: N= Number of randomized subjects in each treatment group

Percentages are based on the number of randomized subjects in each treatment group.

|---|---|---|
| Generon (Ghanghar) Corporation Eta. | 5111051 | 1.0, 2020-03-11 |

Table 14.1.3.2 Major Protocol Deviations for Cycle 1 – Randomized Subjects

| | F-627 | GRAN® | Total |
|---------------------------------------|-----------|-----------|-----------|
| | (N=xx) | (N=xx) | (N=xx) |
| | n(%) | n(%) | n(%) |
| At least one major protocol deviation | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| < major protocol deviations #1> | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| < major protocol deviations #2> | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| < major protocol deviations #3> | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Data Source: Data Listing 16.x.x.x

Note: N= Number of randomized subjects in each treatment group

Percentages are based on the number of randomized subjects in each treatment group.

| Sponsor : Protocol Number : SP11631 | Version, date: 1.0, 2020-03-11 |
|-------------------------------------|--------------------------------|
|-------------------------------------|--------------------------------|

Table 14.2.1 Demographics and Baseline Characteristics – FAS

| Parameter | F-627 | $GRAN^{\circledR}$ | Total |
|---|---|---|---|
| Category/Statistics | (N=xx) | (N=xx) | (N=xx) |
| Age(years) | | | \ |
| n(missing) | xx(xx) | xx(xx) | xx(xx) |
| Mean (SD) | xx.x(xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | xx.x | xx.x |
| Min , Max | xx, xx | XX, XX | XX, XX |
| Sex, n (%) | | | |
| Female | xx (100) | xx (100) | xx (100) |
| missing | XX | XX | XX |
| Nation, n (%) | | | |
| n | XX | XX | XX |
| Han Chinese | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Others | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| missing | xx | XX | XX |
| Height (cm) | | | |
| n(missing) | xx(xx) | xx(xx) | xx(xx) |
| Mean (SD) | xx.x(xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Min , Max | xx, xx | XX, XX | XX, XX |
| Weight (kg) | | | |
| n(missing) | xx(xx) | xx(xx) | xx(xx) |
| Mean (SD) | xx.x(xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Min , Max | xx, xx | XX, XX | XX, XX |
| BMI(kg/m <sup>2</sup> ) | | | |
| n(missing) | xx(xx) | xx(xx) | xx(xx) |
| Mean (SD) | xx.x(xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |

|---|---|---|---|
| Median | XX.X | XX.X | XX.X |
| Min , Max | XX, XX | XX, XX | XX, XX |
| BSA(m <sup>2</sup> ) | | | |
| n(missing) | xx(xx) | xx(xx) | xx(xx) |
| Mean (SD) | xx.x(xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | xx.x | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx |

Data Source: Data Listing 16.x.x.x

Note: Percentages are based on the number of subjects with non-missing values from Full Analysis Set in each treatment group.

Programming note: For categorical variable, the row for missing will not be displayed when the count of missing equals to 0.

|---|---|---|

Similar tables as Table 14.2.1:

## Table 14.2.2.1 Demographics and Baseline Characteristics – PP Analysis Set A

Data Source: Data Listing 16.x.x.x

Note: Percentages are based on the number of subjects with non-missing values from PP Analysis Set A in each treatment group.

# Table 14.2.2.2 Demographics and Baseline Characteristics – PP Analysis Set B

Data Source: Data Listing 16.x.x.x

Note: Percentages are based on the number of subjects with non-missing values from PP Analysis Set B in each treatment group.

| Construction of the construction of the constr | Desta ed Navak en e | Warrian data |
|---|---|---|

# Table 14.2.3 Baseline Characteristics of the Disease – FAS

| Parameter | F-627 | $GRAN^{\circledR}$ | Total |
|---|---|---|---|
| Category/Statistics | (N=xx) | (N=xx) | (N=xx) |
| Diagnosed with breast cancer, n (%) | | | (2.1.113) |
| n | XX | xx | XX |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| missing | XX | xx | xx |
| The time from the date of diagnosis as breast cancer to date of Informed Consent [1] | | | |
| n(missing) | xx(xx) | xx(xx) | xx(xx) |
| Mean (SD) | xx.x(xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | XX.X |
| Min , Max | XX, XX | XX, XX | xx, xx |
| Diagnosed by histopathology, n (%) | | | |
| n | XX | XX | XX |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| missing | XX | XX | XX |
| Fumor stage, n (%) | | | |
| n | XX | XX | XX |
| (T1,N0,M0) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| (T1,N1,M0) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| missing | XX | XX | XX |
| Tumor clinical stage [2], n (%) | | | |
| n | XX | xx | XX |
| 0 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1A | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| IV | | | |
| missing | xx | XX | XX |

|---|---|---|---|
| Chemotherapy within 1 year prior to screening, n (%) | | | |
| n | XX | xx | xx |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| missing | xx | XX | xx |
| Radiotherapy within 1 year prior to screening, n (%) | | | |
| n | XX | xx | xx |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| missing | xx | XX | XX |
| Surgery within 1 year prior to screening, n (%) | | | |
| n | XX | xx | xx |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| missing | xx | XX | XX |
| Other treatments for breast cancer within 1 year proceeding, n (%) | for to | | |
| n | XX | xx | xx |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| missing | xx | XX | XX |
| ECOG score, n (%) | | | |
| n | XX | XX | XX |
| 0 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| missing | XX | XX | XX |

Data Source: Data Listing 16.x.x.x

Note: Percentages are based on the number of subjects with non-missing values from Full Analysis Set in each treatment group.

<sup>[1]</sup> The time in days from diagnosis as breast cancer to Informed Consent= Date of Informed Consent – Date of diagnosis as breast cancer +1.

<sup>[2]</sup> Tumor stage and clinical stage were assessed using breast carcinoma TNM staging system(Version 7). In clinical stage, 0 = (Tis, N0, M0), IA = (T1, N0, M0), IB = (T0, N1mi, M0) or (T1, N1, M0) or (T1, N1, M0) or (T2, N1, M0) or (T2, N2, M0), (T3, N1, M0), IIB = (T2, N1, M0) or (T3, N0, M0), IIIA = (T0, N2, M0), (T1, N2, M0), (T2, N2, M0), (T3, N1 or N2, M0), (T

|---|---|
| l | l |

IIIB = (T4, N0 or N1 or N2, M0), and IV = (any T, any N, M1).

#### Programming notes:

In clinical stage, Only the combination of (T, N, M) with a total number of observations not being 0 is listed.

There are 9 clinical stages: 0, IA, IB, IIA, IIB, IIIA, IIIB, IV, other, Only the categoty where the total number of observations is not 0 is listed.

In ECOG Score, Only the categoty where the total number of observations is not 0 is listed.

|---|---|---|

Similar tables as Table 14.2.3:

#### Table 14.2.4.1 Baseline Characteristics of the Disease – PP Analysis Set A

Data Source: Data Listing 16.x.x.x

Note: Percentages are based on the number of subjects with non-missing values from PP Analysis Set A in each treatment group.

- [1] The time in days from diagnosis as breast cancer to Informed Consent Date of diagnosis as breast cancer +1.
- [2] Tumor stage and clinical stage were assessed using breast carcinoma TNM staging system(Version 7). In clinical stage, 0 = (Tis, N0, M0), IA = (T1, N0, M0), IB = (T0, N1mi, M0) or (T1, N1, M0), IIA = (T0, N1, M0) or (T1, N1, M0) or (T2, N0, M0), IIB = (T2, N1, M0) or (T3, N0, M0).IIIA = (T0, N2, M0), (T1, N2, M0), (T2, N2, M0), (T3, N1 or N2, M0), IIB = (T4, N0 or N1 or N2, M0), and IV = (T3, N1, M1).

## Table 14.2.4.2 Baseline Characteristics of the Disease – PP Analysis Set B

Data Source: Data Listing 16.x.x.x

Note: Percentages are based on the number of subjects with non-missing values from PP Analysis Set B in each treatment group.

- [1] The time in days from diagnosis as breast cancer to Informed Consent= Date of Informed Consent Date of diagnosis as breast cancer +1.
- [2] Tumor stage and clinical stage were assessed using breast carcinoma TNM staging system(Version 7). In clinical stage, 0 = (Tis, N0, M0), IA = (T1, N0, M0), IB = (T0, N1mi, M0) or (T1, N1, M0), IIA = (T0, N1, M0) or (T1, N1, M0) or (T2, N0, M0), IIB = (T2, N1, M0) or (T3, N0, M0). IIIA = (T0, N2, M0), (T1, N2, M0), (T2, N2, M0), (T3, N1 or N2, M0), IIIB = (T4, N0 or N1 or N2, M0), and IV = (T3, N1, M1).

|-------------------------------------|-------------------|-----------------|
| Generon (Shanghai) Corporation Ltd. | SP11631 | 1.0, 2020-03-11 |

Table 14.2.5 Medical History, Symptoms and Surgical History – FAS

| - | F-627 | GRAN® | Total |
|---------------------------|-----------|-----------|-----------|
| MedDRA System Organ Class | (N=xx) | (N=xx) | (N=xx) |
| Preferred Term | n(%) | n(%) | n(%) |
| Prior Diseases | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| <soc #1=""></soc> | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| <pt #1-1=""></pt> | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| <pt #1-2=""></pt> | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| <soc #2=""></soc> | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| <pt #1-1=""></pt> | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| <pt #1-2=""></pt> | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Data Source: Data Listing 16.x.x.x

Note: Prior diseases are coded using MedDRA(Version 22.1).

Percentages are based on the number of subjects from Full Analysis Set in each treatment group.

Prior diseases are these diseases with an end date prior to the date of first chemotherapy.

|---|---|---|

Similar tables as Table 14.2.5:

# Table 14.2.6 Concomitant Diseases and Symptoms - FAS

Data Source: Data Listing 16.x.x.x

Note: Concomitant diseases are coded using MedDRA(Version 22.1).

Percentages are based on the number of subjects from Full Analysis Set in each treatment group.

Concomitant diseases are these diseases starting on or after the date of first chemotherapy, or diseases starting prior to the date of first chemotherapy but continuing after the date of first chemotherapy.

Programming notes: Change the row 1, column 1 "Prior diseases" to "Concomitant Diseases"...

# **Table 14.2.7 Surgical History of Breast Cancer – FAS**

Data Source: Data Listing 16.x.x.x

Note: Surgical history is coded using MedDRA(Version 22.1).

Percentages are based on the number of subjects from Full Analysis Set in each treatment group.

|--|--|---|---|---|
|--|--|---|---|---|

## **Table 14.2.8 Prior Medications – FAS**

| (N=xx) |
|-----------|
| (0/) |
| n(%) |
| xx (xx.x) |
| xx (xx.x) |
| xx (xx.x) |
| xx (xx.x) |

Data Source: Data Listing 16.x.x.x. Note: WHODrug Version B3 September 1, 2019.

Percentages are based on the number of subjects from Full Analysis Set in each treatment group. Prior medications are these drugs with an end date on or prior to the date of first chemotherapy.

|-------------------------------------|-------------------|-----------------|
| Generon (Shanghai) Corporation Ltd. | SP11631 | 1.0, 2020-03-11 |

Similar tables as Table 14. 2.8:

## **Table 14.2.9.1 Concomitant Medications – FAS**

Data Source: Data Listing 16.x.x.x

Note: WHODrug Version B3 September 1, 2019.

Percentages are based on the number of subjects from Full Analysis Set in each treatment group.

Concomitant medications are these medications other than the study drug used from the date of first chemotherapy to the Day 21 of Cycle 4.

Similar tables as Table 14.2.5:

# **Table 14.2.9.2 Concomitant Non-Drug Treatments – FAS**

Data Source: Data Listing 16.x.x.x

Note: Concomitant non-drug treatments are coded using MedDRA(Version 22.1).

Percentages are based on the number of subjects from Full Analysis Set in each treatment group.

Programming notes: Change the row 1, column 1 "Prior diseases" to " Concomitant Non-Drug Treatments".

|-------------------------------------|-------------------|-----------------|
| Generon (Shanghai) Corporation Ltd. | SP11631 | 1.0, 2020-03-11 |

Table 14.2.10 Extent of Exposure to Study Medication(F-627, GRAN®)-Safety Analysis Set

| <b>Table 14.2</b> | .10 Extent of Exposure to Study Medication | n(F-627, GRAN®)–Safety Ana | alysis Set |
|---|---|---|---|
| _ | | F-627 | GRAN® |
| Cycle | | (N=xx) | (N=xx) |
| Cycle 1 | Actual frequency of drug administration | | |
| | n(missing) | xx(xx) | xx(xx) |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X |
| | Min , Max | xx, xx | xx, xx |
| | Actual cumulative dose [1] | | |
| | n(missing) | XX(XX) | xx(xx) |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X |
| | Min , Max | xx, xx | xx, xx |
| | Actual dose intensity [2] | | |
| | n(missing) | XX(XX) | XX(XX) |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X |
| | Min , Max | xx, xx | xx, xx |
| | Relative dose intensity (RDI) (%) [3] | | |
| | n(missing) | XX(XX) | XX(XX) |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X |
| | Min, Max | XX, XX | xx, xx |

| Sponsor :<br>Generon (Shanghai) Corpo | ration Ltd. | Protocol Number :<br>SP11631 | | Version, date : 1.0, 2020-03-11 |
|---|---|---|---|---|
| | Category of relative | dose intensity [4], n (%) | · | |
| | >110% | | xx (xx.x) | xx (xx.x) |
| | >100-110% | | xx (xx.x) | xx (xx.x) |
| | >90 - 100% | | xx (xx.x) | xx (xx.x) |
| | >80 - 90% | | xx (xx.x) | xx (xx.x) |
| | >70 - 80% | | xx (xx.x) | xx (xx.x) |
| | >60 - 70% | | xx (xx.x) | xx (xx.x) |
| | >50 - 60% | | xx (xx.x) | xx (xx.x) |
| | ≤50% | | xx (xx.x) | xx (xx.x) |
| Cycle 2 | | | | |
| Cycle 3 | | | | |
| Cycle 4 | | | | |
| All treatment periods | | | | |

Data Source: Data Listing 16.x.x.x

Note: Treated as misssing for subjects with no drug administration within the cycle.

- [1] Actual cumulative dose, Unit of F-627: mg, Unit of GRAN®: µg.
- [2] For GRAN®, Actual dose intensity( $\mu$ g/kg/day)= (Actual cumulative dose / Weight) / Actual days of drug administration, the weight used for analysis should be the last valid weight value measured before or on the start date of chemotherapy of each cycle. For F-627, Actual dose intensity( $\mu$ g/kg/day) = (Actual cumulative dose / Actual frequency of drug administration.
- [3] Relative dose intensity (RDI) (%) = Actual dose intensity / Planned dose intensity \*100.
- [4] Percentages of category of relative dose intensity are based on the number of evaluable subjects from Safety Analysis Set in each treatment group and each cycle.

Programming notes: relative dose intensity (%) is rounded to integer. The decimal place of each statistics is displayed in SAP.

Programming notes: Total frequency of drug administration in cycle 1 is calculated based on the number of subjects who completed Cycle 1 treatment; Total frequency of drug administration in cycle 2 is calculated based on the number of subjects who completed Cycle 2 treatment; etc.

| Sponsor : | Protocol Number : | Version, date: |
|-------------------------------------|-------------------|-----------------|
| Generon (Shanghai) Corporation Ltd. | SP11631 | 1.0, 2020-03-11 |

Similar tables as Table 14.2.10:

### Table 14.2.11 Extent of Exposure to Chemotherapy drugs(Epirubicin, Cyclophosphamide) -Safety Analysis Set

Data Source: Data Listing 16.x.x.x

Note: Treated as misssing for subjects with no drug administration within the cycle.

- [1] Actual dose intensity (mg/m^2/frequency)=Actual cumulative dose / Body surface area (BSA) / Total frequency of drug administration.
- [2] Relative dose intensity (RDI) (%) = Actual dose intensity / Planned dose intensity \*100.
- [3] According to the Gao Billiangformula: Body surface area (BSA) =  $0.007184 \times \text{Weight}$  (kg) $0.425 \times \text{Height}$ (cm)0.725. The weight used for the analysis should be the last valid weight value measured before or on the start date of chemotherapy of each cycle.
- [4] Percentages of category of relative dose intensity are based on the number of evaluable subjects from Safety Analysis Set in each treatment group and each cycle.

Programming notes: relative dose intensity (%) is rounded to integer. The decimal place of each statistics is displayed in SAP.

| Sponsor: Version, date: Generon (Shanghai) Corporation Ltd. SP11631 1.0, 2020-03-11 | - F | Protocol Number :<br>SP11631 | Version, date: 1.0, 2020-03-11 |
|---|---|---|---|
|---|---|---|---|

Table 14.3.1.1 Duration of Grade 3 or 4 Neutropenia during Cycle 1 – FAS

| | F-627 | GRAN® |
|---|---|---|
| Statistics (Day) | (N=xx) | (N=xx) |
| n(missing) | XX(XX) | XX(XX) |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX |
| (F-627 - GRAN®) Hodges-Lehmann Estimation (95% CI) (F-627 - GRAN®) Hodges-Lehmann Estimation (the upper limit of the one-sided 97.5% CI) $^{[1]}$ | xx.x (xx.xx-xx.xx)<br>xx.x (xx.xx) | |

Note: Missing ANC values within the first 13 days of a cycle will be imputed using the method specified in SAP. Grade 3 or 4 neutropenia is defined as ANC<  $1.0 \times 10^9$ /L or ANC<  $0.5 \times 10^9$ /L.

Programme note: Keep 1 decimal place for Hodges-Lehmann Estimation and 2 decimal places for 97.5% CI

<sup>[1]</sup> The upper limit of the one-sided 97.5% CI is estimated by Hodges-Lehmann method for the difference in duration (day) of Grade 3 or 4 neutropenia between F-627 vs. GRAN® during Cycle 1. If the upper limit of the one-sided 97.5% CI <=1, then the non-inferiority hypothesis test will be valid.

| Sponsor :<br>Generon (Shanghai) Corporation Ltd. | Protocol Number :<br>SP11631 | Version, date: 1.0, 2020-03-11 |
|---|---|---|

Similar tables as Table 14.3.1.1:

## Table 14.3.1.2 Duration of Grade 3 or 4 Neutropenia during Cycle 1 – PP Analysis Set A

Note: Missing ANC values within the first 13 days of a cycle will be imputed using the method specified in SAP.

Grade 3 or 4 neutropenia is defined as ANC<  $1.0 \times 10^9$ /L or ANC<  $0.5 \times 10^9$ /L.

[1] The upper limit of the one-sided 97.5% CI is estimated by Hodges-Lehmann method for the difference in duration (day) of Grade 3 or 4 neutropenia between F-627 vs.  $GRAN^{\otimes}$  during Cycle 1. If the upper limit of the one-sided 97.5% CI <=1, then the non-inferiority hypothesis test will be valid.

Programming notes: Note to add the unit (Day);

Please pay attention to change the "Full Analysis Set" into "PP Analysis Set A" in footnote;

# Table 14.3.1.3 Duration of Grade 3 or 4 Neutropenia during Cycle 1 – FAS (No Imputation for ANC missing data)

Note: Missing ANC values will not be imputed.

Grade 3 or 4 neutropenia is defined as ANC< 1.0  $\times$  10<sup>9</sup>/L or ANC< 0.5  $\times$  10<sup>9</sup>/L.

[1] The upper limit of the one-sided 97.5% CI is estimated by Hodges-Lehmann method for the difference in duration (days) of Grade 3 or 4 neutropenia between F-627 vs. GRAN® during Cycle 1.

Programming notes: Note to add the unit (Day);

Please pay attention to add the subtitle" (No Imputation for ANC missing data)";

| Sponsor :<br>Generon (Shanghai) Corporation Ltd. | Protocol Number :<br>SP11631 | Version, date: 1.0, 2020-03-11 |
|---|---|---|

Table 14.3.1.4 Sensitivity Analysis for Duration of Grade 3 or 4 Neutropenia during Cycle 1
- Subjects with Grade 3 or 4 neutropenia during Cycle 1 in FAS

| 8 / | |
|---|---|
| F-627 | GRAN® |
| (N=xx) | (N=xx) |
| XX | XX |
| xx.x (xx.xx) | xx.x (xx.xx) |
| XX.X | XX.X |
| xx, xx | xx, xx |
| xx.x (xx.xx-xx.xx) | |
| xx.x (xx.xx) | |
| | F-627<br>(N=xx)<br>xx<br>xx.x (xx.xx)<br>xx.x (xx.xx)<br>xx.x xx, xx |

Note: Missing ANC values within the first 13 days of a cycle will be imputed using the method specified in SAP.

Grade 3 or 4 neutropenia is defined as ANC<  $1.0 \times 10^9$ /L or ANC<  $0.5 \times 10^9$ /L.

<sup>[1]</sup> The difference in mean (F-627 minus GRAN®) and its CI for the duration (day) of Grade 3 or 4 neutropenia are estimated by t-test for subjects with Grade 3 or 4 neutropenia during Cycle 1.

| Sponsor :<br>Generon (Shanghai) Corporati | Protocol Number :<br>SP11631 | Version, date: 1.0, 2020-03-11 |
|---|---|---|

Table 14.3.2.1 The Incidence of Grade 3 or 4 Neutropenia for Cycle 1 – FAS

| | F-627 | $GRAN^{	ext{@}}$ |
|---|---|---|
| Statistics | (N = xx) | (N = xx) |
| n | XX | XX |
| Yes, n (%) | xx (xx.x) | xx (xx.x) |
| No, n (%) | xx (xx.x) | xx (xx.x) |
| missing | xx | xx |
| Difference in Incidence (F-627-GRAN®) (95% CI) <sup>[1]</sup> | xx.x (xx.x- xx.x) | |
| P-value [1] | XX.XXX | |

Data Source: Data Listing 16.x.x.x.

Note: Missing ANC values within the first 13 days of a cycle will be imputed using the method specified in SAP.

Grade 3 or 4 neutropenia is defined as ANC<  $1.0 \times 10^9$ /L or ANC<  $0.5 \times 10^9$ /L. Percentages are based on the number of evaluable subjects from Full Analysis Set in each treatment group.

[1] The difference in incidence of Grade 3 or 4 neutropenia between F-627 and GRAN®. and its 95% CI is estimated. P value is calculated based on the chi-square/Fisher (Fisher's exact test will be used if there observed at least one expected frequency less than 1).

Programming notes: All p-values will be rounded to three decimal places. If a p-value is less than 0.001 it will be reported as "<0.001."

| Sponsor : | Protocol Number : | Version, date: |
|-------------------------------------|-------------------|-----------------|
| Generon (Shanghai) Corporation Ltd. | SP11631 | 1.0, 2020-03-11 |

Similar tables as Table 14.3.2.1:

### Table 14.3.2.2 The Incidence of Grade 3 or 4 Neutropenia for Cycle 1 – PP Analysis Set A

Data Source: Data Listing 16.x.x.x.

Note: Missing ANC values within the first 13 days of a cycle will be imputed using the method specified in SAP.

Grade 3 or 4 neutropenia is defined as ANC $< 1.0 \times 10^9/L$  or ANC $< 0.5 \times 10^9/L$ . Percentages are based on the number of evaluable subjects from PP Analysis Set A in each treatment group.

[1] The difference in incidence of Grade 3 or 4 neutropenia between F-627 and GRAN®. and its 95% CI is estimated. P value is calculated based on the chi-square/Fisher (Fisher's exact test will be used if there observed at least one expected frequency less than 1).

Programming notes: Please pay attention to change the "Full Analysis Set" into "PP Analysis Set A" in footnote; Note to add the unit (Days);

| | | D. J. IN. J. | |
|---|---|---|---|
| , | ponsor: | Protocol Number :<br>SP11631 | Version, date :<br>1.0, 2020-03-11 |
| U | eneron (Shanghai) Corporation Ltd. | 3F11031 | 1.0, 2020-03-11 |

Table 14.3.2.3 The Incidence of Grade 3 or 4 Neutropenia for Cycle 2-4 and All Treatment Periods – FAS

| 1 4010 1 11012 | b The includince of Grade of Tricallopenia | | cutificate i ci ious - 1 i k |
|---|---|---|---|
| | • | F-627 | GRAN® |
| Phase | Statistics | (N = xx) | (N = xx) |
| Cycle 2 | n | XX | xx |
| | Yes, n (%) | xx (xx.x) | xx (xx.x) |
| | No, n (%) | xx (xx.x) | xx (xx.x) |
| | missing | XX | XX |
| | Difference in Incidence (F-627-GRAN®) (95% CI) <sup>[1]</sup> | xx.x (xx.x- xx.x) | |
| | P-value [1] | XX.XXX | |
| Cycle 3 | n | XX | XX |
| | Yes, n (%) | xx (xx.x) | xx (xx.x) |
| | No, n (%) | xx (xx.x) | xx (xx.x) |
| | missing | XX | XX |
| | Difference in Incidence (F-627-GRAN®) (95% CI) <sup>[1]</sup> | xx.x (xx.x- xx.x) | |
| | P-value [1] | XX.XXX | |
| Cycle 4 | | | |

All Treatment Periods

Data Source: Data Listing 16.x.x.x.

Note: Missing ANC values within the first 13 days of a cycle will be imputed using the method specified in SAP.

Grade 3 or 4 neutropenia is defined as ANC< 1.0 × 10<sup>9</sup>/L or ANC< 0.5 × 10<sup>9</sup>/L. Percentages are based on the number of evaluable subjects from Full Analysis Set in each treatment group and each cycle.

[1] The difference in incidence of Grade 3 or 4 neutropenia between F-627 and GRAN® and its 95% CI is estimated. P value is calculated based on the chisquare/Fisher (Fisher's exact test will be used if there observed at least one expected frequency less than 1).

Programming notes: All p-values will be rounded to three decimal places. If a p-value is less than 0.001 it will be reported as "<0.001."

| Generon (Shanghai) Corporation Ltd. SP11631 1.0, 2020-03-11 |
|-------------------------------------------------------------|
|-------------------------------------------------------------|

Similar tables as Table 14.3.2.3:

# Table 14.3.2.4 The Incidence of Grade 3 or 4 Neutropenia for Cycle 2-4 and All Treatment Periods – PP Analysis Set B

Data Source: Data Listing 16.x.x.x.

Note: Missing ANC values within the first 13 days of a cycle will be imputed using the method specified in SAP.

Grade 3 or 4 neutropenia is defined as ANC<  $1.0 \times 10^9$ /L or ANC<  $0.5 \times 10^9$ /L. Percentages are based on the number of evaluable subjects from PP Analysis Set B in each treatment group and each cycle.

[1] The difference in incidence of Grade 3 or 4 neutropenia between F-627 and GRAN® and its 95% CI is estimated. P value is calculated based on the chi-square/Fisher (Fisher's exact test will be used if there observed at least one expected frequency less than 1).

Programming notes: Please pay attention to change the "Full Analysis Set" into "PP Analysis Set B" in footnote;

|-------------------------------------|-------------------|-----------------|
| Generon (Shanghai) Corporation Ltd. | SP11631 | 1.0, 2020-03-11 |

Table 14.3.3.1 Duration of Grade 3 or 4 Neutropenia for Cycle 2-4 and All Treatment Periods – FAS

| | | F-627 | $GRAN^{\circledast}$ |
|---|---|---|---|
| Phase | Statistics (Day) | (N = xx) | (N = xx) |
| Cycle 2 | n(missing) | XX(XX) | xx(xx) |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X |
| | Min , Max | XX - XX | xx - xx |
| | (F-627 - GRAN®) Hodges-Lehmann Estimation (95% $CI$ ) <sup>[1]</sup> | xx.x (xx.xx-xx.xx) | |

Cycle 3

Cycle 4

Cycle

All Treatment Periods

Note: Missing ANC values within the first 13 days of a cycle will be imputed using the method specified in SAP. Grade 3 or 4 neutropenia is defined as ANC<  $1.0 \times 10^9$ /L or ANC<  $0.5 \times 10^9$ /L.

[1] Hodges-Lehmann is used to estimate the difference and its 95% CI for duration (days) of Grade 3 or 4 neutropenia between F-627 and GRAN® for Cycle 2-4 and all treatment periods.

Programme note: Hodges-Lehmann Estimation kept 1 decimal place and 2 decimal places reserved for 97.5% CI

| Generon (Shanghai) Corporation Ltd. SP11631 1.0, 2020-03-11 |
|-------------------------------------------------------------|
|-------------------------------------------------------------|

Similar tables as Table 14.3.3.1:

# Table 14.3.3.2 Duration of Grade 3 or 4 Neutropenia during Cycle 2-4 and All Treatment Periods – PP Analysis Set B

Note: Missing ANC values within the first 13 days of a cycle will be imputed using the method specified in SAP. Grade 3 or 4 neutropenia is defined as ANC<  $1.0 \times 10^9$ /L or ANC<  $0.5 \times 10^9$ /L.

[1] Hodges-Lehmann is used to estimate the difference and its 95% CI for duration (days) of Grade 3 or 4 neutropenia between F-627 and GRAN® for Cycle 2-4 and all treatment periods.

Programming notes: Please pay attention to change the "Full Analysis Set" into "PP Analysis Set B" in footnote; Note to add the unit (Day) after "Statistics";

| Generon (Shanghai) Corporation Ltd. SP11631 1.0, 2020-03-11 |
|-------------------------------------------------------------|
|-------------------------------------------------------------|

# Table 14.3.4.1 Duration of Grade 4 Neutropenia during Cycle 1 – FAS

| | F-627 | $GRAN^{\scriptscriptstyle{\circledR}}$ |
|---|---|---|
| Statistics (Day) | (N=xx) | (N=xx) |
| n(missing) | XX(XX) | XX(XX) |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X |
| Min , Max | xx, xx | xx, xx |
| (F-627 - GRAN®) Hodges-Lehmann Estimation (95% CI) | xx.x (xx.x- xx.x) | |

Note: Missing ANC values within the first 13 days of a cycle will be imputed using the method specified in SAP. Grade 4 neutropenia is defined as ANC<  $0.5 \times 10^9$ /L.

| Smanaani | Protocal Nymbor | Varian data |
|---|---|---|
| Sponsor: Generon (Shanghai) Corporation Ltd. | Protocol Number :<br>SP11631 | Version, date :<br>1.0, 2020-03-11 |

Similar tables as Table 14.3.4.1:

## Table 14.3.4.2 Duration of Grade 4 Neutropenia during Cycle 1 – PP Analysis Set A

Note: Missing ANC values within the first 13 days of a cycle will be imputed using the method specified in SAP. Grade 4 neutropenia is defined as ANC<  $0.5 \times 10^9$ /L.

Programming notes: Please pay attention to change the "Full Analysis Set" into "PP Analysis Set A" in footnote; Note to add the unit (Day) after "Statistics";

Similar tables as Table 14.3.3.1:

## Table 14.3.4.3 Duration of Grade 4 Neutropenia during Cycle 2-4 and All Treatment Periods – FAS

Note: Missing ANC values within the first 13 days of a cycle will be imputed using the method specified in SAP. Grade 4 neutropenia is defined as ANC<  $0.5 \times 10^9$ /L.

Programming notes: Note to add the unit (Day) after "Statistics";

# Table 14.3.4.4 Duration of Grade 4 Neutropenia during Cycle 2-4 and All Treatment Periods – PP Analysis Set B

Note: Missing ANC values within the first 13 days of a cycle will be imputed using the method specified in SAP. Grade 4 neutropenia is defined as ANC<  $0.5 \times 10^9$ /L.

Programming notes: Please pay attention to change the "Full Analysis Set" into "PP Analysis Set B" in footnote; Note to add the unit (Day) after "Statistics";

| Sponsor : | Protocol Number : | Version, date: |
|-------------------------------------|-------------------|-----------------|
| Generon (Shanghai) Corporation Ltd. | SP11631 | 1.0, 2020-03-11 |

Similar tables as Table 14.3.2.1:

#### Table 14.3.4.5 The Incidence of Grade 4 Neutropenia for Cycle 1 – FAS

Data Source: Data Listing 16.x.x.x.

Note: Missing ANC values within the first 13 days of a cycle will be imputed using the method specified in SAP.

Grade 4 neutropenia is defined as ANC $< 0.5 \times 10^9/L$ .

Percentages are based on the number of evaluable subjects from Full Analysis Set in each treatment group and each cycle.

[1] The difference in incidence of Grade 4 neutropenia between F-627 and GRAN® and its 95% CI is estimated. P value is calculated based on the chi-square/Fisher (Fisher's exact test will be used if there observed at least one expected frequency less than 1).

#### Table 14.3.4.6 The Incidence of Grade 4 Neutropenia for Cycle 1 – PP Analysis Set A

Data Source: Data Listing 16.x.x.x.

Note: Missing ANC values within the first 13 days of a cycle will be imputed using the method specified in SAP.

Grade 4 neutropenia is defined as ANC<  $0.5 \times 10^9$ /L.

Percentages are based on the number of evaluable subjects from PP Analysis Set A in each treatment group and each cycle.

[1] The difference in incidence of Grade 4 neutropenia between F-627 and GRAN® and its 95% CI is estimated. P value is calculated based on the chi-square/Fisher (Fisher's exact test will be used if there observed at least one expected frequency less than 1).

Programming notes: Please pay attention to change the "Full Analysis Set" into "PP Analysis Set A" in footnote;

Similar tables as Table 14.3.2.3:

## Table 14.3.4.7 The Incidence of Grade 4 Neutropenia for Cycle 2-4 and All Treatment Periods – FAS

Data Source: Data Listing 16.x.x.x.

Note: Missing ANC values within the first 13 days of a cycle will be imputed using the method specified in SAP.

Grade 4 neutropenia is defined as ANC<  $0.5 \times 10^9$ /L.

Percentages are based on the number of evaluable subjects from Full Analysis Set in each treatment group and each cycle.

[1] The difference in incidence of Grade 4 neutropenia between F-627 and GRAN® and its 95% CI is estimated. P value is calculated based on the chi-square/Fisher (Fisher's exact test will be used if there observed at least one expected frequency less than 1).

# Table 14.3.4.8 The Incidence of Grade 4 Neutropenia for Cycle 2-4 and All Treatment Periods – PP Analysis Set B

Data Source: Data Listing 16.x.x.x.

Note: Missing ANC values within the first 13 days of a cycle will be imputed using the method specified in SAP.

Grade 4 neutropenia is defined as ANC<  $0.5 \times 10^9$ /L.

Percentages are based on the number of evaluable subjects from PP Analysis Set B in each treatment group and each cycle.

[1] The difference in incidence of Grade 4 neutropenia between F-627 and GRAN® and its 95% CI is estimated. P value is calculated based on the chi-square/Fisher

| Generon (Shanghai) Corporation Ltd. SP11631 1.0, 2020-03-11 |
|-------------------------------------------------------------|
|-------------------------------------------------------------|

(Fisher's exact test will be used if there observed at least one expected frequency less than 1).

Programming notes: Please pay attention to change the "Full Analysis Set" into "PP Analysis Set B" in footnote;

|---|---|---|

Similar tables as Table 14.3.4.1:

### Table 14.3.5.1 The total Duration of Grade 3 or 4 Neutropenia during 4 Cycles – FAS

Note: Missing ANC values within the first 13 days of a cycle will be imputed using the method specified in SAP. Grade 3 or 4 neutropenia is defined as ANC<  $1.0 \times 10^9$ /L or ANC<  $0.5 \times 10^9$ /L.

The total Duration (day) of Grade 3 or 4 Neutropenia during 4 Cycles = Duration of Grade 3 or 4 Neutropenia during Cycle 1 (day) + Duration of Grade 3 or 4 Neutropenia during Cycle 2 (day) + Duration of Grade 3 or 4 Neutropenia during Cycle 3 (day) + Duration of Grade 3 or 4 Neutropenia during Cycle 4 (day).

Programming notes: Note to add the unit (Day) after "Statistics";

### Table 14.3.5.2 The total Duration of Grade 3 or 4 Neutropenia during 4 Cycles – PP Analysis Set B

Note: Missing ANC values within the first 13 days of a cycle will be imputed using the method specified in SAP. Grade 3 or 4 neutropenia is defined as ANC<  $1.0 \times 10^9$ /L or ANC<  $0.5 \times 10^9$ /L.

The total Duration (day) of Grade 3 or 4 Neutropenia during 4 Cycles = Duration of Grade 3 or 4 Neutropenia during Cycle 1 (day) + Duration of Grade 3 or 4 Neutropenia during Cycle 2 (day) + Duration of Grade 3 or 4 Neutropenia during Cycle 4 (day).

Programming notes: Please pay attention to change the "Full Analysis Set" into "PP Analysis Set B" in footnote; Note to add the unit (Day) after "Statistics";

| Sponsor :<br>Generon (Shanghai) Corporation Ltd. | Protocol Number :<br>SP11631 | Version, date:<br>1.0, 2020-03-11 |
|---|---|---|

Similar tables as Table 14.3.4.1:

#### Table 14.3.6.1 Duration of Grade 2 or Higher Neutropenia during Cycle 1 – FAS

Note: Missing ANC values within the first 13 days of a cycle will be imputed using the method specified in SAP. Grade 2 neutropenia is defined as ANC<  $1.5 \times 10^9$ /L.

Programming notes: Note to add the unit (Day)

## Table 14.3.6.2 Duration of Grade 2 or Higher Neutropenia during Cycle 1 – PP Analysis Set A

Note: Missing ANC values within the first 13 days of a cycle will be imputed using the method specified in SAP. Grade 2 neutropenia is defined as ANC<  $1.5 \times 10^9$ /L.

Programming notes: Please pay attention to change the "Full Analysis Set" into "PP Analysis Set A" in footnote; Note to add the unit (Day) after "Statistics";

Similar tables as Table 14.3.3.1:

#### Table 14.3.6.3 Duration of Grade 2 or Higher Neutropenia during Cycle 2-4 and All Treatment Periods – FAS

Note: Missing ANC values within the first 13 days of a cycle will be imputed using the method specified in SAP. Grade 2 neutropenia is defined as ANC<  $1.5 \times 10^9$ /L.

Programming notes: Note to add the unit (Day) after "Statistics";

# Table 14.3.6.4 Duration of Grade 2 or Higher Neutropenia during Cycle 2-4 and All Treatment Periods – PP Analysis Set B

Note: Missing ANC values within the first 13 days of a cycle will be imputed using the method specified in SAP. Grade 2 neutropenia is defined as ANC<  $1.5 \times 10^9$ /L.

Programming notes: Please pay attention to change the "Full Analysis Set" into "PP Analysis Set B" in footnote; Note to add the unit (Day) after "Statistics";

|-------------------------------------|-------------------|-----------------|
| Generon (Shanghai) Corporation Ltd. | SP11631 | 1.0, 2020-03-11 |

Similar tables as Table 14.3.2.1:

#### Table 14.3.6.5 The Incidence of Grade 2 or Higher Neutropenia for Cycle 1 – FAS

Data Source: Data Listing 16.x.x.x.

Note: Missing ANC values within the first 13 days of a cycle will be imputed using the method specified in SAP.

Grade 2 neutropenia is defined as ANC<  $1.5 \times 10^9$ /L.

Percentages are based on the number of evaluable subjects from Full Analysis Set in each treatment group and each cycle.

[1] The difference in incidence of Grade 4 neutropenia between F-627 and GRAN® and its 95% CI is estimated. P value is calculated based on the chi-square/Fisher (Fisher's exact test will be used if there observed at least one expected frequency less than 1).

### Table 14.3.6.6 The Incidence of Grade 2 or Higher Neutropenia for Cycle 1 – PP Analysis Set A

Data Source: Data Listing 16.x.x.x.

Note: Missing ANC values within the first 13 days of a cycle will be imputed using the method specified in SAP.

Grade 2 neutropenia is defined as ANC $< 1.5 \times 10^9/L$ .

Percentages are based on the number of evaluable subjects from PP Analysis Set A in each treatment group and each cycle.

[1] The difference in incidence of Grade 4 neutropenia between F-627 and GRAN® and its 95% CI is estimated. P value is calculated based on the chi-square/Fisher (Fisher's exact test will be used if there observed at least one expected frequency less than 1).

Programming notes: Please pay attention to change the "Full Analysis Set" into "PP Analysis Set A" in footnote;

Similar tables as Table 14.3.2.3:

# Table 14.3.6.7 The Incidence of Grade 2 or Higher Neutropenia for Cycle 2-4 and All Treatment Periods – FAS

Data Source: Data Listing 16.x.x.x.

Note: Missing ANC values within the first 13 days of a cycle will be imputed using the method specified in SAP.

Grade 2 neutropenia is defined as ANC $< 1.5 \times 10^9$ /L.

Percentages are based on the number of evaluable subjects from Full Analysis Set in each treatment group and each cycle.

[1] The difference in incidence of Grade 4 neutropenia between F-627 and GRAN® and its 95% CI is estimated. P value is calculated based on the chi-square/Fisher (Fisher's exact test will be used if there observed at least one expected frequency less than 1).

# Table 14.3.6.8 The Incidence of Grade 2 or Higher Neutropenia for Cycle 2-4 and All Treatment Periods – PP Analysis Set B

Data Source: Data Listing 16.x.x.x.

Note: Missing ANC values within the first 13 days of a cycle will be imputed using the method specified in SAP.

|--|

Grade 2 neutropenia is defined as ANC< 1.5  $\times$  10 $^{9}$ /L.

Percentages are based on the number of evaluable subjects from PP Analysis Set B in each treatment group and each cycle.

[1] The difference in incidence of Grade 4 neutropenia between F-627 and GRAN® and its 95% CI is estimated. P value is calculated based on the chi-square/Fisher (Fisher's exact test will be used if there observed at least one expected frequency less than 1).

Programming notes: Please pay attention to change the "Full Analysis Set" into "PP Analysis Set B" in footnote;

|-------------------------------------|-------------------|-----------------|
| Generon (Shanghai) Corporation Ltd. | SP11631 | 1.0, 2020-03-11 |

Similar tables as Table 14.3.2.1:

## Table 14.3.7.1 The Incidence of Febrile Neutropenia (FN) for Cycle 1 – FAS

Data Source: Data Listing 16.x.x.x.

Note: Missing ANC values within the first 13 days of a cycle will be imputed using the method specified in SAP.

Febrile neutropenia is defined as ANC <1.0×10<sup>9</sup>/L and a single measurement of body temperature > 38.3 °C or a body temperature ≥ 38.0 °C sustained over 1 hour.

Percentages are based on the number of evaluable subjects from Full Analysis Set in each treatment group and each cycle.

[1] The difference in incidence of Febrile neutropenia between F-627 and GRAN® and its 95% CI is estimated. P value is calculated based on the chi-square/Fisher (Fisher's exact test will be used if there observed at least one expected frequency less than 1).

#### Table 14.3.7.2 The Incidence of Febrile Neutropenia (FN) for Cycle 1 – PP Analysis Set A

Data Source: Data Listing 16.x.x.x.

Note: Missing ANC values within the first 13 days of a cycle will be imputed using the method specified in SAP.

Febrile neutropenia is defined as ANC  $<1.0 \times 10^9$ /L and a single measurement of body temperature >38.3 °C or a body temperature >38.0 °C sustained over 1 hour .

Percentages are based on the number of evaluable subjects from PP Analysis Set A in each treatment group and each cycle.

[1] The difference in incidence of Febrile neutropenia between F-627 and GRAN® and its 95% CI is estimated. P value is calculated based on the chi-square/Fisher (Fisher's exact test will be used if there observed at least one expected frequency less than 1).

Programming notes: Please pay attention to change the "Full Analysis Set" into "PP Analysis Set A" in footnote;

Similar tables as Table 14.3.2.3:

### Table 14.3.7.3 The Incidence of Febrile Neutropenia (FN) for Cycle 2-4 and All Treatment Periods – FAS

Data Source: Data Listing 16.x.x.x.

Note: Missing ANC values within the first 13 days of a cycle will be imputed using the method specified in SAP.

Febrile neutropenia is defined as ANC <1.0×10<sup>9</sup>/L and a single measurement of body temperature > 38.3 °C or a body temperature ≥ 38.0 °C sustained over 1 hour.

Percentages are based on the number of evaluable subjects from Full Analysis Set in each treatment group and each cycle.

[1] The difference in incidence of Febrile neutropenia between F-627 and GRAN® and its 95% CI is estimated. P value is calculated based on the chi-square/Fisher (Fisher's exact test will be used if there observed at least one expected frequency less than 1).

# Table 14.3.7.4 The Incidence of Febrile Neutropenia (FN) for Cycle 2-4 and All Treatment Periods – PP Analysis Set B

Data Source: Data Listing 16.x.x.x.

Note: Missing ANC values within the first 13 days of a cycle will be imputed using the method specified in SAP.

Febrile neutropenia is defined as ANC <1.0×10<sup>9</sup>/L and a single measurement of body temperature > 38.3 °C or a body temperature ≥ 38.0 °C sustained over 1 hour.

Percentages are based on the number of evaluable subjects from PP Analysis Set B in each treatment group and each cycle.

[1] The difference in incidence of Febrile neutropenia between F-627 and GRAN® and its 95% CI is estimated. P value is calculated based on the chi-square/Fisher (Fisher's exact test will be used if there observed at least one expected frequency less than 1).

|---|---|---|

Programming notes: Please pay attention to change the "Full Analysis Set" into "PP Analysis Set B" in footnote;
| Sponsor: | Protocol Number: | Version, date : |
|-------------------------------------|------------------|-----------------|
| Generon (Shanghai) Corporation Ltd. | SP11631 | 1.0, 2020-03-11 |

Table 14.3.8.1 ANC nadir from day 3 to day 13 for Cycle 1 – FAS

| | F-627 | $GRAN^{\circledast}$ |
|---|---|---|
| Statistics (10 <sup>9</sup> /L) | (N=xx) | (N=xx) |
| n(missing) | XX(XX) | xx(xx) |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X |
| Min , Max | XX, XX | xx, xx |
| (F-627 - GRAN®) Hodges-Lehmann Estimation (95% CI) | xx.x (xx.x- xx.x) | |

Data Source: Data Listing 16.x.x.x

Note: Missing ANC values within the first 13 days of a cycle will be imputed using the method specified in SAP.

Similar tables as Table 14.3.8.1:

#### Table 14.3.8.2 ANC nadir from day 3 to day 13 for Cycle 1 – PP Analysis Set A

Data Source: Data Listing 16.x.x.x

Note: Missing ANC values within the first 13 days of a cycle will be imputed using the method specified in SAP.

Programming notes: Please pay attention to change the "Full Analysis Set" into "PP Analysis Set A" in footnote; Note to add the unit  $(10^9/L)$  after "Statistics";

Similar tables as Table 14.3.3.1: (Note to update the unit after the statistics in the header.)

### Table 14.3.8.3 ANC nadir from day 3 to day 13 within a cycle for Cycle 2-4 – FAS

Data Source: Data Listing 16.x.x.x

Note: Missing ANC values within the first 13 days of a cycle will be imputed using the method specified in SAP.

### Table 14.3.8.4 ANC nadir from day 3 to day 13 within a cycle for Cycle 2-4 – PP Analysis Set B

Data Source: Data Listing 16.x.x.x

Note: Missing ANC values within the first 13 days of a cycle will be imputed using the method specified in SAP.

Programming notes: Note to add the unit (10<sup>9</sup>/L) after "Statistics";

|---|---|---|

Similar tables as Table 14.3.4.1:

#### Table 14.3.9.1 Time in days to ANC Recovery Post Nadir for Cycle 1– FAS

Note: Missing ANC values within the first 13 days of a cycle will be imputed using the method specified in SAP.

ANC recovery is defined as an ANC  $\geq 2.0 \times 10^9 / L$  after the expected ANC nadir.

Nadir is the lowest ANC value observed in the first 13 days of a cycle.

If nadir point of ANC  $< 2.0 \times 10^9$ /L during the first 13 days of a cycle, then time in days to ANC Recovery = (Start Date when ANC  $\ge 2.0 \times 10^9$ /L) - (Date of nadir in this cycle) + 1

If ANC  $\ge 2.0 \times 10^9$ /L during the first 13 days of a cycle, then time in days to ANC Recovery equals to 0 days.

#### Table 14.3.9.2 Time in days to ANC Recovery Post Nadir for Cycle 1 – PP Analysis Set A

Note: Missing ANC values within the first 13 days of a cycle will be imputed using the method specified in SAP.

ANC recovery is defined as an ANC  $\geq$  2.0  $\times$  10<sup>9</sup>/L after the expected ANC nadir.

Nadir is the lowest ANC value observed in the first 13 days of a cycle.

If nadir point of ANC  $< 2.0 \times 10^9$ /L during the first 13 days of a cycle, then time in days to ANC Recovery = (Start Date when ANC  $\ge 2.0 \times 10^9$ /L) - (Date of nadir in this cycle) + 1

If ANC  $\ge 2.0 \times 10^9$ /L during the first 13 days of a cycle, then time in days to ANC Recovery equals to 0 days.

Programming notes: Note to add the unit (Day) after "Statistics";

Similar tables as Table 14.3.3.1:

### Table 14.3.9.3 Time in days to ANC Recovery Post Nadir for Cycle 2-4 and All Treatment Periods– FAS

Note: Missing ANC values within the first 13 days of a cycle will be imputed using the method specified in SAP.

ANC recovery is defined as an ANC  $\geq 2.0 \times 10^9 / L$  after the expected ANC nadir.

Nadir is the lowest ANC value observed in the first 13 days of a cycle.

If nadir point of ANC  $< 2.0 \times 10^9$ /L during the first 13 days of a cycle, then time in days to ANC Recovery = (Start Date when ANC  $\ge 2.0 \times 10^9$ /L) - (Date of nadir in this cycle) + 1

If ANC  $\ge 2.0 \times 10^9$ /L during the first 13 days of a cycle, then time in days to ANC Recovery equals to 0 days.

## Table 14.3.9.4 Time in days to ANC Recovery Post Nadir for Cycle 2-4 and All Treatment Periods – PP Analysis Set B

Note: Missing ANC values within the first 13 days of a cycle will be imputed using the method specified in SAP.

ANC recovery is defined as an ANC  $\geq 2.0 \times 10^9 / L$  after the expected ANC nadir.

Nadir is the lowest ANC value observed in the first 13 days of a cycle.

If nadir point of ANC  $< 2.0 \times 10^9/L$  during the first 13 days of a cycle , then time in days to ANC Recovery = (Start Date when ANC  $\ge 2.0 \times 10^9/L$ ) - (Date of nadir in this cycle) +

If ANC  $\ge 2.0 \times 10^9$ /L during the first 13 days of a cycle, then time in days to ANC Recovery equals to 0 days.

|---|---|---|

Programming notes: Note to add the unit (Day) after "Statistics";

| Generon (Shanghai) Corporation Ltd. SP11631 1.0, 2020-03-11 |
|-------------------------------------------------------------|
|-------------------------------------------------------------|

Table 14.4.1 Immunogenicity Results of F-627- Immunogenicity Analysis Set

| | | Binding<br>n (% | - | | atory assay <sup>[2]</sup> | | ation assay <sup>[3]</sup> | | nclusion<br>n (%) |
|---|---|---|---|---|---|---|---|---|---|
| Treatement<br>Group | Visit | Negative | Positive | Negative | Positive | Negative | Positive | Negative <sup>[4]</sup> | Positive <sup>[5]</sup> |
| F-627 (N = xx) | | | | | | | | | |
| | Day 1 of Cycle 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx(xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Day 1 of Cycle 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Day 1 of Cycle 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Data Source: Data Listing 16.x.x.x

Note: Immunogenicity analysis set (IMAS) is defined as all subjects who receive at least one dose of F627 and have at least one result of serum anti-F-627 antibody collected after treatment of F-627.

Binding assay is conducted in all samples. Confirmatory assay is conducted in these samples with positive results in binding assay. Neutralization assay is conducted in these samples with positive results in confirmatory assay. A positive conclusions will be displayed only for the samples with positive results in neutralization assay.

- [1] Positive (or Negative) rate in Binding assay (%) = number of subjects with positive (or negative) results in binding assay / all subjects in binding assay;
- [2] Positive (or Negative) rate in Confirmatory assay (%) = number of subjects with positive (or negative) results in confirmatory assay / number of subjects with positive results in binding assay :
- [3] Positive (or Negative) rate in Neutralization assay (%) = number of subjects with positive (or negative) results in neutralization assay / number of subjects with positive results in confirmatory assay;
- [4] Positive rate in Conclusion (%) = number of subjects with positive results in neutralization assay / all subjects in Binding assay;
- [5] Negative rate in Conclusion (%) = number of subjects with negative results in any assay / all subjects in Binding assay = 1- Positive rate in Conclusion (%).

Programming notes: Visit point for Immunogenicity test: day 1 of each Cycle, day 21 of Cycle 4, 90 days (±7days) after last visit (day 21 of Cycle 4).

|---|---|---|

| Sponsor: General (Shanghai) Corporation Ltd | Protocol Number : | Version, date : |
|---|---|---|
| Generon (Shanghai) Corporation Ltd. | SP11631 | 1.0, 2020-03-11 |

Table 14.5.1.1 Adverse Events – Safety Analysis Set

| | F-627 | $GRAN^{\scriptscriptstyle{\circledR}}$ | Total |
|---|---|---|---|
| | (N = xx) | (N = xx) | (N = xx) |
| Category of Adverse Event | n(%) NE | n (%) NE | n(%) NE |
| $AEs^{[1]}$ | xx(xx.x) xx | xx(xx.x) xx | xx(xx.x) xx |
| TEAEs <sup>[2]</sup> | xx(xx.x) xx | xx(xx.x) xx | xx(xx.x) xx |
| Study-drug-related TEAEs [3] | xx(xx.x) $xx$ | xx(xx.x) $xx$ | xx(xx.x) $xx$ |
| Any TEAE with CTCAE grade 3 or higher <sup>[4]</sup> | xx(xx.x) xx | xx(xx.x) xx | xx(xx.x) xx |
| Any study drug-related TEAE with CTCAE grade 3 or higher | xx(xx.x) xx | xx(xx.x) xx | xx(xx.x) xx |
| Any TEAE leading to discontinuation of study drug | xx(xx.x) xx | xx(xx.x) $xx$ | xx(xx.x) xx |
| SAE <sup>[5]</sup> | xx(xx.x) xx | xx(xx.x) xx | xx(xx.x) xx |
| Any study drug-related SAE | xx(xx.x) xx | xx(xx.x) xx | xx(xx.x) $xx$ |
| Any study drug-related SAE with CTCAE grade 3 or higher | xx(xx.x) $xx$ | xx(xx.x) $xx$ | xx(xx.x) xx |
| Death | xx(xx.x) xx | xx(xx.x) $xx$ | xx(xx.x) xx |

Data Source: Data Listing 16.x.x.x

Note: Percentages are based on the number of subjects from Safety Analysis Set in each treatment group.

- [1] AE = Adverse Event.
- [2] Treatment-emergent adverse event (TEAE) is defined as any adverse event that onset, or worsens in severity on or after the date of first chemotherapy.
- [3] AEs with causality of "Certainly related", "Probably related" and "Possibly related"are categorized to "Related".
- [4] All AEs grade will be assessed with the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
- [5] SAE = Serious Adverse Event.

Programming notes: Subjects will be counted only once when the subject experienced more than one TEAE within each SOC and PT; Subjects will be counted only once for each system organ class and preferred term by selecting the most severe event;

Subjects will be counted only once for each system organ class and preferred term by selecting the most related event.

Those TEAEs with same system organ class and preferred term but having different start date will be considered as different TEAEs.

| Sponsor :<br>Generon (Shanghai) Corporation Ltd. | Protocol Number :<br>SP11631 | Version, date: 1.0, 2020-03-11 |
|---|---|---|

Table 14.5.1.2 Adverse Events by Causality with study drug – Safety Analysis Set

| | F-627 | GRAN® | Total |
|---------------------------|----------|----------|----------|
| | (N = xx) | (N = xx) | (N = xx) |
| Causality with study drug | n(%) | n(%) | n(%) |
| Unrelated | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Unlikely related | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Possibly related | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Probably related | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Definitely related | xx(xx.x) | xx(xx.x) | xx(xx.x) |

Data Source: Data Listing 16.x.x.x

Note: Percentages are based on the number of subjects from Safety Analysis Set in each treatment group.

| Sponsor : Protocol Number : SP11631 | Version, date : 1.0, 2020-03-11 |
|-------------------------------------|---------------------------------|
|-------------------------------------|---------------------------------|

Table 14.5.1.3 TEAEs by System Organ Class and Preferred Term – Safety Analysis Set

| MedDRA System Organ Class | F-627 | $GRAN^{	ext{@}}$ | Total |
|------------------------------|----------|------------------|----------|
| Preferred Term | (N = xx) | (N = xx) | (N = xx) |
| | n (%) | n (%) | n (%) |
| ΓΕ <b>Α</b> Ε <sup>[1]</sup> | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| <soc #1=""></soc> | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| <pt #1-1=""></pt> | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| <pt #1-2=""></pt> | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| ••••• | | | |
| <soc #2=""></soc> | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| <pt #2-1=""></pt> | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| <pt #2-2=""></pt> | xx(xx,x) | xx(xx.x) | xx(xx.x) |

Data Source: Data Listing 16.x.x.x

Note: Percentages are based on the number of subjects from Safety Analysis Set in each treatment group.

Programming notes: Subjects will be counted only once when the subject experienced more than one TEAE within each SOC and PT; Subjects will be counted only once for each system organ class and preferred term by selecting the most severe event;

<sup>[1]</sup> Treatment-emergent adverse event (TEAE) is defined as any adverse event that onset, or worsens in severity on or after the date of first chemotherapy. Adverse events are coded using MedDRA(Version 22.1).

|---|---|---|

Similar tables as Table 14.5.1.3:

### Table 14.5.1.4 Study Drug Related TEAEs by System Organ Class and Preferred Term - Safety Analysis Set

Data Source: Data Listing 16.x.x.x

Note: Percentages are based on the number of subjects from Safety Analysis Set in each treatment group.

[1] Treatment-emergent adverse event (TEAE) is defined as any adverse event that onset, or worsens in severity on or after the date of first chemotherapy. Adverse events are coded using MedDRA(Version 22.1).

# Table 14.5.1.5 TEAEs with CTCAE Grade 3 or Higher by System Organ Class and Preferred Term - Safety Analysis Set

Data Source: Data Listing 16.x.x.x

Note: Percentages are based on the number of subjects from Safety Analysis Set in each treatment group.

[1] Treatment-emergent adverse event (TEAE) is defined as any adverse event that onset, or worsens in severity on or after the date of first chemotherapy. Adverse events are coded using MedDRA(Version 22.1).

# Table 14.5.1.6 Study Drug Related TEAEs with CTCAE Grade 3 or Higher by System Organ Class and Preferred Term - Safety Analysis Set

Data Source: Data Listing 16.x.x.x

Note: Percentages are based on the number of subjects from Safety Analysis Set in each treatment group.

[1] Treatment-emergent adverse event (TEAE) is defined as any adverse event that onset, or worsens in severity on or after the date of first chemotherapy. Adverse events are coded using MedDRA(Version 22.1).

|-------------------------------------|-------------------|-----------------|
| Generon (Shanghai) Corporation Ltd. | SP11631 | 1.0, 2020-03-11 |

Table 14.5.1.7 TEAEs by System Organ Class and Preferred Term and NCI CTCAE V4.03 Grade - Safety Analysis Set

| | | F-627 | GRAN® | Total |
|---|---|---|---|---|
| MedDRA System Organ Class | NCI CTCAE V4.03 grade | (N = xx) | (N = xx) | (N = xx) |
| Preferred Term | | n (%) | n (%) | n (%) |
| TEAE | Total | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Grade 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Grade 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Grade 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Grade 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Grade 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| <soc #1=""></soc> | Total | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Grade 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Grade 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Grade 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Grade 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Grade 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| <pt #1-1=""></pt> | Total | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Grade 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Grade 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Grade 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Grade 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Grade 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| <pt #1-2=""></pt> | Total | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Grade 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Grade 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Grade 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Grade 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Table Shells for Statistical Analyses

|---|---|---|---|
| Grade 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| <soc #2=""></soc> | | | |
| <pt #2-1=""></pt> | | | |
| <pt #2-2=""></pt> | | | |

Data Source: Data Listing 16.x.x.x

Note: Percentages are based on the number of subjects from Safety Analysis Set in each treatment group.

Treatment-emergent adverse event (TEAE) is defined as any adverse event that onset, or worsens in severity on or after the date of first chemotherapy.

Subjects will be counted only once for each system organ class and preferred term by selecting the most severe event;

Adverse events are coded using MedDRA(Version 22.1).

|---|---|---|

Similar tables as Table 14.5.1.7: Replace "TEAE" with "Study drug related TEAE" in row 1.

# Table 14.5.1.8 Study Drug Related TEAEs by System Organ Class and Preferred Term and NCI CTCAE V4.03 Grade - Safety Analysis Set

Data Source: Data Listing 16.x.x.x

Note: Percentages are based on the number of subjects from Safety Analysis Set in each treatment group.

Treatment-emergent adverse event (TEAE) is defined as any adverse event that onset, or worsens in severity on or after the date of first chemotherapy.

Subjects will be counted only once for each system organ class and preferred term by selecting the most severe event;

Adverse events are coded using MedDRA(Version 22.1).

Similar tables as Table 14.5.1.3: Update "TEAE" in row 1 according to the header.

# Table 14.5.1.9 TEAEs leading to Study Drug Withdrawn by System Organ Class and Preferred Term - Safety Analysis Set

Data Source: Data Listing 16.x.x.x

Note: Percentages are based on the number of subjects from Safety Analysis Set in each treatment group.

[1] Treatment-emergent adverse event (TEAE) is defined as any adverse event that onset, or worsens in severity on or after the date of first chemotherapy. Adverse events are coded using MedDRA(Version 22.1).

Programming notes: Only adverse events which action on study drug is "Drug Withdrawn" are summarized in this table...

| Sponsor: | Protocol Number: | Version, date : |
|-------------------------------------|------------------|-----------------|
| Generon (Shanghai) Corporation Ltd. | SP11631 | 1.0, 2020-03-11 |

Table 14.5.1.10 SAE by System Organ Class and Preferred Term - Safety Analysis Set

| MedDRA System Organ Class | F-627 | GRAN® | Total |
|---------------------------|----------|----------|----------|
| Duofamad Tama | (N = xx) | (N = xx) | (N = xx) |
| Preferred Term | n (%) | n (%) | n (%) |
| SAE <sup>[1]</sup> | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| <soc #1=""></soc> | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| <pt #1-1=""></pt> | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| <pt #1-2=""></pt> | xx(xx.x) | xx(xx.x) | xx(xx.x) |

Data Source: Data Listing 16.x.x.x

Note: Percentages are based on the number of subjects from Safety Analysis Set in each treatment group.

[1] Summary of SAE is based on TEAE. Treatment-emergent adverse event (TEAE) is defined as any adverse event that onset, or worsens in severity on or after the date of first chemotherapy.

Adverse events are coded using MedDRA(Version 22.1).

Similar tables as Table 14.5.1.3: Update "TEAE" in row 1 according to the header.

### Table 14.5.1.11 Death by System Organ Class and Preferred Term - Safety Analysis Set

Data Source: Data Listing 16.x.x.x

Note: Percentages are based on the number of subjects from Safety Analysis Set in each treatment group.

[1] Summary of death is based on TEAE. Treatment-emergent adverse event (TEAE) is defined as any adverse event that onset, or worsens in severity on or after the date of first chemotherapy.

Adverse events are coded using MedDRA(Version 22.1).

### Table 14.5.1.12 TEAEs with Incidence > 5% by System Organ Class and Preferred Term - Safety Analysis Set

Data Source: Data Listing 16.x.x.x

Note: Percentages are based on the number of subjects from Safety Analysis Set in each treatment group.

[1] Treatment-emergent adverse event (TEAE) is defined as any adverse event that onset, or worsens in severity on or after the date of first chemotherapy.

Adverse events are coded using MedDRA(Version 22.1).

| Sponsor: | Protocol Number: | Version, date : |
|-------------------------------------|------------------|-----------------|
| Generon (Shanghai) Corporation Ltd. | SP11631 | 1.0, 2020-03-11 |

Table 14.5.2.1.1 Summary of Hematology Results-Safety Analysis Set

| | F-627 | GRAN® | Total |
|----------------------|--------------|--------------|--------------|
| | (N = xx) | (N = xx) | (N = xx) |
| Baseline of cycle xx | | | |
| n(missing) | XX(XX) | xx(xx) | XX(XX) |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Min , Max | xx - xx | xx - xx | xx - xx |
| Day xx of cycle xx | | | |
| n(missing) | XX(XX) | xx(xx) | XX(XX) |

| Willi, Iviax | $\Lambda\Lambda - \Lambda\Lambda$ | AA - AA | $\lambda \lambda - \lambda \lambda$ |
|---|---|---|---|
| Day xx of cycle xx | | | |
| n(missing) | XX(XX) | xx(xx) | XX(XX) |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Min, Max | xx - xx | xx - xx | xx - xx |
| Change from Baseline | | | |
| n(missing) | xx(xx) | XX(XX) | XX(XX) |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Min, Max | xx - xx | xx - xx | xx - xx |

Day xx of cycle xx

Data Source: Data Listing 16.x.x.x

<Hematology Parameter (unit)>

Note: For hematology parameter, baseline of cycle 1 is defined as the last valid value on or prior to the first date of chemotherapy. The baseline of each cycle in cycle 2-4 is defined as the last valid value on or within 3 days prior to the first date of chemotherapy of each cycle.

Programming notes: 1. For hematology parameter, "Day 1 of cycle xx" is not as a analysis visit, its value is included in the baseline analysis of each cycle. Visits not specified in the study flow chart will not be summarized in table.

- 2. Repeat for all hematology parameter: White blood cell count (10^9/L), Neutrophil count (10^9/L), Eosinophil count (10^9/L), Basophil count (10^9/L) etc.
- 3. Please use "Baseline of cycle xx" for baseline of each cycle.

|---|---|---|
|---|---|---|

Table 14.5.2.1.2 Category of Hematology Results by Baseline and Post-Baseline Visit by Cycle – Safety **Analysis Set** 

| <hematolo< th=""><th>m, Paramet</th><th>or (unit)&gt;</th></hematolo<> | m, Paramet | or (unit)> |
|---|---|---|

| | F-627 | GRAN® | Total |
|---|---|---|---|
| | (N = xx) | (N = xx) | (N = xx) |
| | n (%) | n (%) | n (%) |
| Baseline of cycle xx | | | |
| n (missing) | $\mathbf{XX}(\mathbf{xx})$ | XX(xx) | $\mathbf{x}\mathbf{x}(\mathbf{x}\mathbf{x})$ |
| High | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Normal | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Low | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Day xx of cycle xx | | | |
| n (missing) | xx(xx) | xx(xx) | xx(xx) |
| High | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Normal | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Low | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |

Data Source: Data Listing 16.x.x.x

Note: For hematology parameter, baseline of cycle 1 is defined as the last valid value on or prior to the first date of chemotherapy. The baseline of each cycle in cycle 2-4 is defined as the last valid value on or within 3 days prior to the first date of chemotherapy of each cycle.

Percentages are based on the number of non-missing subjects from Safety Analysis Set at each visit in each treatment group.

Programming notes: 1. For hematology parameter, "Day 1 of cycle xx" is not as a analysis visit, its value is included in the baseline analysis of each cycle. Visits not specified in the study flow chart will not be summarized in table.

- 2.Repeat for all hematology parameters: White blood cell count (10^9/L), Neutrophil count (10^9/L), Eosinophil count (10^9/L), Basophil count (10^9/L) etc.
- 3. Please use "Baseline of cycle xx" for baseline of each cycle.

|-------------------------------------|-------------------|-----------------|
| Generon (Shanghai) Corporation Ltd. | SP11631 | 1.0, 2020-03-11 |

Similar tables as Table 14.5.2.1.1:

#### Table 14.5.2.2.1 Summary of Clinical Chemistry Results – Safety Analysis Set

Data Source: Data Listing 16.x.x.x

Note: Baseline is defined as the last valid value on or prior to the first date of chemotherapy during all treatment periods.

#### Programming notes:

- 1. Visits not specified in the study flow chart will not be summarized in table.
- 2. Repeat for all clinical chemistry parameters. Please note that urea will be directly converted to urea nitrogen in table, and the value and unit can be directly converted. But no transformation in listing.
- 3.For laboratory examinations (except for Hematology) and other examinations (physical examination, electrocardiogram, etc.), "Day 1 of cycle 1" is not as a analysis visit for separate summary, its value is included in the baseline analysis according to the baseline definition, but Day 1 of cycle 2-4 will be summarized as analysis visit. The following is the same

Similar tables as Table 14.5.2.1.2:

### Table 14.5.2.2.2 Category of Clinical Chemistry Results by Baseline and Post-Baseline Visit – Safety Analysis Set

Data Source: Data Listing 16.x.x.x

Note: Baseline is defined as the last valid value on or prior to the first date of chemotherapy during all treatment periods.

Percentages are based on the number of non-missing subjects from Safety Analysis Set at each visit in each treatment group.

#### Programming notes:

- 1. Visits not specified in the study flow chart will not be summarized in table.
- 2. Repeat for all clinical chemistry parameters. Please note that urea will be directly converted to urea nitrogen in table, and the value and unit can be directly converted. But no transformation in listing.

Similar tables as Table 14.5.2.1.1:

#### Table 14.5.2.3.1 Summary of Urinalysis Quantitative Parameters – Safety Analysis Set

Data Source: Data Listing 16.x.x.x

Note: Baseline is defined as the last valid value on or prior to the first date of chemotherapy during all treatment periods.

#### Programming notes:

- 1. Visits not specified in the study flow chart will not be summarized in table.
- 2. Repeat for all Urinalysis quantitative parameters: Urine specific gravity, PH.

Similar tables as Table 14.5.2.1.2:

#### Table 14.5.2.3.2 Category of Urinalysis Quantitative Parameters Results by Baseline and Post-Baseline Visit –

Table Shells for Statistical Analyses

| Generon (Shanghai) Corporation Ltd. SP11631 1.0, 2020-03-11 | T - | Version, date:<br>1.0, 2020-03-11 |
|---|---|---|
|---|---|---|

### Safety Analysis Set Data Source: Data Listing 16.x.x.x

Note: Baseline is defined as the last valid value on or prior to the first date of chemotherapy during all treatment periods. Percentages are based on the number of non-missing subjects from Safety Analysis Set at each visit in each treatment group.

#### Programming notes:

- 1. Visits not specified in the study flow chart will not be summarized in table.
- 2. Repeat for all Urinalysis quantitative parameters: Urine specific gravity, PH.

| | | D. J. IN. J. | |
|---|---|---|---|
| , | ponsor: | Protocol Number :<br>SP11631 | Version, date :<br>1.0, 2020-03-11 |
| U | eneron (Shanghai) Corporation Ltd. | 3F11031 | 1.0, 2020-03-11 |

# Table 14.5.2.3.3 Category of Urinalysis Qualitative Parameters Results by Baseline and Post-Baseline Visit – Safety Analysis Set

< Urinalysis qualitative parameters (unit) >

| | F-627 | GRAN® | Total |
|---|---|---|---|
| | (N = xx) | (N = xx) | (N = xx) |
| | n (%) | n (%) | n (%) |
| Baseline | | | |
| n (missing) | $\mathbf{XX}(\mathbf{xx})$ | $\mathbf{x}\mathbf{x}(\mathbf{x}\mathbf{x})$ | $\mathbf{x}\mathbf{x}(\mathbf{x}\mathbf{x})$ |
| Negative | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Positive | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Day xx of cycle xx | | | |
| n (missing) | XX(xx) | XX(xx) | XX(XX) |
| Negative | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Positive | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Data Source: Data Listing 16.x.x.x

Note: Baseline is defined as the last valid value before the first chemotherapy during all treatment periods.

Percentages are based on the number of non-missing subjects from Safety Analysis Set at each visit in each treatment group.

#### Programming notes:

- 1. For Urinalysis qualitative parameters, the laboratory test result is Positive or Negative.
- 2. Repeat for all Urinalysis qualitative parameters: Urine protein, Casts, Blood cells (qualitative), Urine WBC (qualitative), Urine glucose, Urine ketones.
- 3.Please note that Urine RBC (microscopic examination) and Urine WBC (microscopic examination) will be only displayed in listing, not be summaried in table
- 4. Visits not specified in the study flow chart will not be summarized in table.

|-------------------------------------|-------------------|-----------------|
| Generon (Shanghai) Corporation Ltd. | SP11631 | 1.0, 2020-03-11 |

### Table 14.5.2.3.4 Summary of Urinalysis Clinical Evaluation by Baseline and Post-Baseline Visit – Safety **Analysis Set**

< Urinalysis parameters (unit) >

| | F-627 | GRAN® | Total |
|---|---|---|---|
| | (N = xx) | (N = xx) | (N = xx) |
| | n (%) | n (%) | n (%) |
| Baseline | | | |
| n (missing) | $\mathbf{x}\mathbf{x}(\mathbf{x}\mathbf{x})$ | $\mathbf{XX}(\mathbf{XX})$ | $\mathbf{x}\mathbf{x}(\mathbf{x}\mathbf{x})$ |
| Normal | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Abnormal without clinical significance | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Abnormal with clinical significance | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not examined | xx(xx.x) | xx (xx.x) | xx (xx.x) |
| Day xx of cycle xx | | | |
| n (missing) | $\mathbf{x}\mathbf{x}(\mathbf{x}\mathbf{x})$ | XX(XX) | $\mathbf{XX}(\mathbf{xx})$ |
| Normal | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Abnormal without clinical significance | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Abnormal with clinical significance | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not examined | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Data Source: Data Listing 16.x.x.x

Note: Baseline is defined as the last valid value on or prior to the first date of chemotherapy during all treatment periods.

Percentages are based on the number of non-missing subjects from Safety Analysis Set at each visit in each treatment group.

<sup>1.</sup> For Urinalysis parameters (Quantitative / Qualitative Parameters), the clinical evaluation result is Normal, Abnormal without clinical significance, Abnormal with clinical significance.

<sup>2.</sup> Please note that Urine RBC (microscopic examination) and Urine WBC (microscopic examination) will be only displayed in listing, not be summaried in table.

<sup>3.</sup> Visits not specified in the study flow chart will not be summarized in table.

| Sponsor :<br>Generon (Shanghai) Corporation Ltd. | Protocol Number :<br>SP11631 | Version, date: 1.0, 2020-03-11 |
|---|---|---|

Table 14.5.3.1 Vital Signs and Weight – Safety Analysis Set

| < Vital Signs | Parameter | (unit | )> |
|---------------|-----------|-------|----|
|---------------|-----------|-------|----|

| | F-627 | $GRAN^{\scriptscriptstyle{\circledR}}$ | Total |
|---|---|---|---|
| <vital (unit)="" parameter="" signs=""></vital> | (N = xx) | (N = xx) | (N = xx) |
| Baseline | | | |
| n(missing) | XX(XX) | XX(XX) | XX(XX) |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Min , Max | xx-xx | XX-XX | xx-xx |
| Day xx of cycle xx | | | |
| n(missing) | XX(XX) | xx(xx) | XX(XX) |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Min, Max | XX-XX | XX-XX | XX-XX |
| Change from Baseline | | | |
| n(missing) | xx(xx) | xx(xx) | xx(xx) |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Min, Max | XX-XX | XX-XX | xx-xx |

Data Source: Data Listing 16.x.x.x.

Note: Baseline is defined as the last valid value on or prior to the first date of chemotherapy during all treatment periods.

Programming notes: Repeat for all Vital Signs parameters: : Heart rate (beats/minute), Systolic pressure (mmHg), Diastolic pressure (mmHg), Weight(kg).

| Sponsor : Protocol Number : SP11631 | Version, date : 1.0, 2020-03-11 |
|-------------------------------------|---------------------------------|
|-------------------------------------|---------------------------------|

Table 14.5.3.2 Body Temperature Results – Safety Analysis Set

| | F-627 | GRAN® | Total |
|-----------------------|-------------|-------------|-------------|
| Body Temperature (°C) | (N = xx) | (N = xx) | (N = xx) |
| Baseline | | | |
| n(missing) | XX(XX) | XX(XX) | XX(XX) |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Min , Max | xx-xx | xx-xx | XX-XX |
| Day xx of cycle xx | | | |
| n(missing) | XX(XX) | xx(xx) | XX(XX) |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Min, Max | XX-XX | XX-XX | XX-XX |
| Change from Baseline | | | |
| n(missing) | xx(xx) | XX(XX) | XX(XX) |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Min, Max | XX-XX | XX-XX | xx-xx |

Data Source: Data Listing 16.x.x.x.

Note: Baseline is defined as the last valid value on or prior to the first date of chemotherapy during all treatment periods.

|---|---|---|

Table 14.5.3.3.1 Physical Examination – Safety Analysis Set

| - ware - were to the - my shown | 200100, 1111001, 515 200 | | |
|---|---|---|---|
| * | F-627 | GRAN® | Total |
| <physical examination="" parameter=""></physical> | (N = xx) | (N = xx) | (N = xx) |
| | n (%) | n (%) | n (%) |
| Baseline | | | |
| n (missing) | XX(XX) | $\mathbf{x}\mathbf{x}(\mathbf{x}\mathbf{x})$ | $\mathbf{XX}(\mathbf{XX})$ |
| Normal | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Abnormal without clinical significance | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Abnormal with clinical significance | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not examined | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Day xx of cycle xx | | | |
| n (missing) | $\mathbf{XX}(\mathbf{XX})$ | XX(xx) | $\mathbf{x}\mathbf{x}(\mathbf{x}\mathbf{x})$ |
| Normal | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Abnormal without clinical significance | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Abnormal with clinical significance | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not examined | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Data Source: Data Listing 16.x.x.x

Note: Baseline is defined as the last valid value on or prior to the first date of chemotherapy during all treatment periods. Percentages are based on the number of non-missing subjects from Safety Analysis Set at each visit in each treatment group.

Programming notes: Repeat for all Physical Examination parameters: General conditions, Lymph nodes, Skin, etc.

|--|--|---|---|---|
|--|--|---|---|---|

Table 14.5.3.3.2 Shift Change of Physical Examination from Baseline to Post-Baseline – Safety Analysis Set

| | | | | | | Results of Baseline | | |
|---|---|---|---|---|---|---|---|---|
| | Physical | Visit | | - | | n (%) | Not | Total |
| | Examination | | Results of Post- | | Abnormal without | Abnormal with | examined | |
| Treatement Group | parameter | | Baseline | Normal | clinical significance | clinical significance | | |
| | General | Day xx of cycle xx | | | | | | |
| F-627 (N=xx) | conditions | | Normal | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| | | | Abnormal without | | | | | |
| | | | clinical significance | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| | | | Abnormal with | | | | | |
| | | | clinical significance | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| | | | Not examined | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| | | | Total | x (xx.x) | x (xx.x) | x (xx.x) | x(xx.x) | x (xx.x) |
| | | Day xx of cycle xx | Normal | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| | | | Abnormal without | | | | | |
| | | | clinical significance | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| | | | Abnormal with | | | | | |
| | | | clinical significance | x (xx.x) | x (xx.x) | x(xx.x) | x (xx.x) | x (xx.x) |
| | | | Not examined | x (xx.x) | x(xx.x) | x(xx.x) | x (xx.x) | x (xx.x) |
| | | | Total | x(xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |

Skin

Day xx of cycle xx

 $GRAN \circledR \ (N=xx)$ 

Data Source: Data Listing 16.x.x.x

Note: Baseline is defined as the last valid value on or prior to the first date of chemotherapy during all treatment periods. Percentages are based on the number of non-missing subjects from Safety Analysis Set at each visit in each treatment group.

Programming notes: Repeat for all Physical Examination parameters: General conditions, Lymph nodes, Skin, etc.

|-------------------------------------|-------------------|-----------------|
| Generon (Shanghai) Corporation Ltd. | SP11631 | 1.0, 2020-03-11 |

Table 14.5.4.1 12-Lead ECG – Safety Analysis Set

| | F-627 | $GRAN^{	ext{@}}$ | Total |
|---|---|---|---|
| <12-Lead ECG Parameter> | (N = xx) | (N = xx) | (N = xx) |
| Baseline | | , , , | , |
| n(missing) | XX(XX) | XX(XX) | XX(XX) |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Min, Max | XX-XX | XX-XX | xx-xx |
| Day xx of cycle xx | | | |
| n(missing) | XX(XX) | xx(xx) | XX(XX) |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Min, Max | XX-XX | XX-XX | XX-XX |
| Change from Baseline | | | |
| n(missing) | XX(XX) | xx(xx) | xx(xx) |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Min, Max | XX-XX | XX-XX | XX-XX |

Data Source: Data Listing 16.x.x.x.

Note: Baseline is defined as the last valid value on or prior to the first date of chemotherapy during all treatment periods.

Programming notes: Repeat for following 12-Lead ECG Parameter: (Heart rate, PR Interval, QRS Interval, QT Interval, QTc)

|---|
| ı |

Table 14.5.4.2 12-Lead ECG Results in Clinical Evaluation—Safety Analysis Set

| | F-627 | GRAN® | Total |
|---|---|---|---|
| 12-Lead ECG | (N = xx) | (N = xx) | (N = xx) |
| 12-Lead ECG | n (%) | n (%) | n (%) |
| Baseline | | | |
| n (missing) | $\mathbf{x}\mathbf{x}(\mathbf{x}\mathbf{x})$ | $\mathbf{x}\mathbf{x}(\mathbf{x}\mathbf{x})$ | $\mathbf{x}\mathbf{x}(\mathbf{x}\mathbf{x})$ |
| Normal | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Abnormal without clinical significance | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Abnormal with clinical significance | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Day xx of cycle xx | | | |
| n (missing) | $\mathbf{XX}(\mathbf{xx})$ | $\mathbf{XX}(\mathbf{xx})$ | $\mathbf{x}\mathbf{x}(\mathbf{x}\mathbf{x})$ |
| Normal | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Abnormal without clinical significance | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Abnormal with clinical significance | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Data Source: Data Listing 16.x.x.x

Note: Baseline is defined as the last valid value on or prior to the first date of chemotherapy during all treatment periods.

Percentages are based on the number of non-missing subjects from Safety Analysis Set at each visit in each treatment group.

| Sponsor: Generon (Shanghai) Corporation Ltd | Protocol Number :<br>SP11631 | Version, date : |
|---|---|---|
| Generon (Shanghai) Corporation Ltd. | SP11631 | 1.0, 2020-03-11 |

Table 14.5.4.3 Shift Change of 12-Lead ECG Results in Clinical Evaluation from Baseline to Post-Baseline – Safety Analysis Set

| | | | | | Results of Baseline | | |
|---|---|---|---|---|---|---|---|
| Treatement Group | Visit | Results of Post-Baseline | Normal | Abnormal without clinical significance | n (%) Abnormal with clinical significance | Not examined | Total |
| F-627 (N=xx) | Day xx of cycle xx | Normal Abnormal without | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| | | clinical significance<br>Abnormal with clinical | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| | | significance | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| | | Not examined | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| | | Total | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| | Day xx of cycle xx | Normal<br>Abnormal without | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| | | clinical significance<br>Abnormal with clinical | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| | | significance | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| | | Not examined | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| | | Total | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| | 00000 | | | | | | |

000000

Day xx of cycle xx

 $GRAN \circledR \ (N=xx)$ 

Data Source: Data Listing 16.x.x.x

Note: Baseline is defined as the last valid value on or prior to the first date of chemotherapy during all treatment periods.

Percentages are based on the number of non-missing subjects from Safety Analysis Set at each visit in each treatment group.

| Sponsor: Generon (Shanghai) Corporation Ltd | Protocol Number :<br>SP11631 | Version, date : |
|---|---|---|
| Generon (Shanghai) Corporation Ltd. | SP11631 | 1.0, 2020-03-11 |

Table 14.5.4.4 QTc ECG Results – Safety Analysis Set

| | F-627 | GRAN® | Total |
|------------------------------|-----------|-----------|-----------|
| 12-Lead ECG QTC Interval | (N = xx) | (N = xx) | (N = xx) |
| 12-Lead ECG QTC Illierval | n (%) | n (%) | n (%) |
| Baseline | | | |
| n (missing) | xx (xx) | xx (xx) | xx (xx) |
| >450 msec | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >480 msec | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >500 msec | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Change from baseline>30 msec | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Change from baseline>60 msec | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Change from baseline>90 msec | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Day xx of cycle xx | | | |
| n (missing) | xx (xx) | xx (xx) | xx (xx) |
| >450 msec | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >480 msec | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >500 msec | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Change from baseline>30 msec | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Change from baseline>60 msec | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Change from baseline>90 msec | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Data Source: Data Listing 16.x.x.x

Note: Baseline is defined as the last valid value on or prior to the first date of chemotherapy during all treatment periods.

Percentages are based on the number of non-missing subjects from Safety Analysis Set at each visit in each treatment group.

|-------------------------------------|-------------------|-----------------|
| Generon (Shanghai) Corporation Ltd. | SP11631 | 1.0, 2020-03-11 |

Table 14.5.5.1 Results of Abdominal Ultrasound - Safety Analysis Set

| | F-627 | GRAN® | Total |
|---|---|---|---|
| Abdominal Ultrasound | (N = xx) | (N = xx) | (N = xx) |
| | n (%) | n (%) | n (%) |
| Baseline | | | |
| n (missing) | $\mathbf{x}\mathbf{x}(\mathbf{x}\mathbf{x})$ | XX(XX) | $\mathbf{XX}(\mathbf{XX})$ |
| Normal | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Abnormal without clinical significance | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Abnormal with clinical significance | xx(xx.x) | xx (xx.x) | xx (xx.x) |
| Day xx of cycle xx | | | |
| n (missing) | $\mathbf{XX}(\mathbf{xx})$ | $\mathbf{XX}(\mathbf{xx})$ | $\mathbf{XX}(\mathbf{XX})$ |
| Normal | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Abnormal without clinical significance | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Abnormal with clinical significance | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Data Source: Data Listing 16.x.x.x.

Note: Baseline is defined as the last valid value on or prior to the first date of chemotherapy during all treatment periods. Percentages are based on the number of non-missing subjects from Safety Analysis Set at each visit in each treatment group.

Programming note: Visits of Abdominal Ultrasound : Baseline, End of study.

|-------------------------------------|-------------------|-----------------|
| Generon (Shanghai) Corporation Ltd. | SP11631 | 1.0, 2020-03-11 |

Table 14.5.5.2 Shift Change of Abdominal Ultrasound from Baseline to Post-Baseline - Safety Analysis Set

| | | | Results of Baseline n (%) | | | | |
|---|---|---|---|---|---|---|---|
| Treatement Group | Visit | Results of Post-Baseline | Normal | Abnormal without clinical significance | Abnormal with clinical significance | Not examined | Total |
| 7-627 (N=xx) | Day xx of cycle xx | Normal<br>Abnormal without | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| | | clinical significance<br>Abnormal with clinical | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| | | significance | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| | | Not examined | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| | | Total | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| | Day xx of cycle xx | Normal<br>Abnormal without | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| | | clinical significance<br>Abnormal with clinical | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| | | significance | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| | | Not examined | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| | | Total | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |

000000

Day xx of cycle xx

GRAN® (N=xx)

Data Source: Data Listing 16.x.x.x.

Note: Baseline is defined as the last valid value on or prior to the first date of chemotherapy during all treatment periods.

Percentages are based on the number of non-missing subjects from Safety Analysis Set at each visit in each treatment group.

h visit in each treatment group.

|---|---|---|

Listing 16.1.7.1 Enrollment Information and Randomization – All Subjects

| Subject ID | Is the subject eligible for enrollment? (If no, please specify) | Was the subject randomized? (If no, please specify) | Date of randomization | Random no. | Treatement<br>Group |
|---|---|---|---|---|---|
| XXXXXX | Yes | Yes | YYYY-MM-DD | | F-627 |
| XXXXXX | Yes | No | YYYY-MM-DD | | $GRAN^{\circledR}$ |
| XXXXXX | No, xxx | No, xxx | YYYY-MM-DD | | GRAN® |
| XXXXXX | Yes | Yes | YYYY-MM-DD | | F-627 |

Listing 16.2.1.1 Disposition of Subjects –Randomized Subjects

| Treatement Group | Subject ID | Received study drug at least once | Complete the study | Completion or Withdrawal Date | Reason for withdrawal |
|---|---|---|---|---|---|
| F-627 | xxxxxx | Yes | Yes | YYYY-MM-DD | |
| GRAN® | xxxxxx | Yes | No | YYYY-MM-DD | Adverse Event |
| GRAN® | xxxxxx | No | No | YYYY-MM-DD | Adverse Event |
| F-627 | xxxxxx | Yes | Yes | YYYY-MM-DD | |

 $Programming\ notes:\ If\ the\ reason\ for\ with drawal\ is\ ``Adverse\ Event",\ please\ add\ AE\ Reported\ Term\ or\ symptom.$ 

|---|---|---|

Listing 16.2.1.2 Withdrawal from Study-Randomized Subjects

| Treatement Group | Subject ID | Received study drug at least once | Withdrawal Date | Reason for withdrawal |
|---|---|---|---|---|
| F-627 | xxxxxx | Yes | YYYY-MM-DD | Adverse Event |
| GRAN® | xxxxxx | Yes | YYYY-MM-DD | Adverse Event |
| GRAN® | xxxxxx | Yes | YYYY-MM-DD | Adverse Event |
| F-627 | xxxxxx | Yes | YYYY-MM-DD | Adverse Event |

Programming notes: If the reason for withdrawal is "Adverse Event", please add AE Reported Term or symptom.

| Sponsor: | Protocol Number: | Version, date : |
|-------------------------------------|------------------|-----------------|
| Generon (Shanghai) Corporation Ltd. | SP11631 | 1.0, 2020-03-11 |

Listing 16.2.1.3.1 Analysis Sets-Randomized Subjects

| Treatement<br>Group | Subject ID | Full Analysis Set (FAS) | PP Analysis Set A | PP Analysis Set B | Safety<br>Set | Analysis Immunogenicity analysis set |
|---|---|---|---|---|---|---|
| F-627 | xxxxxx | Yes | Yes | Yes | Yes | Yes |
| GRAN® | xxxxxx | Yes | Yes | No | Yes | Yes |
| GRAN® | xxxxxx | Yes | Yes | Yes | No | No |
| F-627 | xxxxxx | Yes | Yes | Yes | Yes | Yes |

Listing 16.2.1.3.2 Reasons for Subjects Excluded from FAS/SS/PP Set – Randomized Subjects

| Treatement<br>Group | Subject<br>ID | FAS | Reason Excluded from FAS | SS | Reason Excluded from SS | PP Set A | Reason Excluded from PP Set A | PP Set B | Reason Excluded from PP Set B |
|---|---|---|---|---|---|---|---|---|---|
| F-627 | xxxxxx | | | | | | | | |
| $GRAN^{\mathbb{R}}$ | XXXXXX | | | | | | | | |
| GRAN® | XXXXXX | | | | | | | | |
| F-627 | XXXXXX | | | | | | | | |

|-------------------------------------|-------------------|-----------------|
| Generon (Shanghai) Corporation Ltd. | SP11631 | 1.0, 2020-03-11 |

Listing 16.2.1.4 Major Protocol Deviations—Randomized Subjects

| Treatement Group | Subject ID | Phase | Category | Description |
|---------------------|------------|---------|----------|-------------|
| F-627 | xxxxxx | Screen | xxxxxxxx | xxxxxxxx |
| $GRAN^{\mathbb{R}}$ | xxxxxx | Cycle 1 | xxxxxxxx | xxxxxxxx |
| GRAN® | xxxxxx | Cycle 1 | xxxxxxxx | xxxxxxxx |
| F-627 | xxxxxx | Cycle 2 | xxxxxxxx | xxxxxxxx |

Programming notes: Phase of Protocol Deviations: Screen, Cycle 1, Cycle 2, Cycle 3, Cycle 4

|---|---|---|

**Listing 16.2.1.5 Protocol Deviations— Randomized Subjects** 

| Treatement Group | Subject ID | Phase | Category | Description | Severity |
|---|---|---|---|---|---|
| F-627 | XXXXXX | Screen | xxxxxxxx | XXXXXXXX | Major |
| GRAN® | XXXXXX | Cycle 1 | XXXXXXXX | xxxxxxxx | Mild |
| GRAN® | xxxxxx | Cycle 1 | XXXXXXXX | xxxxxxxx | |
| F-627 | XXXXXX | Cycle 2 | xxxxxxxx | xxxxxxxx | |
| ••••• | | | | | |

Programming notes: Phase of Protocol Deviations: Screen, Cycle 1, Cycle 2, Cycle 3, Cycle 4

|---|---|---|
| Generon (Ghanghan) Corporation Eta. | 5111031 | 1.0, 2020-03-11 |

**Listing 16.2.2.1 Demographics – FAS** 

| Treatement<br>Group | Subject ID | Date of Informed Consent | Age (years) | Sex | Natio<br>n | Height (cm) | Weight (kg) | BMI<br>(kg/m²) | Body surface area (m <sup>2</sup> ) |
|---|---|---|---|---|---|---|---|---|---|
| F-627 | xxxxxx | YYYY-MM-DD | XX | Femal | Other | XXX.X | XX.X | XX.X | XX.X |
| GRAN® | XXXXXX | YYYY-MM-DD | XX | Femal | Han | XXX.X | XX.X | XX.X | XX.X |
| GRAN® | xxxxxx | YYYY-MM-DD | XX | Femal | Han | XXX.X | XX.X | XX.X | XX.X |
| F-627 | xxxxxx | YYYY-MM-DD | XX | Femal | Han | XXX.X | XX.X | XX.X | XX.X |

Programming notes: Height and Weight measurements in screening will be used here.
|---|---|
| Generon (Shanghar) corporation Eta. | 1.0, 2020 03 11 |

### Listing 16.2.2.2 Disease Diagnosis, Chemotherapy History, Physical Status – FAS

| Treatement<br>Group | Subject<br>ID | Date of disease diagnosis | Diagnosed with breast cancer | Diagnosed by histopathology | Tumor stage (T,N,M) <sup>[1]</sup> | Tumor<br>clinical<br>stage | Medication<br>history [2] | Date of ECOG performance status | ECOG<br>score |
|---|---|---|---|---|---|---|---|---|---|
| F-627 | xxxxxx | YYYY-MM-DD | Yes | Yes, xxxxxxx | T1,N0,M0 | I | Yes | YYYY-MM-DD | 0 |
| GRAN® | xxxxxx | YYYY-MM-DD | No | No | T1,N1,M0 | IIB | No | YYYY-MM-DD | 1 |
| GRAN® | xxxxxx | YYYY-MM-DD | No | No | T1,N1,M0 | IIB | No | YYYY-MM-DD | 1 |

 $<sup>\</sup>begin{bmatrix} 1 \end{bmatrix} \text{ In tumor clinical stage, } 0 = (\text{Tis, N0, M0}), \text{ IA} = (\text{T1, N0, M0}), \text{ IB} = (\text{T0, N1mi, M0}) \text{ or } (\text{T1, N1, M0}), \text{ IIA} = (\text{T0, N1, M0}) \text{ or } (\text{T1, N1, M0}) \text{ or } (\text{T2, N0, M0}), \text{ IIB} = (\text{T2, N1, M0}) \text{ or } (\text{T3, N0, M0}), \text{ IIB} = (\text{T0, N2, M0}), (\text{T1, N2, M0}), (\text{T2, N2, M0}), (\text{T3, N1 or N2, M0}), \text{ IIB} = (\text{T4, N0 or N1 or N2, M0}), \text{ and IV} = (\text{any T, any N, M1}).$ 

<sup>[2]</sup> Medications refers to drugs taken within 3 months and chemotherapy drugs received within 1 year prior to the date of first chemotherapy.

|---|---|---|

# **Listing 16.2.2.3 History of Surgery–FAS**

| Treatement Group | Subject ID | Date of surgery | MeDRA System Organ Class | Preferred Term | Name of surgery |
|---|---|---|---|---|---|
| F-627 | xxxxxx | YYYY-MM-DD | xxxxxx | xxxxxx | XXXXXX |
| $GRAN^{\scriptscriptstyle{\circledR}}$ | XXXXXX | YYYY-MM-DD | xxxxxx | XXXXXX | XXXXXX |
| $GRAN^{\mathbb{R}}$ | xxxxxx | YYYY-MM-DD | xxxxxx | xxxxxx | xxxxxx |
| F-627 | xxxxxx | YYYY-MM-DD | xxxxxx | xxxxxx | xxxxxx |

Note: Surgery history is coded using MedDRA(Version 22.1).

|---|---|---|

### **Listing 16.2.2.4 Prior / Concomitant Disease – FAS**

| Treatement<br>Group | Subject<br>ID | Disease name | Category for Disease [1] | MedDRA System Organ<br>Class | Preferred<br>Term | Start date | End date |
|---|---|---|---|---|---|---|---|
| F-627 | XXXXXX | xxxxxx | Concomitant disease | XXXXXX | xxxxxx | YYYY-MM-DD | YYYY-MM-DD |
| GRAN® | XXXXXX | XXXXXX | Prior disease | XXXXXX | xxxxxx | YYYY-MM-DD | YYYY-MM-DD |
| GRAN® | XXXXXX | xxxxxx | | XXXXXX | xxxxxx | YYYY-MM-DD | YYYY-MM-DD |
| F-627 | XXXXXX | XXXXXX | | XXXXXX | xxxxxx | YYYY-MM-DD | YYYY-MM-DD |

Note: Prior diseases are coded using MedDRA(Version 22.1).

Prior diseases are these diseases with an end date prior to the date of first chemotherapy. Concomitant diseases are these diseases starting on or after the date of first dose of chemotherapy, or diseases starting prior to the date of first dose of chemotherapy but continuing after the date of first dose of chemotherapy.

| Sponsor : | Protocol Number : | Version, date : |
|-------------------------------------|-------------------|-----------------|
| Generon (Shanghai) Corporation Ltd. | SP11631 | 1.0, 2020-03-11 |

### Listing 16.2.2.5 Cardiac Doppler Ultrasound- FAS

| Treatement Group | Subject ID | Date of examination | Left ventricular ejection fraction (%) | Results | If abnormal, please specify |
|---|---|---|---|---|---|
| F-627 | XXXXXX | YYYY-MM-DD | XX.X | XXXXXX | XXXXXX |
| GRAN® | XXXXXX | YYYY-MM-DD | XX.X | XXXXXX | XXXXXX |
| GRAN® | xxxxxx | YYYY-MM-DD | XX.X | xxxxxx | xxxxxx |
| F-627 | XXXXXX | YYYY-MM-DD | XX.X | xxxxxx | xxxxxx |
| | •••• | | | | |

|--|--|---|---|---|
|--|--|---|---|---|

### Listing 16.2.2.6 Chest (Lateral) Examination- FAS

| Treatement Group | Subject ID | Date of examination | Results | If abnormal, please specify |
|---|---|---|---|---|
| F-627 | XXXXXX | YYYY-MM-DD | Normal | XXXXXX |
| GRAN® | xxxxxx | YYYY-MM-DD | Normal | xxxxxx |
| GRAN® | xxxxxx | YYYY-MM-DD | Abnormal without clinical | XXXXXX |
| F-627 | xxxxxx | YYYY-MM-DD | Normal | XXXXXX |

|---|---|---|

### **Listing 16.2.2.7 Concomitant medications – FAS**

| Treatement | Subject | Category for | Drugs' generic | ATC II/ Preferred | Indication | Reasons | Single dose | Dosing | Route of | Start date / End |
|---|---|---|---|---|---|---|---|---|---|---|
| Group | ID | Medication [1] | names | Name | | for use | / unit | frequency <sup>[2]</sup> | administration | date |
| F-627 | xxxxxx | Prior medications | xxxxxx | xxxxxx/ xxxxxx | xxxxxx | xxxxxx | xxxxxx | QD | IM | YYYY-MM-DD/<br>YYYY-MM-DD |
| GRAN® | xxxxxx | Prior medications | xxxxxx | xxxxxx/ xxxxxx | xxxxxx | xxxxxx | xxxxxx | BID | IV | YYYY-MM-DD/<br>YYYY-MM-DD |
| GRAN® | xxxxxx | Concomitant medications | xxxxxx | xxxxxx/ xxxxxx | xxxxxx | xxxxxx | xxxxxx | ID | IVGTT | YYYY-MM-DD/<br>YYYY-MM-DD |
| F-627 | xxxxxx | Prior medications | xxxxxx | xxxxxx/ xxxxxx | xxxxxx | xxxxxx | xxxxxx | QID | PO | YYYY-MM-DD/<br>YYYY-MM-DD |
| | ••••• | | | | | | | | | |

Note: WHODrug Version B3 September 1, 2019.

<sup>[1]</sup> Prior medications are defined as these medications with an end date on or prior to the date of first chemotherapy. Concomitant medications are these medications other than the study drug used from the date of first chemotherapy to the Day 21 of Cycle 4.

<sup>[2]</sup> QD = One dose daily, BID = Two doses daily, TID = Three doses daily, QID = Four doses daily, QOD = Every other day;

IM = Intramuscular injection, IV = Intravenous injection, IVGTT = Intravenous guttae, PO = Oral administration, TO = Topical.

| Sponsor : Protocol Number : SP11631 | Version, date : 1.0, 2020-03-11 |
|-------------------------------------|---------------------------------|
|-------------------------------------|---------------------------------|

**Listing 16.2.2.8 Concomitant Non-Drug Treatments – FAS** 

| Treatement<br>Group | Subject<br>ID | Type<br>treatment | of MedDRA SOC | Preferred Term | Indication | Reasons for treatment | Start date / End date |
|---|---|---|---|---|---|---|---|
| F-627 | xxxxxx | xxxxxx | xxxxxx | xxxxxx | xxxxxx | xxxxxx | YYYY-MM-DD/<br>YYYY-MM-DD |
| GRAN® | xxxxxx | xxxxxx | xxxxxx | xxxxxx | xxxxxx | xxxxxx | YYYY-MM-DD/<br>YYYY-MM-DD |
| GRAN® | xxxxxx | xxxxxx | xxxxxx | xxxxxx | xxxxxx | xxxxxx | YYYY-MM-DD/<br>YYYY-MM-DD |
| F-627 | xxxxxx | xxxxxx | xxxxxx | xxxxxx | xxxxxx | xxxxxx | YYYY-MM-DD/<br>YYYY-MM-DD |

Note: Concomitant non-drug treatments are coded using MedDRA(Version 22.1).

| Sponsor :<br>Generon (Shanghai) Corporation Ltd. | | ration Ltd. | Protocol Number : SP11631 | | Version, date: 1.0, 2020-03-11 | |
|---|---|---|---|---|---|---|
| Listing 1<br>reatement<br>Group | | | Ficacy Endpoints – FAS Efficacy Endpoints | Re | sults (not imputed) | Results (imputed) |
| F-627 | xxxxxx | Cycle 1 | Duration of Grade 3 or 4 Neutropenia during (day) Duration of Grade 4 Neutropenia (day) Duration of Grade 2 or Higher Neutropenia (day) ANC nadir (10 <sup>9</sup> /L) Time in days to ANC Recovery Post Nadir (day) | | | |
| | | Cycle 2 Cycle 3 Cycle 4 All Treatment periods | Duration of Grade 3 or 4 Neutropenia during (day) | | | |
| GRAN®<br>GRAN®<br>7-627 | XXXXXX<br>XXXXXX<br>XXXXXX | Cycle 1 | | | | |

Note: Method for imputation is specified in SAP.

| Sponsor :<br>Generon (Shanghai) Corporation Ltd. | Protocol Number :<br>SP11631 | Version, date: 1.0, 2020-03-11 |
|---|---|---|

Listing 16.2.3.1 Immunogenicity test of F-627 - Immunogenicity Analysis Set

| Treatement<br>Group | Subject ID | Visit | Date of examination | Binding assay -<br>Bridge enzyme-<br>linked<br>immunosorbent<br>assay | Confirmatory<br>assay - Pre-<br>binding<br>inhibition<br>assay | Neutralization<br>assay - Cell<br>function<br>Neutralization<br>assay | Conclusion Notes |
|---|---|---|---|---|---|---|---|
| F-627 | XXXXXX | Day xx of cycle xx | YYYY-MM-DD | Negative | Negative | Negative | Negative |
| | xxxxxx | Day xx of cycle xx | YYYY-MM-DD | Negative | Negative | Negative | Negative |
| | xxxxxx | Day xx of cycle xx | YYYY-MM-DD | Negative | Negative | Negative | Negative |
| F-627 | xxxxxx | Day xx of cycle xx | YYYY-MM-DD | Positive | Positive | Positive | Positive |
| | ••••• | | | | | | |

|---|---|---|

Listing 16.2.4.1.1 Exposure of Study Drug (F-627, GRAN®) for Cycle 1 – Safety Analysis Set

| Treatement Group | Subject ID | Visit | Dosing date / time | Actual cumulative dose (unit) | Relative dose intensity (RDI) (%) <sup>[1]</sup> |
|---|---|---|---|---|---|
| F-627 | xxxxxx | Day xx of cycle xx | YYYY-MM-DD HH:MM | xxx (mg) | xx.x |
| GRAN® | xxxxxx | Day xx of cycle xx | YYYY-MM-DD HH:MM | xxx (μg) | XX.X |
| GRAN® | xxxxxx | Day xx of cycle xx | YYYY-MM-DD HH:MM | xxx (μg) | XX.X |
| F-627 | xxxxxx | Day xx of cycle xx | YYYY-MM-DD HH:MM | xxx (mg) | XX.X |

Note: [1]Relative dose intensity (%)=(Actual dose intensity / Planned dose intensity)\*100;

For F-627, Actual dose intensity = Actual cumulative dose / Total frequency of drug administration;

For GRAN®, Actual dose intensity = Actual cumulative dose / Weight / Actual days of drug administration. The last valid weight value measured before each chemotherapy cycle will be used for analysis.

Programming notes: For visit of GRAN®, please specify the day of visit rather than list '4-21 days'.

Programming notes: relative dose intensity (%) is rounded to integer.

|---|---|---|

Listing 16.2.4.1.2 Exposure of Study Drug (F-627, GRAN®) for All Treatment Periods – Safety Analysis Set

| Treatement Group | Subject ID | Visit Visit | Dosing date / time | Actual cumulative dose (unit) | Relative dose intensity (RDI) (%)[1] |
|---|---|---|---|---|---|
| F-627 | xxxxxx | Day xx of cycle xx | YYYY-MM-DD HH:MM | xxx (mg) | XX.X |
| GRAN® | xxxxxx | Day xx of cycle xx | YYYY-MM-DD HH:MM | xxx (mg) | XX.X |
| GRAN® | xxxxxx | Day xx of cycle xx | YYYY-MM-DD HH:MM | xxx (mg) | XX.X |
| F-627 | xxxxxx | Day xx of cycle xx | YYYY-MM-DD HH:MM | xxx (mg) | xx.x |

Note: [1] Relative dose intensity (%) = (Actual dose intensity/ Planned dose intensity)\*100;

For F-627, Actual dose intensity = Actual cumulative dose / Total frequency of drug administration;

For GRAN®, Actual dose intensity = Actual cumulative dose / Weight / Actual days of drug administration. The last valid weight value measured before each chemotherapy cycle will be used for analysis.

Programming notes: For visit of GRAN®, please specify the day of visit rather than list '4-21 days'.

Programming notes: relative dose intensity (%) is rounded to integer.

|---|---|---|
|---|---|---|

Listing 16.2.4.1.3 Overdose of Study Drug (F-627, GRAN®) for All Treatment Periods – Safety Analysis Set

| Planned Treatem<br>Group | ent Subject ID | Actual Treatement<br>Grou | Overdose | Visit | Dosing date / time | Actual cumulative dose(unit) | Relative dose intensity (RDI) (%)[1] |
|---|---|---|---|---|---|---|---|
| F-627 | xxxxxx | GRAN® | | Day xx of cycle xx | YYYY-MM-D<br>HH:MM | xxx (mg) | XX.X |
| GRAN® | xxxxxx | F-627 | | Day xx of cycle xx | YYYY-MM-D<br>HH:MM | xxx (mg) | XX.X |
| GRAN® | xxxxxx | F-627 | Overdose | Day xx of cycle xx | YYYY-MM-D<br>HH:MM | xxx (mg) | XX.X |
| F-627 | xxxxxx | GRAN® | | Day xx of cycle xx | YYYY-MM-D<br>HH:MM | xxx (mg) | XX.X |

Note: [1] Relative dose intensity (%) = (Actual dose intensity/ Planned dose intensity)\*100;

For F-627, Actual dose intensity = Actual cumulative dose / Total frequency of drug administration;

For GRAN®, Actual dose intensity = Actual cumulative dose / Weight / Actual days of drug administration. The last valid weight value measured before each chemotherapy cycle will be used for analysis.

Overdose is defined as equal to or more than 20% of the prescribed dose.

Programming notes: relative dose intensity (%) is rounded to integer, and statistics for decimal places refer to SAP.

|--|--|---|---|---|
|--|--|---|---|---|

# Listing 16.2.4.1.4 Exposure of Chemotherapy drugs (Epirubicin, Cyclophosphamide) for Cycle 1– Safety Analysis Set

| Treatement<br>Group | Subject ID | Dosing date / time | Actual cumulative dose of Epirubicin (unit) | Relative dose intensity (%) | Dosing date / time | Actual cumulative dose of Cyclophosphamide | Relative dose intensity (%)[1] |
|---|---|---|---|---|---|---|---|
| F-627 | xxxxxx | YYYY-MM-DD<br>HH:MM | xxx (mg) | XX.X | YYYY-MM-DD<br>HH:MM | xxx (mg) | XX.X |
| GRAN® | xxxxxx | YYYY-MM-DD<br>HH:MM | xxx (mg) | XX.X | YYYY-MM-DD<br>HH:MM | xxx (mg) | XX.X |
| GRAN® | xxxxxx | YYYY-MM-DD<br>HH:MM | xxx (mg) | xx.x | YYYY-MM-DD<br>HH:MM | xxx (mg) | xx.x |
| F-627 | xxxxxx | YYYY-MM-DD<br>HH:MM | xxx (mg) | XX.X | YYYY-MM-DD<br>HH:MM | xxx (mg) | XX.X |

Note: [1] For chemotherapy drugs, Relative dose intensity (%) = (Actual dose intensity / Planned dose intensity)\*100, Actual dose intensity (mg/m^2/frequency) = Actual cumulative dose / Body surface area (BSA) / Total frequency of drug administration, According to the high ratio formula, Body surface area (BSA) =0.007184 × Weight (kg) ^0.425 × Height(cm) ^0.725

The last valid weight value value measured before each chemotherapy cycle will be used for calculating Body surface area (BSA).

Programming notes: relative dose intensity (%) is rounded to integer, and statistics for decimal places refer to SAP. Height is only tested once during screening.

|-------------------------------------|-------------------|-----------------|
| Generon (Shanghai) Corporation Ltd. | SP11631 | 1.0, 2020-03-11 |

Listing 16.2.4.1.5 Exposure of Chemotherapy drugs (Epirubicin, Cyclophosphamide) for All Treatment Periods – Safety Analysis Set

| Treatement<br>Group | Subject ID | Phase | Dosing date /<br>time | Actual cumulative<br>dose of Epirubicin<br>(unit) | Relative dose intensity (RDI) (%) | Dosing date / time | Actual cumulative dose of Cyclophosphamide (unit) | Relative dose intensity (RDI) (%) [1] |
|---|---|---|---|---|---|---|---|---|
| F-627 | xxxxxx | Cycle x | YYYY-MM-DD<br>HH:MM | xxx (mg) | XX.X | YYYY-MM-<br>DD HH:MM | xxx (mg) | XX.X |
| GRAN® | xxxxxx | Cycle x | YYYY-MM-DD<br>HH:MM | xxx (mg) | XX.X | YYYY-MM-<br>DD HH:MM | xxx (mg) | XX.X |
| GRAN® | xxxxxx | Cycle x | YYYY-MM-DD<br>HH:MM | xxx (mg) | xx.x | YYYY-MM-<br>DD HH:MM | xxx (mg) | XX.X |
| F-627 | xxxxxx | Cycle x | YYYY-MM-DD<br>HH:MM | xxx (mg) | XX.X | YYYY-MM-<br>DD HH:MM | xxx (mg) | xx.x |

Note: [1] For chemotherapy drugs, Relative dose intensity (%) = (Actual dose intensity / Planned dose intensity)\*100, Actual dose intensity ( $mg/m^2$ /frequency) = Actual cumulative dose / Body surface area (BSA) / Total frequency of drug administration, According to the high ratio formula, Body surface area (BSA) =0.007184 × Weight (kg)<sup>0.425</sup>× Height(cm)<sup>0.725</sup>. The last valid weight value and height value measured before each chemotherapy cycle will be used for calculating Body surface area (BSA).

Programming notes: relative dose intensity (%) is rounded to integer, and statistics for decimal places refer to SAP.

Listing 16.2.4.2.1 Adverse Event – Safety Analysis Set

| | , | | ~ | 525 200 | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatem<br>ent<br>Group | Subject ID | MedDRA SOC/ PT<br>/AE Term | Start date/<br>End date | Course<br>of AE | CTCAE<br>Grade | Causality<br>with study<br>drug | Actions on study drug | Concomitant<br>medication or<br>treatment for<br>AE | Outcome | TEA<br>E | SAE | SAE<br>Category |
| F-627 | xxxxxx | xxxxxx/ xxxxxx/<br>xxxxxx | YYYY-MM-DD /<br>YYYY-MM-DD | Day 1 of<br>Cycle 1 | Grade 1 | Possibly related | Dose reduction | Yes | Persistin<br>g | Yes | Yes | 死亡 |
| GRAN® | xxxxxx | xxxxxx/ xxxxxx/<br>xxxxxx | YYYY-MM-DD /<br>YYYY-MM-DD | Day xx<br>of Cycle<br>xx | Grade 2 | Unlikely<br>related | Dose reduction | Yes | Persistin<br>g | Yes | No | |

| Sponsor :<br>Generon ( | (Shanghai) Cor | poration Ltd. | Protocol Number :<br>SP11631 | , | Version, date : 1.0, 2020-03-11 | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| GRAN® | xxxxxx | xxxxxx/ xxxxxx/<br>xxxxxx | | YY-MM-DD /<br>YY-MM-DD | Grade 3 | Unrelated | Dose discontinu ation | Not applicable | Resolved | Yes | No |
| F-627 | xxxxxx | xxxxx/ xxxxxx/<br>xxxxxx | | YY-MM-DD /<br>YY-MM-DD | Grade 5 | Possibly related | Dose<br>discontinu<br>ation | Unknown | Cured | No | No |

Note: Adverse events are coded using MedDRA(Version 22.1).

Course of AE: the start date of AE was on day x of cycle x (day 1 of each cycle was the first day of chemotherapy in each cycle), and the Course of AEs with the start date before the first day of chemotherapy in cycle 1 was classified as "screening period".

Similar listing as listing 16.2.4.2.1:

### Listing 16.2.4.2.2 TEAE Related to Study Drug – Safety Analysis Set

Programming notes: Delete the column "Causality with study drug" in Listing 16.2.4.2.1.

### **Listing 16.2.4.2.3 Serious Adverse Event – Safety Analysis Set**

Programming notes: Delete the column "SAE" in Listing 16.2.4.2.1. Column "Course of AE" should be updated to "Course of SAE".

### Listing 16.2.4.2.4 Adverse Event leading to Study Drug Withdrawn – Safety Analysis Set

Programming notes: Only adverse events which action on study drug is "Drug Withdrawn" are displayed in this listing.

| Sponsor :<br>Generon (Shanghai) Corporati | Protocol Number :<br>SP11631 | Version, date: 1.0, 2020-03-11 |
|---|---|---|

Listing 16.2.4.3.1 Hematology - Safety Analysis Set

| Treatement<br>Group | Subject<br>ID | Parameters (unit) | Visit | Date of collection | Measurement<br>Results | High/low/Normal | Normal Range | Data source |
|---|---|---|---|---|---|---|---|---|
| F-627 | XXXXXX | White blood cell count (10^9/L) | l Screen | YYYY-MM-<br>DD | XX.X | | (xx, xx) | Local Laboratory |
| | | | Day xx of cycle xx | YYYY-MM-<br>DD | XX.X | | | Center<br>Laboratory |
| | | Neutrophil coun (10 <sup>^9</sup> /L) | t Screen | YYYY-MM-<br>DD | xx.x | Н | | |
| | | | Day xx of cycle xx | YYYY-MM-<br>DD | XX.X | | | |
| GRAN® | xxxxxx | | | | | | | |

Note: H: Above the Normal value, L: Below the Normal value, N: Normal value.

Programming notes: Visits of Hematology test: Screen, Day xx of Cycle xx, End of study.

hematology parameter specified in protocol: White blood cell count (10^9/L), Neutrophil count (10^9/L), Eosinophil count (10^9/L), Basophil count (10^9/L) etc.

| Sponsor: | Protocol Number: | Version, date : |
|-------------------------------------|------------------|-----------------|
| Generon (Shanghai) Corporation Ltd. | SP11631 | 1.0, 2020-03-11 |

Similar listing as Listing 16.2.4.3.1

Listing 16.2.4.3.2 Clinical Chemistry - Safety Analysis Set

| Treatement<br>Group | Subject<br>ID | Parameters (unit) | Visit | Date of collection | Measurement<br>Results | High/low/Normal | Normal Range |
|---|---|---|---|---|---|---|---|
| F-627 | xxxxxx | White blood cell count $(10^{9}/L)$ | Screen | YYYY-MM-DD | XX.X | | (xx, xx) |
| | | | Day xx of cycle xx | YYYY-MM-DD | XX.X | | |
| | | Neutrophil count (10^9/L) | Screen | YYYY-MM-DD | xx.x | Н | |
| | | | Day xx of cycle xx | YYYY-MM-DD | XX.X | | |
| CD ANI® | | | | | | | |
| GRAN® | xxxxxx | | | | | | |

Programming notes: Clinical Chemistry parameters specified in protocol: Alanine transaminase (ALT) IU/L), Aspartate transaminase (AST) IU/L), etc.

|-------------------------------------|-------------------|-----------------|
| Generon (Shanghai) Corporation Ltd. | SP11631 | 1.0, 2020-03-11 |

# **Listing 16.2.4.3.3 Urinalysis - Safety Analysis Set**

| Treatemen<br>t Group | Subject<br>ID | Visit | Parameters | | Measureme<br>nt Results | Unit | Date of collection | Normal Range | Clinical evaluation |
|---|---|---|---|---|---|---|---|---|---|
| F-627 | xxxxxx | Screen | PH | | XX.X | | YYYY-MM-DD | (xx, xx) | Normal |
| | | Day xx of cycle xx | Urine specific gr | avity | XX.X | | YYYY-MM-DD | | Abnormal without clinical significance |
| | | | Urine protein | | | | | | |
| | | | Casts | | | | | | Abnormal with clinical significance |
| | | Screen | Blood<br>(qualitative) | cells | XX.X | | YYYY-MM-DD | | |
| | | Day xx of cycle xx | Urine (microscopic | RBC | XX.X | | YYYY-MM-DD | | |
| | | | Urine<br>(qualitative) | WBC | | | | | |
| | | | Urine (microscopic | WBC | | | | | |
| | | | Urine glucose | | | | | | |
| | | | Urine ketones | | | | | | |
| GRAN® | xxxxxx | | | | | | | | |

|---|---|---|

Programming notes: Visits of Urinalysis test: Screen, Day xx of Cycle 1-4, End of study.

For Urinalysis test, if the result is missing and test status is "Not examined", set the value of Urinalysis parameters value as "Not examined"; if both the result and test status are missing, set the value of each Urinalysis parameters value as missing.

Urinalysis quantitative parameters: PH, Urine specific gravity, Urine protein, Casts, Blood cells (qualitative), Urine RBC (microscopic examination). Urine WBC (qualitative), Urine WBC (microscopic examination). Urine glucose, Urine ketones.

|---|---|---|
| Generon (Ghanghar) Corporation Eta. | 5111051 | 1.0, 2020-03-11 |

Listing 16.2.4.3.4 Pregnancy Test - Safety Analysis Set

| Treatement Group | Subject ID | Visit | Date of collection | Results | Data source |
|---|---|---|---|---|---|
| F-627 | xxxxxx | Screen | YYYY-MM-DD | XX.X | Local Laboratory |
| | | Day xx of cycle xx | YYYY-MM-DD | XX.X | Center Laboratory |
| | | Screen | YYYY-MM-DD | XX.X | XX.X |
| | | Day xx of cycle xx | YYYY-MM-DD | XX.X | XX.X |
| GRAN® | xxxxxx | | | | |

| Sponsor : | Protocol Number : | Version, date: |
|-------------------------------------|-------------------|-----------------|
| Generon (Shanghai) Corporation Ltd. | SP11631 | 1.0, 2020-03-11 |

Listing 16.2.4.4.1 Vital Signs - Safety Analysis Set

| Treatement<br>Group | Subject<br>ID | Visit | Date of measurement | Heart rate (beats/minute) | Systolic<br>pressure<br>(mmHg) | Diastolic<br>pressure<br>(mmHg) | Weight (kg) | Height (cm) | Weight change<br>from baseline (%) |
|---|---|---|---|---|---|---|---|---|---|
| F-627 | xxxxxx | Screen | YYYY-MM-DD | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | Day xx of cycle xx | YYYY-MM-DD | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | End of study | YYYY-MM-DD | XX.X | xx.x | xx.x | xx.x | XX.X | XX.X |
| GRAN® | | | | | | | | | |

Programming notes: Weight change from baseline (%) is rounded to integer.

| Sponsor : | Protocol Number : | Version, date: |
|-------------------------------------|-------------------|-----------------|
| Generon (Shanghai) Corporation Ltd. | SP11631 | 1.0, 2020-03-11 |

Listing 16.2.4.4.2 Body Temperature- Safety Analysis Set

| Treatement Group | Subject ID | Visit | Date of measurement | Method of measurement | Results ( $^{\circ}$ C) |
|---|---|---|---|---|---|
| F-627 | xxxxxx | Screen | YYYY-MM-DD | Oral | XX.X |
| | | Day xx of cycle xx | YYYY-MM-DD | Oral | XX.X |
| | | Screen | YYYY-MM-DD | Axillary | xx.x |
| | | Day xx of cycle xx | YYYY-MM-DD | Oral | XX.X |
| GRAN® | xxxxxx | | | | |

|-------------------------------------|-------------------|-----------------|
| Generon (Shanghai) Corporation Ltd. | SP11631 | 1.0, 2020-03-11 |

| Treatement<br>Group | Subject<br>ID | Items | Visit | Date of examination | Results | Description abnormality | of | the |
|---|---|---|---|---|---|---|---|---|
| F-627 | xxxxxx | General conditions | Screen | YYYY-MM-DD | Normal | | | |
| | | | Day xx of cycle xx | YYYY-MM-DD | Normal | | | |
| | | Neck | Screen | YYYY-MM-DD | Abnormal without clinical significance | xxxxxx | | |
| | | | Day xx of cycle xx | YYYY-MM-DD | Normal | | | |
| GRAN® | xxxxxx | | | | | | | |

|-------------------------------------|-------------------|-----------------|
| Generon (Shanghai) Corporation Ltd. | SP11631 | 1.0, 2020-03-11 |

Listing 16.2.4.5.1 12-Lead ECG - Safety Analysis Set

| Treatement<br>Group | Subject<br>ID | Visit | Date of<br>Examination | Heart rate (beats/minute) | RR<br>Interval<br>(ms) | P wave<br>Interval<br>(ms) | PQ<br>Interval<br>(ms) | PR<br>Interval<br>(ms) | QRS<br>Interval<br>(ms) | QT<br>Interval<br>(ms) | QTc<br>Interval<br>(ms) | Results / abnormal, specify |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| F-627 | XXX<br>XXX | Screen | YYYY-<br>MM-DD | XXXX | xxxx | xxxx | xxxx | xxxx | xxxx | xxxx | xxxx | Normal |
| | | Day xx of | YYYY-<br>MM-DD | xxxx | xxxx | xxxx | xxxx | xxxx | xxxx | xxxx | xxxx | Normal |
| | | | YYYY-<br>MM-DD | xxxx | xxxx | xxxx | xxxx | xxxx | xxxx | xxxx | xxxx | Abnormal without clinical significance |
| GRAN® | | | | | | | | | | | | |

| Sponsor:<br>Generon (Shanghai) Corporation Ltd. | Protocol Number :<br>SP11631 | Version, date : 1.0, 2020-03-11 |
|---|---|---|

Listing 16.2.4.5.2 Abdominal Ultrasound - Safety Analysis Set

| Treatement | Subject ID | Visit | Date of examination | Results | If abnormal, please specify |
|---|---|---|---|---|---|
| F-627 | xxxxxx | Screen | YYYY-MM-DD | Normal | |
| | | Day xx of cycle xx | YYYY-MM-DD | Abnormal with clinical significance | xxxxxxxxxx |
| | | End of study | YYYY-MM-DD | | |
| GRAN® | xxxxxx | | | | |

| Sponsor:<br>Generon (Shanghai) Corporation Ltd. | Protocol Number :<br>SP11631 | Version, date : 1.0, 2020-03-11 |
|---|---|---|

Figure 14.1.1.1 Changes of ANC Mean (log-transformed) by Time during Cycle 1 - FAS

Figure 14.1.1.1 Changes of ANC Mean (log-transformed) by Time during Cycle 1 - FAS



According to the above figure, drawn a figure about the relationship between ANC mean and days of cycle 1 by each Treatement Group (F627,GRAN®).

Programming notes: Delete the title in Figure, On the Y-axis, only values such as 0.5, 1.0, 2.0, 10 and 100 are retained;

Data point of Log values should be kept in each graph;

For each Cycle, drawn an independent graph.

|-------------------------------------|-------------------|-----------------|
| Generon (Shanghai) Corporation Ltd. | SP11631 | 1.0, 2020-03-11 |

#### Similar Figures as Figure 14.1.1.1:

- Figure 14.1.1.2 Changes of ANC Mean (log-transformed) by Time during Cycle 1 PP Analysis Set A
- Figure 14.1.1.3 Changes of ANC Median (log-transformed) by Time during Cycle 1 FAS
- Figure 14.1.1.4 Changes of ANC Median (log-transformed) by Time during Cycle 1 PP Analysis Set A
- Figure 14.1.2.1 Changes of ANC Mean (log-transformed) by Time during Cycle 2 FAS
- Figure 14.1.2.2 Changes of ANC Mean (log-transformed) by Time during Cycle 2 –PP Analysis Set B
- Figure 14.1.2.3 Changes of ANC Median (log-transformed) by Time during Cycle 2 FAS
- Figure 14.1.2.4 Changes of ANC Median (log-transformed) by Time during Cycle 2 PP Analysis Set B
- Figure 14.1.3.1 Changes of ANC Mean (log-transformed) by Time during Cycle 3 FAS
- Figure 14.1.3.2 Changes of ANC Mean (log-transformed) by Time during Cycle 3 PP Analysis Set B
- Figure 14.1.3.3 Changes of ANC Median (log-transformed) by Time during Cycle 3 FAS
- Figure 14.1.3.4 Changes of ANC Median (log-transformed) by Time during Cycle 3 PP Analysis Set B
- Figure 14.1.4.1 Changes of ANC Mean (log-transformed) by Time during Cycle 4 FAS
- Figure 14.1.4.2 Changes of ANC Mean (log-transformed) by Time during Cycle 4 PP Analysis Set B
- Figure 14.1.4.3 Changes of ANC Median (log-transformed) by Time during Cycle 4 FAS
- Figure 14.1.4.4 Changes of ANC Median (log-transformed) by Time during Cycle 4 PP Analysis Set B